# Statistical Analysis Plan



| Sponsor | Alkahest, Inc. |
|---|---|
| Protocol Title: | A Randomized, Double-Blind, Placebo-Controlled Study to<br>Assess the Safety and Tolerability of GRF6021 Infusions in<br>Subjects with Parkinson's Disease and Cognitive Impairment |
| Protocol Number: | ALK6021-201 |
| Premier Research PCN: | ALKA7951 |
| Document Version: | Version 4.0 |
| Document Date: | 17-Aug-2020 |

# Approvals

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| Lead<br>Biostatistician | Print Name: | |
| Premier Statistical<br>Reviewer | Print Name: Sign PMasia end by: | |
| Alkahest<br>Representative | Print Name: Sign के क्षित्रकृत by: | |



# **Document History**

| Version | Date | Section | Description of<br>Change/Purpose |
|---|---|---|---|
| 1.0 | 05-Feb-2019 | N/A | N/A |
| 2.0 | 21-May-2019 | 3.5 | Added additional detail about timing of randomization. |
| 2.0 | 21-May-2019 | 3.6 | Added additional detail about measures to ensure blinding of vial and drip chamber. Stated laboratory results will remain blinded until study end except for the screening value. Clarified the personnel who remain blinded and unblinded. |
| 2.0 | 21-May-2019 | 3.7 | Replaced Schedule of Events table. |
| 2.0 | 21-May-2019 | 4.2 | Clarified table presentations will be displayed in aggregate at interim analyses and no subject level listings will be provided. Added external consultants to the list of parties that may be |
| 2.0 | 21-May-2019 | 5 | involved in the Safety<br>Evaluation Meetings.<br>Updated definition of |
| | | | Evaluable Set to reflect 5 planned doses for consistency with the end of first treatment |



| | | | period. Listed additional reasons for exclusion from the Per Protocol Set. |
|---|---|---|---|
| 2.0 | 21-May-2019 | 8.3.1 | Clarified the visit in which the blood sample will be obtained for ApoE analysis |
| 2.0 | 21-May-2019 | 9.1 | Added language describing tabulations of TEAEs, AEs leading to withdrawal, Deaths and SAEs, and AESIs from previous drafts that was erroneously omitted due to subheading formatting. |
| 2.0 | 21-May-2019 | 9.1.3 | Removed the AESI criteria as these are left to the discretion of the PI. Added text describing new table presenting AEs associated with blood pressure changes by infusion period, SOC, PT, and treatment. |
| 2.0 | 21-May-2019 | 9.2 | Added descriptions of screening, pre-infusion, and exit safety laboratory evaluations from previous drafts that was erroneously omitted due to subheading formatting. Explicitly stated the visits in which |





| | | | would be listed. |
|---|---|---|---|
| | | | Stated shifts from baseline in coagulation and quantitative urinalysis parameters will also be provided. |
| 2.0 | 21-May-2019 | 9.3 | Clarified the visits in which orthostatic vital signs will be presented pre- and post-infusion. |
| | | | Clarified the position of abnormal vital signs and added criterion of orthostatic hypotension. |
| | | | Included reference to<br>the blood pressures of<br>special interest that will<br>be summarized<br>separately. |
| 2.0 | 21-May-2019 | 10 | Stated that BPSIs were identified and summarized in the SAP, but are not in the current protocol version. |
| 2.0 | 21-May-2019 | 11.1 | Clarified the Hoehn<br>and Yahr will be used,<br>not the modified Hoehn<br>and Yahr. |
| 2.0 | 21-May-2019 | 11.3 | Added a subsection to detail the echocardiogram results that will be listed. |
| 2,0 | 21-May-2019 | 13.1 | Indicated which demographic and safety TFLs will also be provided at the efficacy IA. |



| 2.0 | 21-May-2019 | 14.2 | Updated footnotes,<br>titles, and table shell<br>formatting for<br>consistency with text<br>and other shells. |
|---|---|---|---|
| | | | Added a table of AEs with terms associated with blood pressure changes. |
| | | | Added summary and shift tables of coagulation and quantitative urinalysisf laboratory parameters. |
| | | | Added a table of blood pressure values of special interest. |
| 2.0 | 21-May-2019 | 14.3 | Added listings of coagulation, immunology, and serology laboratory parameters. |
| | | | Added a column to the protocol deviations listing to indicate which deviations exclude someone from the Per Protocol analysis Set. |
| 3.0 | 01-May-2020 | 8.3.2 | Added subsections for<br>Volumetric MRI,<br>Resting fMRI, and<br>ASL MRI describing<br>what tests, locations<br>and laterality will be<br>presented. |
| 3.0 | 01-May-2020 | 13.2 | Removed the 'X' from<br>ANCOVA tables as<br>they were not provided |



| | | | and the interim efficacy<br>analysis |
|---|---|---|---|
| 3.0 | 01-May-2020 | 14.2 | Added table shells for<br>Volumetric MRI and<br>ASL MRI |
| 3.0 | 01-May-2020 | 14.3 | Added listing shells for<br>Volumetric MRI and<br>ASL MRI |
| 3.0 | 01-May-2020 | 14.4 | Added figure shells for<br>the individual MDS-<br>UPDRS scores (Part 1,<br>Part 2, and Part 3) |
| 4.0 | 17-Aug-2020 | 5 | Refined Per Protocol<br>set definition, Added<br>Complete population |
| 4.0 | 17-Aug-2020 | 7.1 | Added description of subjects who did not complete the study due to COVID-19 |
| 4.0 | 17-Aug-2020 | 9.1.1 | Added derived action taken variable for AEs |
| 4.0 | 17-Aug-2020 | 13 | Added medical history<br>table by LLT, added<br>efficacy tables in the<br>Complete Set |
| 4.0 | 17-Aug-2020 | 14 | Added medical history<br>table shell and efficacy<br>table shells for<br>Complete Set |
| | | | Updated footnotes,<br>titles, columns for<br>consistency with text |





# **Table of Contents**

| Document History | 1 |
|---|---|
| List of Tables List of Figures 1. Overview 2. Study Objectives and Endpoints 2.1. Study Objectives 2.1.1 Primary Objective 2.1.2. Secondary Objectives 2.1.3. Exploratory Objectives | 2 |
| List of Figures | 7 |
| 1. Overview | 9 |
| 2. Study Objectives and Endpoints 2.1. Study Objectives 2.1.1. Primary Objective 2.1.2. Secondary Objectives 2.1.3. Exploratory Objectives | 9 |
| 2.1. Study Objectives 2.1.1 Primary Objective 2.1.2 Secondary Objectives 2.1.3 Exploratory Objectives | 10 |
| 2.1.1. Primary Objective | 10 |
| Secondary Objectives 2.1.3. Exploratory Objectives | 10 |
| 2.1.3. Exploratory Objectives | 10 |
| | 10 |
| 2.2. Study Endpoints | 10 |
| | 11 |
| 2.2.1. Safety Endpoints | |
| 2.2.2. Efficacy Endpoints | |
| 3. Overall Study Design and Plan | 12 |
| 3.1. Overall Design | 12 |
| 3.2. Sample Size and Power | 12 |
| 3.3. Study Population | 13 |
| 3.4. Treatments Administered | 13 |
| 3.5. Method of Assigning Subjects to Treatment Groups | 13 |
| 3.6. Blinding and Unblinding | 13 |
| 3.7. Schedule of Events | 14 |
| 4. Statistical Analysis and Reporting | 18 |
| 4.1. Introduction | 18 |
| 4.2. Interim Analysis and Data Monitoring | 18 |
| 5. Analysis Sets | 19 |
| General Issues for Statistical Analysis | 22 |
| 6.1. Statistical Definitions and Algorithms | 22 |
| 6.1.1. Baseline | |
| 6.1.2. Adjustments for Covariates | |
| 6.1.3. Multiple Comparisons | 22 |
| 6.1.4. Handling of Dropouts or Missing Data | 23 |
| 6.1.5. Analysis Visit Windows | |
| 6.1.6. Pooling of Sites | 23 |
| 6.1.7. Derived Variables | |
| 6.1.8. Data Adjustments/Handling/Conventions | |





| 7. | St | udy Subjects and Demographics | . 2 |
|---|---|---|---|
| | 7.1. | Disposition of Subjects and Withdrawals | . 27 |
| | 7.2. | Protocol Violations and Deviations | . 27 |
| | 7.3. | Demographics and Other Baseline Characteristics | . 2 |
| | 7.4. | Exposure | |
| 8. | Ef | ficacy Analysis | . 28 |
| | 8.1. | Primary Efficacy Analysis | |
| | 8.2. | Secondary Efficacy Analysis | |
| | 8.2.1. | Montreal Cognitive Assessment (MoCA) | . 28 |
| | 8.2.2. | Cognitive Drug Research Computerized Cognition Battery (CDR-CCB) | 29 |
| | 8.2.3. | Delis-Kaplan Executive Function Verbal Fluency (D-KEFS) | |
| | 8.2.4. | Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | |
| | 8.2.5. | Schwab and England Activities of Daily Living Scale (SE-ADL) | . 30 |
| | 8.2.6. | Clinical Impression of Severity Index - Parkinson's Disease (CISI-PD) | 32 |
| | 8.2.7. | Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39) | . 32 |
| | 8.2.8. | Geriatric Depression Scale-15 (GDS-15) | . 33 |
| | 8.2.9. | Digital Clock Drawing Test (dCDT) | . 33 |
| | 8.3. | Exploratory Efficacy Analysis | . 34 |
| | 8.3.1. | Apolipoprotein E (ApoE) Genotype Testing | 34 |
| | 8.3.2. | Magnetic Resonance Imaging (MRI) | 34 |
| 9. | Sa | fety and Tolerability Analysis | 36 |
| | 9.1. | Adverse Events | 36 |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 37 |
| | 9.1.2. | Deaths and Serious Adverse Events | 38 |
| | 9.1.3. | Other Significant Adverse Events | 38 |
| | 9.2. | Laboratory Evaluations | 38 |
| | 9.3. | Vital Signs | 39 |
| | 9.4. | Electrocardiograms (ECGs) | 40 |
| | 9.5. | Further Safety Evaluations | 40 |
| | 9.5.1. | Physical Examination | 40 |
| | 9.5.2. | Sheehan-Suicidality Tracking Scale (S-STS) | 40 |
| | 9.6. | Concomitant Medication | 41 |
| 10. | Cl | anges from Planned Analysis | 41 |
| 11. | | her Planned Analysis | |
| | 11.1. | Hoehn and Yahr Scale | 41 |
| | 11.2. | Modified Hachinski Ischemic Scale (MHIS) | |
| | 11.3. | Echocardiogram | 42 |
| AD- | ST-33.05 | Effective date: 22-Jan-2018 | |



| Statistical Analysis Plan, |
|-----------------------------|
| Sponsor Alkahest, Inc. |
| Protocol Number ALK6021-201 |
| PCN Number ALK A7951 |

| - | rer | Number ACKA751 | |
|------|---------|-------------------------------------------------------|-----|
| 12. | R | eferences | 42 |
| 13. | Ta | ables, Listings, and Figures | 42 |
| | 13.1. | Planned Table Descriptions | 43 |
| | 13.2. | Efficacy Data Tabulations | 44 |
| | 13.3. | Safety Data | 48 |
| | 13.4. | Planned Listing Descriptions | 50 |
| | 13.5. | Planned Figure Descriptions | 51 |
| 14. | Ta | ables, Listings, and Figures (TLF) Shells | 54 |
| | 14.1. | Standard Layout for all Tables, Listings, and Figures | 54 |
| | 14.2. | Planned Table Shells | 56 |
| | 14.3. | Planned Listing Shells | 111 |
| | 14.4. | Planned Figure Shells | 145 |
| App | endix | 1: Premier Research Library of Abbreviations | 152 |
| App | endix | 2: Bracket Statistical Analysis Plan for CDR | 156 |
| | | Γables | |
| Tab | le 1: S | Schedule of Events | 15 |
| Tab | le 2: I | Demographic Data Summary Tables and Figures | 44 |
| Tab | le 3: I | Efficacy Data | 44 |
| Tab | le 4: S | Safety Data | 48 |
| Tab | le 5: I | Planned Listings | 50 |
| Tab | le 6: I | Planned Figures | 51 |
| Lis | t of l | Figures | |
| Figu | re 1: | Study Schema | 12 |
| 100 | | Standardized Layout | |



### Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Alkahest protocol number ALK6021-201 (A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Tolerability of GRF6021 Infusions in Subjects with Parkinson's Disease and Cognitive Impairment), dated 08MAR2019 V4.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup> All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>2</sup> and the Royal Statistical Society<sup>3</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to Alkahest's study ALK6021-201.

# 2. Study Objectives and Endpoints

### 2.1. Study Objectives

# 2.1.1. Primary Objective

The primary objective of the study is to assess the safety and tolerability of GRF6021, a human fraction administered by intravenous (IV) infusion, in subjects with Parkinson's disease (PD) and cognitive impairment.

### 2.1.2. Secondary Objectives

As a secondary objective, the study aims to assess the effects of GRF6021 on cognitive and motor function.

# 2.1.3. Exploratory Objectives

The exploratory objectives include blood and plasma collection to identify specific biomarkers associated with cognitive and motor function and/or indicators of PD with mild cognitive impairment (PD-MCI) and PD with dementia (PDD) progression. In addition, magnetic resonance imaging (MRI) of the brain will be conducted after the second dosing period in consenting subjects to identify potential therapeutic effects of GRF6021.

### 2.2. Study Endpoints

### 2.2.1. Safety Endpoints

### 2.2.1.1. **Primary Safety Endpoints**

The primary safety endpoints of this study include the following:

Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) identified by the Medical Dictionary for Regulatory Activities (MedDRA) preferred term (PT) and grouped by MedDRA System Organ Class (SOC).

### 2.2.1.2. Secondary Safety Endpoints

The secondary safety endpoints include the following:

- Change from baseline in clinical laboratory parameters.
- Change from baseline in vital sign measurements.
- Change from baseline in body weight.
- Change from baseline in the S-STS.

### 2.2.2. **Efficacy Endpoints**

### 2.2.2.1. Primary Efficacy Endpoint

Not Applicable.

### 2.2.2.2. Secondary Efficacy Endpoint(s)

The secondary efficacy endpoints of this study include the following:

- Change from baseline in the Montreal Cognitive Assessment (MoCA).
- Change from baseline in Continuity and Power of Attention, Working Memory, and Episodic Memory on the Cognitive Drug Research Computerized Cognition Battery (CDR-CCB).
- Change from baseline in Delis-Kaplan Executive Function System (D-KEFS) Verbal
- Change from baseline in the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) 1, 2, 3, and total score.
- Change from baseline in the Schwab and England Activities of Daily Living (SE-ADL) Scale.
- Change from baseline in the Clinical Impression of Severity Index PD (CISI-PD).
- Change from baseline in the PD Quality of Life Questionnaire-39 (PDQ-39).
- Change from baseline in the Geriatric Depression Scale-15 (GDS-15).
- Change from baseline in the digital clock drawing test (dCDT).

### 2.2.2.3. Exploratory Efficacy Endpoint(s)

The exploratory efficacy endpoints of this study include the following:



- Serial compositional analysis of individual subject's plasma to identify specific biomarkers associated with cognitive functional changes and/or indicators of disease progression.
- Epigenetic changes.
- Change from baseline in the following assessments (in consenting subjects):
  - Brain morphometry as measured by MRI.
  - Functional connectivity as measured by task-free functional MRI (tf-fMRI), where available.
  - Cerebral blood flow assessments as measured by arterial-spin labeling (ASL) MRI, where available.

# 3. Overall Study Design and Plan

# 3.1. Overall Design

This is a randomized, double-blind, placebo-controlled study to assess the safety and tolerability of GRF6021, a human human fraction, administered by IV infusion to subjects with PD and cognitive impairment.

All subjects will undergo a screening visit, including an MRI scan, baseline visit, 2 dosing periods, follow-up visits, and an end-of-study/early-termination visit. Each dosing period (Treatment 1, starting at Week 1; and Treatment 2, starting at Week 13) consists of 5 consecutive days ("pulsed dosing") of IV infusions of of either GRF6021 or placebo. During each 5-day dosing period, subjects will reside in inpatient units and can be discharged after the fifth day of dosing. The subject participation period is approximately 7 months from Screening through End of Study, unless prematurely discontinued.

Safety and tolerability assessments will occur at every visit. Cognitive and motor testing will be performed at Baseline and at periodic interim visits following dosing.

The overall schema of the study is presented in Figure 1:

Figure 1: Study Schema



### 3.2. Sample Size and Power

A total of approximately 90 subjects will be randomized in a 2:1 ratio to active treatment (approximately 60 subjects) or placebo (approximately 30 subjects), with the intent of obtaining ~68 evaluable subjects who have received at least 5 doses and completed the study through Visit



Subjects who discontinue before completing Visit 8 may be replaced. Subjects who withdraw or are withdrawn during screening will be replaced.

The study is not statistically powered to detect differences in measures of clinical efficacy or biomarker endpoints. To evaluate potential safety signals, the statistical approximation described by Hanley (aka the "Rule of Threes" in which the upper bound of the 95% confidence interval [CI] for the frequency of an unreported AE is at most 3/n %, where n represents the number of subjects who received active GRF6021 in the study) will be used. In a sample of 60 subjects, the upper bound of the 95% CI for the frequency of an unobserved AE is approximately 5%. In addition, the proposed sample size may be sufficient to identify trends in efficacy endpoints that will be used to determine the appropriate sample size for subsequent studies.

### 3.3. Study Population

This study includes male and female subjects, aged 40-85 years old, with a diagnosis of either PD-MCI or PDD.

### 3.4. Treatments Administered

| GRF6021 is a human | fraction made from pooled human plasma product |
|---|---|
| | that serves as a viable source of soluble, |
| infusible plasma proteins from h | ealthy male and female donors. It is administered by IV infusior |
| of to subjects. The place | bo control agent will be 0.9% sodium chloride injection, USP |
| (saline). Each infusion will have | a duration of approximately with a maximum of |
| . The infusion of active and | placebo agents will be identical to maintain blinding. Subjects |
| will receive one infusion of | per day for 5 consecutive days at Weeks 1 and 13. |

# 3.5. Method of Assigning Subjects to Treatment Groups

Subjects will be randomized to GRF6021 (Group 1: active dosing in both dosing periods) or placebo (Group 2: placebo dosing in both dosing periods) in a 2:1 ratio. Randomization will be stratified by sex to ensure a balanced distribution of male and female subjects in both treatment groups. Subjects will be randomized at the conclusion of Visit 2, after eligibility has been confirmed (including MRI and echocardiography results).

### 3.6. Blinding and Unblinding

The following measures will be taken to ensure adequate allocation concealment during infusions: blinding of subjects, trial partners, study coordinators, physicians, and cognitive/motor test administrators to treatment allocation; use of blinded Outcomes Assessors and unblinded Infusion Nurses; and measures to block view of the vial or bag, infusion pump, IV tubing, and catheter throughout the infusion.

The study agent/placebo to be administered will be dispensed by an unblinded pharmacist (or other qualified personnel responsible for drug accountability) to an unblinded Infusion Nurse. Administration of the study agent/placebo will be performed by the unblinded Infusion Nurse, and all study outcome measures will be assessed by a blinded Outcomes Assessor.

To ensure that Outcomes Assessors, raters, and other study personnel, as well as subjects and trial partners are unaware of the allocation, appropriate measures will be taken to mask the study agent/placebo containers and IV setup such that they will only be visible as necessary to the unblinded Infusion Nurse. In addition, the vial and drip chamber will be covered with an opaque black bag or equivalent; a curtain, drape, or equivalent will be used to shield the infusion


Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



administration setup; used vials/containers of the study agent or placebo will be concealed during transport and returned to the pharmacy at the end of the Infusion Period.

To avoid potential unblinding based on subject levels, lab results (aside from those tested at screening) will remain blinded until the conclusion of the study. Unblinding lab results would only occur for emergent safety reasons.

Communication between the blinded Outcomes Assessor and the unblinded Infusion Nurse will be restricted to only that required to ensure the immediate safety of subjects. Except for the designated personnel whose sole responsibility necessitates access to unblinding information (e.g. the unblinded CRA whose sole responsibility is to ensure study agent or placebo accountability, the unblinded clinical supply manager, etc.) and the unblinded statistician performing the interim analyses, the study Sponsor and their representatives will be blinded with respect to subjects' treatment allocation through database lock unless breaking the blind is required for safety reasons. The study blind can be broken for safety reasons if the information is required for the management of SAEs or severe AEs.

### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 1.



# Table 1: Schedule of Events

| | Screening | Baseline<br>Visit | | Ţ | Treatment | 1 | | Follow-up | | | Treat | Treatment | | - | | <b>F</b> оВоя-up | H | End of<br>Study/Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1. | . 2 | 3 | * | 5 | 9 | 7 8 | 6 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 81 | 61 |
| Infusion Number | | | - | 2 | 3 | 4 | | | | | | 00 | 0, | $\overline{}$ | | | | |
| Day | Day -35 to -8 | Day -7 to -1 | | 2 | 3 | 7 | 5 6+3 days. | | 28 ± 7 days 56 ± 7 days | 85=7 days | 86 | 87 | 88 | 89 90 | +3 days | 112 ± 7 days | 90+3 days 112±7 days 140±7 days 168±7 days | 168 ± 7 days |
| Week | 1 | | | | | 1 | | 7 | 8 | | | | 3 | | | 16 | 20 | 24 |
| Informed Consent/Opnonal MRI Consent | X | | | | - | H | | | | | | | | - | ľ | | | |
| Medical History | X | | | | | | | | | | | 1 | | - | | | | |
| Demographics | X | | | | | | | | | | | | | H | Ī | | | |
| Vital Signs | × | X | × | X | X | X | X X | x | X | × | X | × | × | N | × | X | X | × |
| Physical Exam | × | | | | | - | | | | | | | | - | | | | X |
| Height | Х | | | | | V | | | | | 1 | | | | | | | |
| Weight | X | | X | įX | 1X | X X | $X \mid X$ | | | X | 7/2 | i.X | H | X. | X | | | X |
| Supme and Standing Blood Pressure | X | | $X_{\Pi}$ | r <sub>X</sub> | X:3 ) | X PX | X TX | | | FX | Z. | N. | N. | X13 | × | | | |
| 12-lead ECG | X | | | | - | 2 | X. | | | × | | | | 1/2 | | | | |
| Echocardiogram | .X. | | | | | | | | | | | | | | | | | |
| MRI | .X. | | | | | | | | | | | | | | N | | | |
| Randomization | | X | | | | | | | | | | | | | | | | |
| Targeted Physical Exam | | | × | | X | _ | 7. | | | × | | 1 | | - N | | | | |
| Concomitant Medication Review | X | X | × | ,X | X | X <sub>1</sub> X | X | x | × | W | N. | X | 1× | Z. | × | X | 1. | × |
| Adverse Event Review | | X | X | × | - | - | X, X | × | × | X | × | 74 | 'n | - X | × | × | X | X |
| GRE6021/Placebo Infusion | | | 1 | × | V | 1 | 1 | | | 1 | 4 | 1 | X | X | | | | |
| Blood/Urine Sampling | | | | | | | | | | | | | | | | | | |
| Screening Safety Lab Panel | X | | | | | | | | | | | | | - | | | | |
| Exit Safety Lab Panel | | | | | | | | | | | | | | | | | | × |
| Pre-Infusion Safety Labs (performed onsite) | | | × | ī×, | | I.V. | | | | × | P. | | × | - | | | | |
| Pregnancy Testing* | X | | Z. | | | 7 | | | | , X | | | | | | | | |
| Comprehensive Labs' | | | | | | X, | × | × | | | | | Z, | | × | X | | |
| Proteomics/Epigenetics/Biobanking | | | X, | | 1 | | X | Х | X | X | | | | | X | X | X | X |
| ApoE Genotype Testing | | | X. | | | | | | | | | | | | | | | |
| Cognitive and Motor Testing | | | | | | | | | | | | | | | | | | |
| NHIS | X | | | | Ü | | | 1 | | | | | | | | | | |
| S-STS | X | | X | | | | X. | | | | | | | | | | | |
| MoCA | X | | | | | | | X | | | | | | | | X | | |
| Hoelm and Yahr | X | | | | | | | | | | | | | | | | | |
| CDR-CCB | 1/4 | X | | | | - | × | × | × | | | | | | × | X | X | 4 |
| D-KEFS | | X | | | | - | X | | X | | L | | | | X | | Х | |
| ACDI | | X | | | | | × | | X | | | | | | × | | X | |
| MDS-UPDRS 1/2/3 | | X | | | - | - | X | X | X | | 1 | | | | X | × | × | × |
| SE-ADL | | X | | | - | - | | | × | | | | | | | | | x |
| CISI-PD | | X | | | | 100 | | 7 - 7 | X | | | | | | | | | X |
| PDQ-39 | | × | | | | 8 | | X | X | | | | | | | | X | × |
| GDS-15 | | X | | | | - | | | × | | | | | | | | X | |

Notes: \*It is recommended, but not required, that the echocardiogram and screening MRI be performed after all other screening criteria have been met. The echocardiogram and screening MRI may be performed in any order.

X1: To be performed prior to infusion start.



| T. C. L. | Intrision. |
|----------|------------|
| d | aller |
| L. C. | Delionined |
| 1 | ğ |
| E | 07 |
| 77 | < |

X<sup>2</sup>: To be performed post-infusion (approximately

X4: If shipping of study agent to the study site will be required, subjects should be randomized at least 3 days prior to treatment start to ensure study agent availability. a: The Screening Visit may be split to allow for sufficient time to complete all procedures. AEs and concomitant medications should be reviewed during split visits, as applicable.

b: The treatment window is 5 days. Visits 8 and/or 16 may occur 1-3 days later.

c: The visit window for Visit 11 is Day 85 ±7 days. Visits 12-15 should follow consecutively.

d: Blood pressure (BP) should be taken after the subject has been lying down for at least 10 minutes (supine). The subject should then stand for 3 minutes, and the BP should be taken again.

B6), thiamine (vitamin B1), TSH, direct antiglobulin test, BNP, serum 1gA, haptoglobin, and C1 inhibitor (availability of C1 e: Includes all comprehensive labs, infectious serology (HIV, HBV, HCV), cobalamin (vitamin B12), pyridoxine (vitamin inhibitor lab results not required for evaluation of I/E criteria). Urine drug screen: cannabinoids, benzodiazepine, barbiturates, opiates, cocaine, amphetamines, methadone, phencyclidine, propoxyphene. Urinalysis: UPCR.

f. Includes all comprehensive labs, infectious serology, and direct antiglobulin test.

g: Samples for local pre-infusion labs should be collected and results interpreted PRIOR to the following day's infusion start. The following should be measured: sodium, potassium, ionized calcium, BUN, creatinine, hematocrit, hemoglobin, platelets.

h: Serum pregnancy test required at screening. Serum and/or urine pregnancy test may be used at subsequent timepoints. Results from pregnancy tests conducted at Visits 3 and 11 must be available prior to dosing.

magnesium, phosphate, potassium, protein total, sodium, triglycerides, BUN, albumin, aPTT, PT/INR, CBC with differential chloride, cholesterol, LDL, HDL, CK, creatinine, GGT, glucose (random), iron, lactate dehydrogenase (LDH or LD), lipase, gravity, nitrite, leukocytes, bilirubin, urobilinogen, urine creatinine, urine albumin, albumin/creatinine ratio, urine sodium, (basophils, eosinophils, lymphocytes, monocytes, neutrophils). Urinalysis: blood, glucose, ketone, protein, pH, specific i: Comprehensive labs: ALP, ALT, amylase, AST, bicarbonate, bilirubin (direct, indirect, and total), ionized calcium, sodium/creatinine ratio, urine potassium, potassium/creatinine ratio, and reflex urine microscopy if indicated.

The second, additional MRI will be performed in consenting subjects only and should be performed at Visit 16 + 7 days.



Task-free functional MRI and arterial-spin labeling MRI will be performed only at a subset of sites.

k: The CDR-CCB will require two training sessions prior to the baseline assessment. These training sessions can be performed at any time during the screening period.





### 4. Statistical Analysis and Reporting

### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for each treatment group, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population with non-missing data at each visit.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified. Percentages will not be displayed when the numerator for a cell is 0.

Unless otherwise indicated, all statistical tests will be conducted at the 0.05 significance level using 2-tailed tests, and P values will be reported. Corresponding 95% CIs will be presented for statistical tests.

### 4.2. Interim Analysis and Data Monitoring

An unblinded interim analysis of the safety endpoints, including the primary endpoint and secondary safety endpoints, is planned when approximately 20 subjects have completed Visit 8 (end of first dosing period). The requirement that subjects remain in an inpatient unit during each dosing period was included in the protocol to enable safety monitoring during dosing. Once the Sponsor has reviewed the safety data from this interim analysis, the need for inpatient stays during dosing will be reassessed.

An unblinded interim analysis of the MoCA, CDR-CCB, and MDS-UPDRS Part 3 secondary efficacy endpoints is planned when approximately 40 subjects have completed Visit 8 (end of first dosing period). As the study is not powered for efficacy and no decisions will be made regarding stopping the trial, statistical testing will be performed at the 0.05 level using two-tailed tests on both the Evaluable and Per Protocol sets. To minimize potential bias of the remaining efficacy and safety data, only aggregated summary tables will be provided. The data will be provided in aggregate fashion so the difference between study agent and placebo is compared but individual treatment allocation remains blinded. An independent statistician other than the author of this plan will perform the unblinded analysis.



Safety will be monitored on an ongoing basis. If safety events of potential concern occur during the trial (i.e., 3 related events in the same SOC or a suspicious overall pattern), a Safety Evaluation Meeting will be triggered and an ad hoc interim safety analysis will be performed. Dosing may be temporarily halted based on the observations. The purpose of the meeting is for investigators, the Sponsor, external consultants with expertise relevant to the specific safety signal(s) detected as necessary, and the contract research organization (CRO) Medical Monitor(s) to discuss and evaluate the safety of the subjects using available aggregated safety data and without compromising study blinding, unless the Sponsor deems unblinding necessary for safety evaluation.

The results that will be presented for each interim analysis are flagged in the table of contents. A separate analysis plan will be prepared for the CDR-CCB endpoints.

### 5. Analysis Sets

The following analysis sets are planned for this study:

- Safety Set: The Safety Set includes all subjects all subjects who receive at least 1 dose of
  the study agent. All safety analyses will be performed using the Safety Set, based on
  treatment received.
- Intent-To-Treat Set (ITT): The ITT Set includes all randomized participants. The
  presentation of baseline characteristics will be conducted on the ITT Set.
- Evaluable Set: The Evaluable Set includes all subjects who receive at least 5 of the 10 planned doses and complete through Visit 8. All efficacy analyses will be performed using the Evaluable Set, based on randomized treatment.
- Per Protocol Set (PP): The PP Set is a subset of the Evaluable set comprised of subjects who receive all 10 planned doses, who complete Visit 18 and Visit 19 in window, and who do not have any of the deviations listed below or any other deviation that could potentially affect the assessment of efficacy identified prior to database lock. Visit windows are found in Section 6.1.5. Deviations related to novel coronavirus disease 2019 (COVID-19) will also be evaluated in determining Per Protocol population eligibility prior to database lock. All efficacy analyses will be repeated in the Per Protocol Set, based on randomized treatment.
- Complete Set: The Complete Set is a subset of the PP Set comprised of subjects who did not have any changes to any of the following concomitant medications preferred terms reported at any time on study: Dopaminergic agents (e.g. Rotigotine [Neupro Patch], Duopa Pump, Sinemet [Carbidopa, Levodopa], Carbidopa, Rytary), Pregabalin (Lyrica), Amantadine, Antipsychotics (e.g. Pimavanserin Tartate [Nuplazid], Clozapine, Quetiapine Fumarate [Seroquel]), or benzodiazepines (e.g. Alprazolam). This includes those that were stable per protocol prior to first dose and either changed dose or stopped on study as well as those that began on study.

| Deviation D<br>Type | eviation | Major/Minor | Excluded<br>from Per<br>Protocol Set | Additional<br>Clarification |
|---|---|---|---|---|
|---|---|---|---|---|



| Eligibility | I2. Diagnosis of clinically established or clinically probable PD according to MDS-PD criteria (Postuma 2015)(Appendix 8) with at least 1 year of PD symptoms | Major | Yes | |
|---|---|---|---|---|
| Eligibility | I3. Diagnosis of PD-MCI (Level I, i.e. impairment on a scale of global cognitive abilities validated for use in PD) or probable or possible PDD according to MDS criteria (Litvan 2012, Emre 2007)(Appendix 9) | Major | Yes | |
| Eligibility | I4. Score on the MoCA of<br>13-25, inclusive (Nasreddine<br>2005)(Appendix 1) | Major | Yes | |
| Eligibility | I5. Hoehn and Yahr Stages 1-4 | Major | Yes | |
| Eligibility | I6. If on dopaminergic therapy (e.g., levodopa, dopamine agonists, monoamine oxidase inhibitors, catechol-O-methyl transferase inhibitors, amantadine), must be on stable dosage at least 4 weeks prior to baseline | Major | Yes | only if<br>change in the<br>last 2 weeks |
| Eligibility | I7. If on medications for cognition (e.g., rivastigmine, galantamine, donepezil, memantine), must be on stable dosage for at least 8 weeks prior to baseline | Major | Yes | only if<br>change in the<br>last 4 weeks |
| Eligibility | I8. If on antidepressant medications, must be on stable dosage for at least 8 weeks prior to baseline | Major | Yes | only if<br>change in the<br>last 4 weeks |



| Eligibility | <ul><li>If on clozapine,</li><li>quetiapine, or pimavanserin,</li><li>must be on stable dosage for</li><li>8 weeks prior to baseline</li></ul> | Major | Yes | only if<br>change in the<br>last 4 weeks |
|---|---|---|---|---|
| Eligibility | I12. Modified Hachinski<br>Ischemic Scale (MHIS) score<br>of 4 or less (Rosen 1980) | Major | Yes | |
| Eligibility | E4. Treatment with any human blood product, including transfusions and IV immunoglobulin, during the 6 months prior to screening | Major | Yes | |
| Eligibility | E19. Positive urine drug screen. The presence of opioids, benzodiazepines, and/or amphetamines in the urine drug screen may be allowed if these are prescribed and the dose stable for at least 8 weeks prior to screening | Major | Yes | |
| Eligibility | E23. Concurrent participation in any other therapeutic treatment trial. If there was prior clinical trial participation, subject must have discontinued investigational agents for at least 30 days for small molecules, and 1 year for active or passive immunotherapies prior to screening | Major | Yes | |
| Eligibility | E24. If on deep brain stimulation (DBS), DBS surgery within 12 months of screening and/or a change in DBS settings within 12 weeks of screening. DBS settings must not be changed at any point during the subject's participation in the trial | Major | Yes | |



| Eligibility | E26. More than 2 lacunar strokes or other clinically relevant imaging abnormality on screening MRI | Major | Yes | |
|---|---|---|---|---|
| Eligibility | E27. Any other condition<br>and/or situation that the<br>investigator believes may<br>interfere with the safety of<br>the subject, study conduct, or<br>interpretation of study data | Major | Yes | Only when<br>interfering<br>with the<br>interpretation<br>of study data |
| Compliance | Incorrect treatment dispensed and administered to subject | Major | Yes | |
| Out of<br>Window | Efficacy Procedures performed outside of the protocol window which are a consistent pattern or potential risk to study data outcomes | Major | Yes | |
| Study Drug<br>Temp<br>Excursion | Study drug temperature<br>excursions when determined<br>to have impacted the quality<br>of the study drug | Major | Yes | |
| Concomitant<br>meds | Use of prohibited concomitant medications as defined in the protocol that have an effect on cognition | Case by Case | | |

# 6. General Issues for Statistical Analysis

# 6.1. Statistical Definitions and Algorithms

### 6.1.1. Baseline

The last observation recorded before the first dose will be used as the baseline observation for all calculations of change from baseline.

# 6.1.2. Adjustments for Covariates

If there is a statistical difference among treatment groups with respect to baseline characteristics or values, that variable may be added to the statistical models as covariate to determine the effect on treatment. Baseline scores will be added as a covariate in models to assess efficacy.

### 6.1.3. Multiple Comparisons

No adjustments will be made for multiple comparisons for any endpoint.



# 6.1.4. Handling of Dropouts or Missing Data

Subjects who discontinue or are unblinded before Visit 8 may be replaced. Subjects who withdraw or are withdrawn during screening will be replaced. Subjects who have received at least 1 dose but are withdrawn or withdraw from the study will be encouraged to complete the end of study procedures within 4-6 weeks of their last visit.

Missing data will not be imputed.

# 6.1.5. Analysis Visit Windows

Visits will be analyzed as scheduled. Unscheduled and/or repeated measurements will only be included if a scheduled measurement is not available and the unscheduled/repeated measurement falls within the analysis visit windows as described below. The windows follow the Schedule of Events in Table 1. Unscheduled/repeated measurements will be listed.

| Visit | Target Start Day | Lower Limit | Upper Limit |
|-------|------------------|-------------|-------------|
| 1 | | -35 | -8 |
| 2 | | -7 | -1 |
| 3 | -1 | 1 | 1 |
| 4 | 2 | 2 | 2 |
| 5 | 3 | 3 | 3 |
| 6 | 4 | 4 | 4 |
| 7 | 5 | 5 | 5 |
| 8 | 6 | 6 | 9 |
| 9 | 28 | 21 | 35 |
| 10 | 56 | 49 | 63 |
| 11 | 85 | 78 | 92 |
| 12 | 86 | 79 | 93 |
| 13 | 87 | 80 | 94 |
| 14 | 88 | 81 | 95 |
| 15 | 89 | 82 | 96 |
| 16 | 90 | 83 | 100 |
| 17 | 112 | 105 | 119 |
| 18 | 140 | 133 | 147 |
| 19 | 168 | 161 | 175 |

### 6.1.6. Pooling of Sites

Not Applicable.

# 6.1.7. Derived Variables

MoCA Total score = sum of individual item scores, with a range from 0 to 30.



- D-KEFS Letter Fluency Total Correct Score = sum of F+A+S correct responses from 1-15, 16-30, 31-46, and 46-60 seconds.
- D-KEFS Category Fluency Total Correct Score = sum of Animals and Boys' Names correct responses from 1-15, 16-30, 31-46, and 46-60 seconds
- D-KEFS Category Switching Total Correct Score = sum of Fruits/Furniture correct responses from I-15, 16-30, 31-46, and 46-60 seconds.
- D-KEFS Total Correct Score = sum of D-KEFS Letter Fluency Total Correct Score, Category Fluency Total Correct Score, and D-KEFS Category Switching Total Correct Score.
- MDS-UPDRS Part 1 score = sum of all Part 1 individual item scores. Part 1 consists of 13 items on a scale of 0 (normal) to 4 (severe), so the Part 1 score ranges from 0 to 52. If an individual item is missing, it will be imputed as the average score for that part.
- MDS-UPDRS Part 2 score = sum of all Part 2 individual item scores. Part 2 consists of 13 items on a scale of 0 (normal) to 4 (severe), so the Part 2 score ranges from 0 to 52. If an individual item is missing, it will be imputed as the average score for that part.
- MDS-UPDRS Part 3 score = sum of all Part 3 individual item scores. Part 3 consists of 33 items on a scale of 0 (normal) to 4 (severe), so the Part 3 score ranges from 0 to 132. If an individual item is missing, it will be imputed as the average score for that part.
- MDS-UPDRS Parts 1-3 total score = sum of Part 1, Part 2, and Part 3 scores. If any of the
  individual part scores are missing, the total score will be set to missing.
- CISI-PD total score = sum of the four individual item scores (motor signs, disability, motor complications, and cognitive status) rated 0 (not at all) to 6 (very severe or disabled), with a range of 0 to 24.
- PDQ-39 Mobility subscore = sum of 10 items in the Mobility domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Activities of Daily Living subscore = sum of 6 items in the Activities of Daily Living domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Emotional Well-Being subscore = sum of 6 items in the Emotional Well-Being domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.



- PDQ-39 Stigma subscore = sum of 4 items in the Stigma domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Social Support subscore = sum of 3 items in the Social Support domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Cognitions subscore = sum of 4 items in the Cognitions domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Communication subscore = sum of 3 items in the Communication domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Bodily Discomfort subscore = sum of 3 items in the Bodily Discomfort domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.
- PDQ-39 Total score = mean of all of the PDQ-39 subscores.
- GDS-15 Total score = sum of the 15 item questionnaire, with a range of 0 to 15. Each question is answered "yes" or "no". Question numbers 1, 5, 7, 11, 13 indicate presence of depression when answered positively (yes) while the remaining questions indicate presence of depression when answered negatively (no). One point is counted for each depressive answer. A score of 0-4 indicates no depression, a score of 5-10 is suggestive of a mild depression, and a score of 11 or more is suggestive of severe depression.
- Modified Hachinski Ischemic Scale Total score = sum of the 8 item scores, with a range of 0-8.
- Change from baseline = value at current time point value at baseline.
- TEAE = any adverse event with an onset date/time after first dose of medication.
- Disease duration (years) = [Enrollment date PD onset date (as recorded on the Medical History case report form) + 1] / 365.25.

### 6.1.8. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

All P values will be displayed in four decimals and rounded using standard scientific notation (e.g., 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001.





Adverse events will be coded using the MedDRA version 21.0 thesaurus or higher.

A treatment related AE is any AE with a relationship to the study drug of possibly related or definitely related.

If partial AE or medication dates occur, the convention for replacing missing dates for the purpose of statistical analysis is as follows:

For partial AE and medication start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - If the year matches the year of first dose date and the end date (if present) is after first dose date, then impute as the month and day of the first dose date.
  - Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:
  - If the month and year match the month and year of the first dose date, then impute as the day of the first dose date.
  - o Otherwise, assign 01.

For partial AE and medication end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known, but the month or month and day is unknown, then:
  - If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
  - Otherwise, assign 31 December.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

If partial times occur, the convention is as follows:



- if the missing time occurs on the day of the first dose and both the hour and minute are
  missing then the time assigned is the time of the first dose, otherwise if both the hour and
  minute are missing and the date is not the date of first dose the time assigned is 12:00;
- · if the date is the same as the date of the first dose and
  - only hour is missing the hour assigned is 12 or the hour of first dose, whichever is later;
  - only the minute is missing the minute assigned is 30 or the minute of first dose, whichever is later;
- Otherwise if the date is not the same as the date of first dose, the hour assigned is 12 if the hour is missing and the minute assigned is 30 if the minute is missing.

# 7. Study Subjects and Demographics

# 7.1. Disposition of Subjects and Withdrawals

Disposition will include tabulations of the number of subjects randomized into each treatment group, the number of subjects who completed each series of infusions in Dosing Period 1 and Dosing Period 2, the number of subjects completing the study, tabulated reasons for discontinuation from the study, and number of subjects in each analysis dataset. The number of subjects completing each visit will also be presented, as will the number of subjects who did not complete the study per protocol due to COVID-19. A subject is considered to not have completed the study per protocol due to COVID-19 if they had any missing visits that affected treatment administration or collection of end of study efficacy assessments due to COVID-19. If a subject did not complete the study per protocol due to COVID-19, this category will supersede their study status on the study completion CRF page.

This summary will be based on the ITT Set.

### 7.2. Protocol Violations and Deviations

Protocol deviations will be listed.

### 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age, sex, race, ethnicity, height, weight, disease duration, and apolipoprotein E (ApoE) genotype will be presented by treatment group using summary statistics or frequencies, as appropriate. See Section 6.1.7 for derivation of disease duration.

The means of continuous demographic variables will be tested using Wilcoxon rank-sum test and the proportions of categorical demographic variables will be tested using a Chi-square test or Fisher's Exact test, as appropriate, in order to evaluate the effectiveness of the randomization in producing homogeneous pre-treatment groups.

These analyses will be conducted for the ITT Set.



The number and percent of subjects reporting various medical histories grouped by MedDRA system organ class and preferred term, will be tabulated. Medical histories of Parkinson's disease will also be presented by SOC, PT, and lower level term (LLT). Subject and family medical history as well as tobacco smoking, alcohol, and illicit substance use will be listed. Social history and exercise level will also be listed.

### 7.4. Exposure

All subjects will receive 5 consecutive days of therapy at the beginning of Weeks 1 and 13. Thus, the cumulative duration of therapy for all subjects will be 10 exposure days. The duration of therapy for a subject to be considered evaluable is 5 exposure days. Exposure days and volume administered will be summarized by treatment group and dosing period. The proportion of subjects who are considered evaluable over both dosing periods will also be displayed.

### 8. Efficacy Analysis

All secondary endpoints will be summarized using the Evaluable, Per Protocol, and Complete Sets. All efficacy data, regardless of population, will be presented in data listings.

# 8.1. Primary Efficacy Analysis

Not applicable. The primary analysis for this study is safety.

# 8.2. Secondary Efficacy Analysis

Normality assumptions will be tested using the Anderson-Darling method. If the P value for the normality test is >0.05 the data will be considered normally distributed and will be analyzed as specified in subsequent sections. Otherwise, if the P value is  $\leq$ 0.05 the data will be considered non-normal. If the data are non-normal, the Wilcoxon rank sum test will be used for comparisons between treatments and a non-parametric ANCOVA model will be run on the ranks. If the data is considered non-normal, the Wilcoxon signed rank test will be used to assess the within-subject changes.

### 8.2.1. Montreal Cognitive Assessment (MoCA)

The MoCA is a 1-page, 30-point test designed as a rapid screening instrument for mild cognitive dysfunction. The questionnaire assesses several different cognitive domains, including attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. Higher scores indicate better cognitive function; the total possible score is 30 and a score of 26 or more is considered normal. Derivation for the MoCA total score is described in Section 6.1.7.

The MoCA will be collected at Screening (Visit 1), Week 4 (Visit 9), and Week 16 (Visit 17).

Change from baseline to study visit in the MoCA total score and individual domains will be summarized by treatment group. Boxplots of the MoCA total score will also be provided by treatment group and visit. A test of hypothesis comparing mean total scores between baseline and subsequent study visits will be conducted using a 2-sided paired t-test or Wilcoxon signed



rank test, as appropriate. The null hypothesis is that the change from baseline to subsequent visit is 0.

Additionally, the mean change from baseline in MoCA total score will be compared between treatment groups using an ANCOVA model with treatment, visit, and treatment by visit interaction as a main effects and baseline MoCA total score, age, and ApoE genotype as covariates.

### 8.2.2. Cognitive Drug Research Computerized Cognition Battery (CDR-CCB)

The CDR-CCB assesses both enhancement and impairment of human cognitive function. In this study, the following will be measured using the CDR-CCB system: Continuity and Power of Attention, Working Memory, and Episodic Memory. Subjects will have two CDR-CCB training sessions during the screening period to ensure adequate performance at the Baseline Visit (Visit 2). CDR-CCB will also be assessed at Week 1 (Visit 8), Week 4 (Visit 9), Week 8 (Visit 10), Week 13 (Visit 16), Week 16 (Visit 17), Week 20 (Visit 18), and Week 24 (Visit 19).

Please refer to the separate SAP for the analysis of the CDR-CCB.

### 8.2.3. Delis-Kaplan Executive Function Verbal Fluency (D-KEFS)

The D-KEFS Verbal Fluency Test has three conditions: Letter Fluency, Category Fluency, and Category Switching. In the Letter Fluency condition, subjects are asked to say as many words that start with a particular letter (e.g., F, A, S) as possible over three trials of 60 seconds. The Category Fluency condition requires subjects to say as many words belonging to a particular semantic category (e.g., animals, tools) as they can in two trials of 60 seconds. In the final condition, subjects are asked to switch between words belonging to two different semantic categories in one trial of 60 seconds (e.g., fruits and furniture). D-KEFs is measured at Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 16), and Week 20 (Visit 18).

The number of correct F, A, and S responses from 1-15, 16-30, 31-46, and 46-60 seconds will be presented by treatment group and visit. Change from baseline in total score will be presented by treatment group. Derivation for the D-KEFS Total score is described in Section 6.1.7. Boxplots of the D-KEFSs total score will also be provided by treatment group and visit. A test of hypothesis comparing mean scores between baseline and subsequent study visits will be conducted using a 2-sided paired t-test or Wilcoxon signed rank test, as appropriate. The null hypothesis is that the mean change from baseline to subsequent visit is 0.

Mean change from Baseline will be compared between treatment groups using an ANCOVA model with treatment, visit, and treatment by visit interaction as a main effects and baseline score, age, and ApoE genotype as covariates.

### 8.2.4. Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

The MDS-UPDRS has four components (Part 1, Mentation, Behavior, and Mood; Part 2, Activities of Daily Living; Part 3, Motor; Part 4, Complications). Only Parts 1, 2, 3 and total score will be utilized for this study. Part 1 has 13 items that address mental dysfunction, mood,





and nonmotor aspects of experiences of daily living. Part 2 has 13 items that assess motor disability and aspects of experiences of daily living. Part 3 has 33 items that assess motor impairment and motor examination. The rating for each item is from 0 (normal) to 4 (severe) and the descriptions of each rating are provided in the table below.

| Scale for the MDS-UPDRS Rating | Description |
|---|---|
| 0 = normal | No symptoms/signs |
| 1 = slight | Symptoms/signs with sufficiently low frequency or intensity to cause no impact on function |
| 2 = mild | Symptoms/signs of frequency or intensity sufficient to cause a modest impact on function |
| 3 = moderate | Symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent, function |
| 4 = severe | Symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent, function |

The total score for each part is obtained from the sum of the corresponding item scores. Derivation for the MDS-UPDRS Total score is described in Section 6.1.7.

MDS-UPDRS is measured at Baseline (Visit 2), Week 1 (Visit 8), Week 4 (Visit 9), Week 8 (Visit 10), Week 13 (Visit 16), Week 16 (Visit 17), Week 20 (Visit 18), and Week 24 (Visit 19). Change from baseline to study visit in MDS-UPDRS scores will be summarized by treatment group. A test of hypothesis comparing mean scores between baseline and subsequent study visits will be conducted using a 2-sided paired t-test or Wilcoxon signed rank test, as appropriate. The null hypothesis is that the mean change from baseline to subsequent visit is 0.

Mean change from baseline in Total score will be compared between treatment groups using an ANCOVA model with treatment, visit, and treatment by visit interaction as a main effects and baseline score and age as covariates.

Boxplots of the MDS-UPDRS Part 3 score will also be provided by treatment group and visit.

# 8.2.5. Schwab and England Activities of Daily Living Scale (SE-ADL)

The SE-ADL evaluates patients' perceptions of global functional capacity and dependence. Scoring is expressed in terms of percentage, in 10 steps from 100 to 0 (100%, normal status; 0%, bedridden with vegetative dysfunction), so that the lower the score, the worse the functional status. The scoring is as follows:





| Scale for the SE-ADL Rating | Description |
|---|---|
| 100% | Completely independent. Able to do all chores without slowness, difficulty, or impairment. Essentially normal. Unaware of any difficulty. |
| 90% | Completely independent. Able to do all chores with some degree of slowness, difficulty and impairment. May take twice as long. Beginning to be aware of difficulty. |
| 80% | Completely independent in most chores. Takes twice as long. Conscious of difficulty and slowing. |
| 70% | Not completed independent. More difficulty with some chores. X3-4 as long in some. May spend a large part of the day with chores. |
| 60% | Some dependency. Can do most chores, but exceedingly slowly and with much effort. Errors; some impossible. |
| 50% | More dependent. Help with ½ of chores. Difficulty with everything. |
| 40% | Very dependent. Can assist with all chores but few alone. |
| 30% | With effort, now and then does a few chores alone or begins alone. Much help needed. |
| 20% | Nothing alone. Can do some slight help with some chores. Severe invalid. |
| 10% | Totally dependent, helpless. Complete invalid |
| 0% | Vegetative functions such as swallowing, bladder and bowel functions are not functioning. Bedridden. |

The SE-ADL is measured at Baseline (Visit 2), Week 8 (Visit 10), and Week 24 (Visit 19). The number and percentage of subjects falling in each category at each time point will be displayed by treatment group. A 2-sided Cochran-Mantel-Haenszel (CMH) test will be performed at the 5% significance level to determine whether there is a significant relationship between treatment group and level of independence.



# 8.2.6. Clinical Impression of Severity Index – Parkinson's Disease (CISI-PD)

The CISI-PD is a severity index formed by four items (motor signs, disability, motor complications, and cognitive status), rated 0 (not at all) to 6 (very severe or completely disabled). CISI-PD is measured at Baseline (Visit 2), Week 8 (Visit 10), and Week 24 (Visit 19). Change from baseline to study visit in each item will be summarized by treatment group. A test of hypothesis comparing mean scores between baseline and subsequent study visits will be conducted using a 2-sided paired t-test or Wilcoxon signed rank test, as appropriate. The null hypothesis is that the mean change from baseline to subsequent visit is 0.

Mean change from baseline in Total score will be compared between treatment groups using an ANCOVA model with treatment, visit, and treatment by visit interaction as a main effects and baseline score, age, and ApoE genotype as covariates.

# 8.2.7. Parkinson's Disease Quality of Life Questionnaire-39 (PDO-39)

The long form of the PDQ has 39 questions, with eight dimensions:

- Mobility (10 items)
- Activities of daily living (6 items)
- Emotional well-being (6 items)
- Stigma (4 items)
- Social support (3 items)
- Cognitions (4 items)
- Communication (3 items)
- Bodily discomfort (3 items)

The frequency of each event is recorded as one of five options, with each option assigned a numeric value as indicated: never (0), occasionally (1), sometimes (2), often (3), or always/cannot do at all (4). It is scored on a scale of 0-100 with lower scores indicating better health and high scores indicating more severe symptoms. Derivations for each of the subscores and total score are described in Section 6.1.7.

The PDQ-39 will be collected at Baseline (Visit 2), Week 4 (Visit 9), Week 8 (Visit 10), Week 20 (Visit 18), and Week 24 (Visit 19).

Change from baseline to study visit in the PDQ-39 Mobility, Activities of Daily Living, Emotional Well-Being, Stigma, Social Support, Cognitions, Communication, and Bodily Discomfort subscores and PDQ-39 Total score will be summarized by treatment group. A test of hypothesis comparing mean scores between baseline and subsequent study visits will be conducted using a 2-sided paired t-test or Wilcoxon signed rank test, as appropriate. The null hypothesis is that the mean change from baseline to subsequent visit is 0.

Mean change from baseline in Total score will be compared between treatment groups using an ANCOVA model with treatment, visit, and treatment by visit interaction as a main effects and baseline score, age, and ApoE genotype as covariates.



### 8.2.8. Geriatric Depression Scale-15 (GDS-15)

The GDS-15 is a shortened form of a 30-item questionnaire in which participants are asked to respond by answering yes or no in reference to how they felt over the past week. Of the 15 items, 10 indicate the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicate depression when answered negatively. Each item is recorded as yes or no which is assigned a numeric value of 1 or 0, respectively. The final score is the tally of the number of depressive answers with the following scores indicating depression:

- 0-4 No depression
- 5-10 Suggestive of a mild depression
- 11 + Suggestive of severe depression

Derivations for the final score is described in Section 6.1.7. The GDS-15 will be collected at Baseline (Visit 2), Week 8, (Visit 10) and Week 20 (Visit 18). The number and percentages of subject responses will be summarized by treatment group and visit. Change from baseline to study visit in GDS-15 total score will be summarized by treatment group.

### 8.2.9. Digital Clock Drawing Test (dCDT)

The pen-like dCDT device gathers the x-y coordinates that describe the movement of the stylus as it changes its position during the assessment. It also assesses when the stylus or writing device is not exerting pressure on the writing surface (i.e., in-air movements performed by the hand while transitioning from one stroke to the next).

The dCDT will be collected at Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 16), and Week 20 (Visit 18).

The dCDT score is a number from 0 and 100 that represents a person's overall cognitive function as assessed by DCTclock. The score will be classified as within normal limits, indeterminate, outside normal limits, or unanalyzable based on cut scores and test performance.

Change from baseline to study visit in dCDT score will be summarized by treatment group. A test of hypothesis comparing mean scores between baseline and subsequent study visits will be conducted using a 2-sided paired t-test or Wilcoxon signed rank test, as appropriate. The null hypothesis is that the mean change from baseline to subsequent visit is 0.

Mean change from baseline in dCDT score will be compared between treatment groups using an ANCOVA model with treatment, visit, and treatment by visit interaction as a main effects and baseline score, age, and ApoE genotype as covariates.

The number and percentage of subjects falling in each classification at each time point will be displayed by treatment group.

The cognitive features within the drawing efficiency, simple motor, information processing, and spatial reasoning composite scales will be listed.





### 8.3. **Exploratory Efficacy Analysis**

### Apolipoprotein E (ApoE) Genotype Testing 8.3.1.

DNA for ApoE analysis will be obtained from a blood serum sample collected at Visit 3 to determine ApoE genotype at baseline. ApoE genotype will be listed and summarized as part of demographics and baseline characteristics. See Section 7.3. The number and proportion of subjects with the genotype for each allele will be presented.

### 8.3.2. Magnetic Resonance Imaging (MRI)

MRI will be used to evaluate subjects' eligibility for inclusion in the study at screening. Structural images will be interpreted by a central reader at screening and any exclusionary findings will be reported. Where available, functional imaging will also be acquired to assess for functional connectivity as measured by tf-fMRI and cerebral blood flow as measured by ASL MRI. In consenting subjects, an additional MRI at Visit 16 will assess for changes in brain atrophy as measured by MRI, functional connectivity as measured by tf-fMRI, and cerebral blood flow as measured ASL MRI. During the MRI, the subject will be asked to lie on a narrow bed in a large tunnel while images are captured by the MRI machine. Participation in the screening MRI is required, while participation in the additional MRI at Visit 16 is optional and not required for inclusion in the study.

### 8.3.2.1. Safety MRI

The number and percentage of subjects with presence of screening safety MRI abnormalities along with the type of abnormality and primary location of abnormality reported will be presented by treatment group. Additionally, abnormality sequence, abnormality status, and presence of white matter disease will be tabulated by treatment group. The number and percentage of subjects whose screening safety MRI findings suggest there is a potential alternative diagnosis to PD will also be presented.

Screening safety MRI results will be listed.

### 8.3.2.2. Volumetric MRI

Volume will be summarized using descriptive statistics for the left, right, and bilateral sides of the following locations:

- Whole brain (bilateral only)
- Lateral ventricles (bilateral only)
- Intracranial (bilateral only)
- Cortical
- Hippocampus

Cerebral cortex average thickness will be summarized using descriptive statistics for the left, right, and bilateral sides of the following locations:

Cortical

premier

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

- Mayo (bilateral only)
- Prefrontal lobe
- Whole temporal lobe
- Superior temporal lobe
- Medial temporal lobe
- Lateral parietal lobe
- · Inferior parietal lobe
- Precuneus
- Isthmus-cingulate
- Entorhinal cortex

Atrophy absolute change and cerebral cortex thickness average change will be summarized using descriptive statistics for the left, right, and bilateral sides of the following locations at follow-up:

- Whole brain (bilateral only)
- · Lateral ventricles (bilateral only)
- Cortical
- Hippocampus

Additionally, cerebral cortex thickness average change will be summarized using descriptive statistics for the left, right, and bilateral sides of the following locations at follow-up:

- Cortical
- Hippocampus
- · Mayo (bilateral only)
- Prefrontal lobe
- Whole temporal lobe
- Superior temporal lobe
- Medial temporal lobe
- Lateral parietal lobe
- Inferior parietal lobe
- Precuneus
- · Isthmus-cingulate
- Entorhinal cortex

Volumetric MRI results will also be listed.

### 8.3.2.3. Resting fMRI

Since there are 85 correlations between regions, fMRI data will not be summarized or listed due to file size. If summaries or listings are desired, they will be provided on an ad hoc basis.

### 8.3.2.4. ASL MRI

Cerebral blood flow measurements will be summarized using descriptive statistics for the left, right, and bilateral sides of the following locations:

Frontal lobe



- Cingulate cortex
- Parietal lobe
- Temporal lobe
- Occipital lobe
- Striatum
- Cerebellum
- Thalamus
- Pallidum
- Substantia nigra
- Hippocampus

ASL MRI results will also be listed.

# 9. Safety and Tolerability Analysis

The primary endpoint of this study is the incidence of TEAEs and SAEs identified by MedDRA PT and grouped by MedDRA SOC.

The secondary safety endpoints are as follows:

- Change from baseline in clinical laboratory parameters
- Change from baseline in vital sign measurements
- · Change from baseline in body weight
- Change from baseline in the S-STS

Safety will also be evaluated from electrocardiogram (ECG) results and physical examination results.

All safety analyses will be performed on the Safety Set.

### 9.1. Adverse Events

All AEs that occur after the time of treatment with the study agent will be considered TEAEs. Events meeting this definition will be those events that are a change from the subject's baseline conditions, including an increase in frequency or severity (these will be entered as new AEs). For AEs occurring on the date of first dose, if the time of onset is missing, the AE will be assumed to be treatment emergent.

All AEs, TEAEs, and SAEs will be coded using the MedDRA Version 20.1 or higher coding dictionary. The AE analyses will focus on those that are treatment emergent, however any AEs that are reported after consent has been signed and before initial dosing will be considered intercurrent events and flagged in the listings as such.

The causal relationship of the AE to the study drug is determined by the investigator as Unrelated, Possibly Related, or Definitely Related. These can be mapped to Unrelated (*Unrelated*) and Related (*Possibly Related* and *Definitely Related*). Adverse event summaries will be repeated for treatment related TEAEs.


Adverse events severity grades are reported as mild, moderate, or severe.

Summaries of incidence rates (frequencies and percentages) of individual TEAEs will be presented by SOC, PT, and treatment group. Such summaries will be displayed for all TEAEs, TEAEs by maximum severity, and TEAEs by relationship.

Each subject will be counted only once within each summation level (SOC and PT). If a subject experiences more than 1 TEAE within each summation level only, the TEAE with the strongest relationship or the maximum severity, as appropriate, will be included in the summaries of relationship and severity. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = definitely related).

Incidences will be presented by descending frequency of SOC and PT within SOC, and then alphabetically within PT where the incidence is the same; this is based on overall subjects then alphabetically in case of a tie.

Missing and partially missing AE start and/or stop dates will be imputed, for the purpose of statistical analysis, according to the specifications described in Section 6.1.8.

In the AE data listings, all AEs will be displayed. AEs that are treatment emergent will be flagged.

A test of hypothesis comparing the proportion of subjects reporting a TEAE throughout the study will be conducted using a Chi-square test or Fisher's exact test, as appropriate. The null hypothesis is that there is no difference in proportion between treatment groups, with a two-sided alternative that considers the possibility of a difference in either direction. The number and percentage of subjects reporting a TEAE and the 95% Wilson confidence interval (CI) for the proportion will be presented for each treatment group. In addition, the difference in proportions between the GRF6021 and placebo groups and the 95% Wilson CI will be presented. The same statistics and hypothesis testing will be performed for subjects reporting an SAE throughout the study.

### 9.1.1. Adverse Events Leading to Withdrawal

A derived action taken variable will be created for subjects who withdrew from the study or study drug due to an AE as noted on the study completion (DS) CRF. If the reason for discontinuation entered on the DS CRF was "Adverse Event" and the AE occurred between the start of the first infusion in Period 1 through the final infusion in Period 2, the derived action taken will be set to "study drug withdrawn" regardless of what action taken was entered on the AE CRF. Since treatment is administered during two distinct periods and not on a continuous basis, if an AE that causes withdrawal occurs between the two infusion periods, action taken may not accurately indicate "study drug withdrawn" unless it was decided that subject would not get a second infusion since the subject will not actively be receiving treatment between the two periods.

A summary of incidence rates (frequencies and percentages) of TEAEs leading to withdrawal of study drug, by treatment group, SOC, and PT will be prepared for the Safety Dataset. No inferential statistical tests will be performed. These summaries will be based on the derived action taken.



A data listing of AEs leading to withdrawal of study drug will be provided, displaying details of the event(s) captured on the CRF. Both derived and CRF action taken variables will be presented in the listing.

### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.

Serious adverse events will be listed and tabulated by SOC, PT, and treatment group.

### 9.1.3. Other Significant Adverse Events

AEs of special interest (AESI) are defined in the protocol. These are to be considered as Adverse Events by the PI in order to be recorded:

A summary tabulating these criteria for safety will be presented by SOC, PT, and treatment group. All AESIs will be flagged in the AE listings.

Adverse events with preferred terms associated with blood pressure changes will also be presented by infusion period, SOC, PT, and treatment group. Infusion period will be further categorized by whether the event start date occurred during the infusion period or after the infusion period. Examples of such events can be identified by the following preferred terms: blood pressure decreased, blood pressure diastolic decreased, blood pressure systolic decreased, blood pressure increased, increased blood pressure, blood pressure diastolic increased, blood pressure systolic increased, hypotension, hypertension, low blood pressure, high blood pressure. This is a non-exhaustive list and a review of AE MedDRA coding will be conducted prior to lock to identify all events associated with blood pressure changes.

### 9.2. Laboratory Evaluations

The screening safety lab panel includes: all comprehensive labs (hematology, chemistry, coagulation, urinalysis, urine chemistry, ionized calcium), immunochemistry (HIV, hepatitis B, hepatitis C, thyroid-stimulating hormone (TSH), brain natriuretic peptide (BNP)), cobalamin (vitamin B12), pyridoxine (vitamin B6), thiamine (vitamin B1), direct antiglobulin test, IgA, haptoglobin, and C1 inhibitor. The urine drug screen includes cannabinoids, benzodiazepine, barbiturates, opiates, cocaine, amphetamines, methadone, phencyclidine, and propoxyphene.

Pre-infusion safety labs will be performed onsite and should be collected and results interpreted prior to the following day's infusion start. The following should be measured at Visit 3, Visit 4, Visit 6, Visit 11, Visit 12, and Visit 14: sodium (Na), potassium (K), ionized calcium, urea nitrogen (BUN)/urea, creatinine (Crea), hematocrit, hemoglobin, platelets. These results are only available at each site and will therefore not be summarized.

The exit safety lab panel includes all comprehensive labs, immunochemistry, direct antiglobulin test, and ionized calcium.



Comprehensive labs will be performed at screening/Visit 1, Visit 6, Visit 8, Visit 9, Visit 14, Visit 16, Visit 17, and upon exit/Visit 19.

Laboratory test results, excluding the site's pre-infusion safety labs mentioned above, will be summarized descriptively by treatment and visit as both observed values and change from baseline values for each parameter. Categorical urinalysis results will be summarized using frequencies by treatment group and visit.

Shifts from baseline for clinical laboratory values below, within, or above the normal range will be provided for hematology, chemistry, coagulation, and quantitaive urinalysis results by visit and treatment. See Section 6.1.1 for the definition of baseline.

Subjects with significant laboratory abnormalities will be identified in data listings. If any laboratory tests are collected at an unscheduled visit post-baseline, the results will be included in listings.

Pregnancy test results from Screening (Visit 1), Visit 3, and Visit 11 will be listed.

### 9.3. Vital Signs

Descriptive summaries of actual values and changes from baseline will be calculated for seated systolic blood pressure, standing systolic blood pressure, and supine systolic blood pressure, seated diastolic blood pressure, standing diastolic blood pressure, and supine diastolic blood pressure, heart rate, respiration rate, and body temperature. These summaries will be presented by visit and treatment group. Vital signs are collected at all study visits. During the infusion periods (Visit 3-Visit 7 and Visit 11- Visit 15), orthostatic vital signs (supine systolic and supine diastolic blood pressure compared to standing systolic and standing diastolic blood pressure) should be measured prior to infusion start and at approximately after infusion start. Seated systolic and seated diastolic blood pressure is measured at multiple timepoints during and after each infusion. Abnormal vital sign values will be flagged in the listings. Abnormal vital sign values are as follows:

- Seated systolic blood pressure value < 90 mmHg</li>
- Seated systolic blood pressure value > 180 mmHg
- Seated diastolic blood pressure value < 50 mmHg</li>
- Seated diastolic blood pressure value > 110 mmHg
- Incidence of orthostatic hypotension (a decrease in systolic blood pressure of > 20 mm Hg and/or a decrease in diastolic blood pressure of > 10 mm Hg between supine and standing)
- Heart rate > 100 beats per minute
- Temperature > 37.5°C
- Temperature < 36.5°C</li>
- Respiration rate > 20 breaths per minute
- Respiration rate < 12 breaths per minute</li>



The vital sign measurements that meet the criteria for blood pressures of special interest (listed below) will also be identified from the vital signs source data and summarized separately by study visit, timepoint, and treatment.

- Seated systolic blood pressure >180 mmHg
- Seated systolic blood pressure > 200 mmHg
- Seated systolic blood pressure < 90 mmHg</li>
- Seated diastolic blood pressure > 110 mmHg
- Seated diastolic blood pressure > 120 mmHg
- Seated diastolic blood pressure < 50 mmHg</li>
- A change of ≥ 30% from baseline in seated systolic and/or seated diastolic blood pressure

### 9.4. Electrocardiograms (ECGs)

12-Lead Electrocardiograms will be obtained at Screening, Week 1 (Visit 7) and Week 13 (Visits 11 and 15).

Descriptive summaries will be presented for ECG measures of QT interval, QTc interval, and HR. Corrected QTc intervals will be calculated using Fridericia's correction formula. These summaries will be presented by treatment group and visit.

The number and percentage of subjects with normal, abnormal but not clinically significant, and abnormal and clinically significant ECG results will be summarized for the Safety Dataset by treatment group and visit.

### 9.5. Further Safety Evaluations

### 9.5.1. Physical Examination

A full physical examination will be performed to assess the following organ systems: skin; ears, nose, and throat (ENT); head; eyes; lungs/chest; heart; abdomen; musculoskeletal; extremities; neurologic system; and lymphatic system. The neurological exam will include cranial nerves (visual fields, fundoscopic exam, pupillary light reflex, extraocular muscles, facial sensation and symmetry, palate and tongue, and head turning and shoulder shrug); muscle strength, tone, and bulk; reflexes (biceps, triceps, knees, ankles, and plantar); coordination (finger-to-nose, heel-knee-shin); sensory function (light touch and pinprick); and gait. Height will be measured at screening and weight will be monitored during the trial.

While the subject is inpatient, a targeted physical exam, including auscultation of the heart and lungs, an assessment of peripheral edema, and weight, will be performed per the study schedule.

All physical exam results will be listed.

### 9.5.2. Sheehan-Suicidality Tracking Scale (S-STS)

The S-STS is a 16-item scale that assesses the seriousness of suicidality phenomena on a Likert-type scale (0-4) ranging from "not at all" (0) to "extremely" (4). It also assesses the frequency of key phenomena and the overall time spent in suicidality. This study is only collecting the total



scale score. S-STS total scores will be summarized descriptively by treatment and visit as both observed values and change from baseline values.

### 9.6. Concomitant Medication

Prior and concomitant medications, coded using World Health Organization drug dictionary (WHO-DDE) (March 2018), will be summarized descriptively by Anatomical Therapeutic Chemical (ATC) classification Level 4 and PT (i.e., ATC classification Level 5), if applicable, and by treatment group using counts and percentages. Additionally, the number of subjects with prior medications for PD and cognition will be presented by treatment group. Medications for PD will be identified from the indication field on the CRF as well as those in ATC Classes N04, N04A, and N04B. Medications for cognition will be identified by ATC Class N06D and N06DX. A review of prior and concomitant medications along with their indications will be performed prior to database lock.

Prior medications will be presented separately from concomitant medications. The assignment of medications as prior and/or concomitant will be done as follows:

- Prior medications: Medications that started before first dose will be considered prior medications whether or not they were stopped before dose.
- Concomitant medications: Any medications continuing or starting after the first dose through the end of study will be considered to be concomitant.

If a medication starts prior to the first dose and continues after the first dose it will be considered both prior and concomitant. Prior and concomitant medications will also be listed.

### 10. Changes from Planned Analysis

The protocol will be amended such that blood pressure values, in conjunction with signs and symptoms of hypo/hypertension, will be at the discretion of the PI as to whether or not they constitute an AESI. As such, ranges for blood pressures of special interest (BPSI) were identified and will be used for consideration in determining whether events are BPSIs going forward. Separate summaries of these measurements will be presented. See Section 9.3.

### 11. Other Planned Analysis

### 11.1. Hoehn and Yahr Scale

The Hoehn and Yahr Scale is used to describe the symptom progression of PD. The scale is as follows:

| Stage | Description |
|---|---|
| 0 | No signs of disease |
| 1.0 | Symptoms are very mild; unilateral involvement only |
| 2 Bilateral involvement without impairment of balance | |



| Stage | Description |
|---|---|
| 3 | Mild to moderate involvement; some postural instability but physically independent; needs assistance to recover from pull test |
| 4 | Severe disability; still able to walk or stand unassisted |
| 5 Wheelchair bound or bedridden unless aided | |

The Hoehn and Yahr Scale will be assessed at Screening (Visit 1) only and will be listed.

### Modified Hachinski Ischemic Scale (MHIS)

The MHIS is an 8-item scale that examines clinical features that may be consistent with vascular dementia and is commonly used as a screening tool to exclude patients with multi-infarct dementia. Scores for the 8 items are added together for a total score. Subjects who score 5 or greater are more likely to have a dementia of vascular etiology and thus are excluded from participating in this trial.

The MHIS will be assessed at Screening (Visit 1) only and the presence of the clinical features will be listed.

### 11.3. Echocardiogram

During Screening (Visit 1), an echocardiogram will be performed to evaluate the subject's left ventricular (LV) systolic function to ensure the subject's ejection fraction percentage is ≥ 55%. Echocardiogram results will be listed.

### 12. References

- 1. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.

### 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (listing number).



### 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number ALK6021-201. The table numbers and page numbers are place holders only and will be determined when the tables are produced.



### Table 2: Demographic Data Summary Tables and Figures

| Number | Set | Title | Safety IA | Efficacy IA |
|---|---|---|---|---|
| Table 14.1.1 | ITT | Summary of Subject Disposition | Х | х |
| Table 14.1.2.1 | ITT | Demographics and Baseline Characteristics | х | х |
| Table 14.1.3.1 | Safety | Summary of Medical History by SOC, PT, and Treatment | | |
| Table 14.1.3.2 | Safety | Summary of Parkinson's Disease Medical History by SOC, PT, LLT, and Treatment | | |
| Table 14.1.4 | Safety | Summary of Prior Medications by ATC Class Level 4, PT, and Treatment | | |
| Table 14.1.5 | Safety | Summary of Exposure by Treatment | x | X |

### 13.2. Efficacy Data Tabulations

Table 3: Efficacy Data

| Number | Set | Title | Include in Interim<br>Efficacy Analysis? |
|---|---|---|---|
| Table<br>14.2.1.1 | Evaluable | Summary of Change from Baseline in MoCA Scores by Treatment | х |
| Table<br>14.2.1.2 | Evaluable | Mean Change from Baseline in MoCA Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table 14.2.1.3 | Per<br>Protocol | Summary of Change from Baseline in MoCA Scores by Treatment | х |
| Table<br>14.2.1.4 | Per<br>Protocol | Mean Change from Baseline in MoCA Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.1.5 | Complete | Summary of Change from Baseline in MoCA Scores by Treatment | |
| Table<br>14.2.1.6 | Complete | Mean Change from Baseline in MoCA Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.2.1 | Evaluable | Summary of Change from Baseline in D-KEFS Total Score by Treatment | |
| Table<br>14.2.2.2 | Evaluable | Mean Change from Baseline in D-KEFS Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table 14.2.2.3 | Per<br>Protocol | Summary of Change from Baseline in D-KEFS Total Score by<br>Treatment | |



| Number | Set | Title | Include in Interim<br>Efficacy Analysis? |
|---|---|---|---|
| Table<br>14.2.2.4 | Per<br>Protocol | Mean Change from Baseline in D-KEFS Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.2.5 | Complete | Summary of Change from Baseline in D-KEFS Total Score by Treatment | |
| Table<br>14.2.2.6 | Complete | Mean Change from Baseline in D-KEFS Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table 14.2,3.1 | Evaluable | Summary of Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Scores by Treatment | х |
| Table<br>14.2.3.2 | Evaluable | Mean Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.3.3 | Per<br>Protocol | Summary of Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Scores by Treatment | х |
| Table 14.2.3.4 | Per<br>Protocol | Mean Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table 14.2.3.5 | Complete | Summary of Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Scores by Treatment | |
| Table<br>14.2.3.6 | Complete | Mean Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and<br>Parts 1-3 Total Score by Study Visit and Treatment, Tabulation of<br>Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.4.1 | Evaluable | Summary of SE-ADL by Study Visit and Treatment | |
| Table<br>14.2.4.2 | Per<br>Protocol | Summary of SE-ADL by Study Visit and Treatment | |
| Table<br>14.2.4.3 | Complete | Summary of SE-ADL by Study Visit and Treatment | |
| Table<br>14.2.5.1 | Evaluable | Summary of Change from Baseline in CISI-PD Scores by Treatment | |
| Table<br>14.2.5.2 | Evaluable | Mean Change from Baseline in CISI-PD Total Score by Study Visit<br>and Treatment, Tabulation of Fitted Summary Statistics from<br>ANCOVA | |
| Table<br>14.2.5.3 | Per<br>Protocol | Summary of Change from Baseline in CISI-PD Scores by Treatment | |
| Table<br>14.2.5.4 | Per<br>Protocol | Mean Change from Baseline in CISI-PD Total Score by Study Visit<br>and Treatment, Tabulation of Fitted Summary Statistics from<br>ANCOVA | |



| Number | Set | Title | Include in Interim<br>Efficacy Analysis? |
|---|---|---|---|
| Table 14.2.5.5 | Complete | Summary of Change from Baseline in CISI-PD Scores by Treatment | |
| Table<br>14.2.5.6 | Complete | Mean Change from Baseline in CISI-PD Total Score by Study Visit<br>and Treatment, Tabulation of Fitted Summary Statistics from<br>ANCOVA | |
| Table<br>14.2.6.1 | Evaluable | Summary of Change from Baseline in PDQ-39 Scores by Treatment | |
| Table<br>14.2.6.2 | Evaluable | Mean Change from Baseline in PDQ-39 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.6.3 | Per<br>Protocol | Summary of Change from Baseline in PDQ-39 Scores by Treatment | |
| Table<br>14.2.6.4 | Per<br>Protocol | Mean Change from Baseline in PDQ-39 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.6.5 | Complete | Summary of Change from Baseline in PDQ-39 Scores by Treatment | |
| Table<br>14.2.6.6 | Complete | Mean Change from Baseline in PDQ-39 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.7.1 | Evaluable | Summary of GDS-15 Categories by Study Visit and Treatment | |
| Table<br>14.2.7.2 | Evaluable | Summary of Change from Baseline in GDS-15 Score by Treatment | |
| Table<br>14.2.7.3 | Evaluable | Mean Change from Baseline in GDS-15 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.7.4 | Per<br>Protocol | Summary of GDS-15 Categories by Study Visit and Treatment | |
| Table<br>14.2.7.5 | Per<br>Protocol | Summary of Change from Baseline in GDS-15 Score by Treatment | |
| Table<br>14.2.7.6 | Per<br>Protocol | Mean Change from Baseline in GDS-15 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.7.7 | Complete | Summary of GDS-15 Categories by Study Visit and Treatment | |
| Table<br>14.2.7.8 | Complete | Summary of Change from Baseline in GDS-15 Score by Treatment | |



| Number | Set | Title | Include in Interim<br>Efficacy Analysis? |
|---|---|---|---|
| Table<br>14.2.7.9 | Complete | Mean Change from Baseline in GDS-15 Total Score by Study Visit and Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.8.1 | Evaluable | Summary of Change from Baseline in dCDT Score by Treatment | |
| Table<br>14.2.8.2 | Evaluable | Mean Change from Baseline in dCDT Score by Study Visit and<br>Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.8.3 | Per<br>Protocol | Summary of Change from Baseline in dCDT Score by Treatment | |
| Table<br>14.2,8,4 | Per<br>Protocol | Mean Change from Baseline in dCDT Score by Study Visit and<br>Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.8.5 | Complete | Summary of Change from Baseline in dCDT Score by Treatment | |
| Table<br>14.2.8.6 | Complete | Mean Change from Baseline in dCDT Score by Study Visit and<br>Treatment, Tabulation of Fitted Summary Statistics from ANCOVA | |
| Table<br>14.2.8.7 | Evaluable | Summary of dCDT Classification by Study Visit and Treatment | |
| Table<br>14.2.8.8 | Per<br>Protocol | Summary of dCDT Classification by Study Visit and Treatment | |
| Table<br>14.2.8.9 | Complete | Summary of dCDT Classification by Study Visit and Treatment | |
| Table<br>14.2.9.1 | Evaluable | Summary of Screening Safety MRI Results by Treatment | |
| Table<br>14.2.9.2 | Per<br>Protocol | Summary of Screening Safety MRI Results by Treatment | |
| Table<br>14.2.9.3 | Evaluable | Summary of Volumetric MRI Results by Treatment | |
| Table<br>14.2.9.4 | Evaluable | Summary of ASL MRI Results by Treatment | |





### 13.3. Safety Data

Table 4: Safety Data

| Number | Set | Title | Include in<br>Interim Safety<br>Analysis? | Include in<br>Interim<br>Efficacy<br>Analysis? |
|---|---|---|---|---|
| 14.3.1 Di | splays o | f Adverse Events | Kanada ara | |
| Table<br>14.3.1.1 | Safety | Summary of Adverse Events by Treatment | x | х |
| Table<br>14.3.1.2 | Safety | Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment | х | х |
| Table<br>14.3.1.3 | Safety | Incidence of Treatment Emergent Adverse Events by<br>Maximum Severity, SOC, PT, and Treatment | Х | |
| Table<br>14.3,1.4 | Safety | Incidence of Treatment Emergent Adverse Events by<br>Relationship, SOC, PT, and Treatment | X | |
| | 4.3.2 St | ummary of Deaths, Other Serious and Significant Adverse | Events | |
| Table<br>14.3.2.1 | Safety | Incidence of Adverse Events Leading to Withdrawal by SOC, PT, and Treatment | х | х |
| Table<br>14,3,2,2 | Safety | Incidence of Serious Adverse Events by SOC, PT, and X Treatment | | Х |
| Table<br>14.3.2.3 | Safety | Incidence of Adverse Events of Special Interest by SOC, PT, and Treatment | x | х |
| Table<br>14.3.2.4 | Safety | Incidence of Adverse Events with Terms Associated with<br>Blood Pressure Changes by Infusion Period, SOC, PT, and<br>Treatment | х | х |
| 14.3.3 N | arrative | s of Deaths, Other Serious and Certain Other Significant | Adverse Events | |
| Table<br>14.3.3.1 | Safety | Listing of Adverse Events Leading to Study Drug<br>Discontinuation | | |
| Table<br>14.3.3.2 | Safety | Listing of Serious Adverse Events | | |
| Table<br>14.3.3.3 | Safety | Listing of Deaths | | |
| Table<br>14.3,3.4 | Safety | Listing of Adverse Events of Special Interest | | |
| 14.3.4 Ab | normal | Laboratory Value | | |
| NA | | | | |
| 14.3.5 Lal | boratory | y Data Summary Tables | | |



| Number | Set | Title | Include in<br>Interim Safety<br>Analysis? | Include in<br>Interim<br>Efficacy<br>Analysis? |
|---|---|---|---|---|
| Table 14.3.5.1.1 | Safety | Summary of Hematology Laboratory Results by Study<br>Visit and Treatment | х | |
| Table<br>14.3.5.1.2 | Safety | Shift from Baseline in Hematology Laboratory Results by<br>Study Visit and Treatment | х | |
| Table<br>14.3.5.2.1 | Safety | Summary of Serum Chemistry Laboratory Results by<br>Study Visit and Treatment | х | |
| Table<br>14.3.5.2.2 | Safety | Shift from Baseline in Serum Chemistry Laboratory<br>Results by Study Visit and Treatment | х | |
| Table<br>14.3.5.3.1 | Safety | Summary of Quantitative Urinalysis Laboratory Results by Study Visit and Treatment | х | |
| Table<br>14.3.5.3.2 | Safety | Shift from Baseline in Quantitative Urinalysis Laboratory<br>Results by Study Visit and Treatment | х | |
| Table<br>14.3.5.3.3 | Safety | Summary of Qualitative Urinalysis Laboratory Results by Study Visit and Treatment | х | |
| Table<br>14.3.5.4.1 | Safety | Summary of Coagulation Laboratory Results by Study<br>Visit and Treatment | х | |
| Table<br>14.3.5.4.2 | Safety | Shift from Baseline in Coagulation Laboratory Results by<br>Study Visit and Treatment | x | |
| 14.3.6 Otl | er Safe | ty Data Summary Tables | | |
| Table<br>14.3.6.1.1 | Safety | Summary of Vital Signs by Study Visit and Treatment | Х | |
| Table<br>14.3.6.1.2 | Safety | Summary of Blood Pressures of Special Interest by Study<br>Visit and Treatment | Х | |
| Table<br>14.3.6.2.1 | Safety | Summary of 12-Lead Electrocardiogram by Study Visit and Treatment | | |
| Table<br>14.3.6.2.2 | Safety | Summary of 12-Lead Electrocardiogram Interpretation by<br>Study Visit and Treatment | | |
| Table<br>14.3.6.3 | Safety | Summary of Sheehan-Suicidality Tracking Scale (S-STS) by Study Visit and Treatment | х | |
| Гаblе<br>14.3.6.4 | Safety | Summary of Concomitant Medications by ATC Class<br>Level 4, PT, and Treatment | | |



### 13.4. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number ALK6021-201.

In general, one listing will be produced per CRF domain. All listings will be sorted by treatment, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

Table 5: Planned Listings

| Number | Dataset | Title / Summary |
|---|---|---|
| 16.2.1 Subject Disc | ontinuations/Com | pletions |
| Listing 16.2.1 | All Subjects | Subjects Subject Disposition |
| 16.2.2 Protocol Dev | viations | No. 10 To 10 |
| Listing 16.2.2.1 | All Subjects | Inclusion and Exclusion Criteria Not Met |
| Listing 16.2.2.2 | All Subjects | Protocol Deviations |
| 16.2.3 Subjects Exc | cluded from the E | fficacy Analyses |
| Listing 16.2.3 | All Subjects | Analysis Sets |
| 16.2.4 Demographi | c Data and Other | Baseline Characteristics |
| Listing 16.2.4.1 | All Subjects | Demographics and Baseline Characteristics |
| Listing 16.2.4.2.1 | All Subjects | Medical History |
| Listing 16.2.4.2.2 | All Subjects | Family Medical History |
| Listing 16.2.4.2.3 | All Subjects | Social History and Exercise/Activity Level |
| Listing 16.2.4.3 | All Subjects | Alcohol, Tobacco, and Substance Use |
| Listing 16.2.4.4 | All Subjects | Modified Hachinski Ischaemia Scale (MHIS) |
| Listing 16.2.4.5 | All Subjects | Hoehn and Yahr Scale |
| 16.2.5 Compliance | and/or Drug Cond | centration Data |
| Listing 16.2.5 | All Subjects | Drug Infusion |
| 16.2.6 Individual E | fficacy Response | Data |
| Listing 16.2.6.1 | All Subjects | MoCA |
| Listing 16.2.6.2 | All Subjects | D-KEFS Verbal Fluency Test |
| Listing 16.2.6.3 | All Subjects | MDS-UPDRS |
| Listing 16,2.6,4 | All Subjects | SE-ADL Scale |





| Number | Dataset | Title / Summary |
|---|---|---|
| Listing 16.2.6.5 | All Subjects | CISI-PD |
| Listing 16.2.6.6 | All Subjects | PDQ-39 |
| Listing 16.2.6.7 | All Subjects | GDS-15 |
| Listing 16.2.6.8 | All Subjects | dCDT |
| Listing 16.2.6.9 | All Subjects | Patient Questionnaire Status |
| Listing 16.2.6.10 | All Subjects | Safety MRI Results |
| Listing 16.2.6.11 | All Subjects | Volumetric MRI Results |
| Listing 16.2.6.12 | All Subjects | ASL MRI Results |
| 16.2.7 Adverse Eve | ent Listings (by Su | bject) |
| Listing 16.2.7.1 | All Subjects | Adverse Events |
| 16.2.8 Laboratory | Values and Other | Clinical Observations and Measurements (by Subject) |
| Listing 16.2.8.1.1 | All Subjects | Clinical Laboratory Data: Hematology |
| Listing 16.2.8.1.2 | All Subjects | Clinical Laboratory Data: Serum Chemistry |
| Listing 16.2.8.1.3 | All Subjects | Clinical Laboratory Data: Urinalysis |
| Listing 16.2.8.1.4 | All Subjects | Clinical Laboratory Data: Urine Drug Screen and Pregnancy Tests |
| Listing 16.2.8.1.5 | All Subjects | Clinical Laboratory Data: Coagulation |
| Listing 16.2.8.1.6 | All Subjects | Clinical Laboratory Data: Immunology |
| Listing 16.2.8.1.7 | All Subjects | Clinical Laboratory Data: Serology |
| Listing 16.2.8.2.1 | All Subjects | Vital Signs |
| Listing 16.2.8.2.2 | All Subjects | Blood Pressure |
| Listing 16.2.8.3 | All Subjects | 12-Lead Electrocardiogram (ECG) Results |
| Listing 16.2.8.4 | All Subjects | Echocardiogram Results |
| Listing 16.2.8.5.1 | All Subjects | Physical Examination |
| Listing 16.2.8.5.2 | All Subjects | Targeted Physical Examination |
| Listing 16.2.8.6 | All Subjects | S-STS |
| Listing 16.2.8.7 | All Subjects | Prior and Concomitant Medications |

### 13.5. Planned Figure Descriptions

**Table 6: Planned Figures** 



| Number | Population | Title | Safety IA | Efficacy<br>IA |
|---|---|---|---|---|
| Figure 14.2.1.1 | Evaluable | Boxplots of MoCA Total Scores by Visit and Treatment | | 207 |
| Figure 14.2.1.2 | Per<br>Protocol | Boxplots of MoCA Total Scores by Visit and Treatment | | |
| Figure 14.2.2.1 | Evaluable | Boxplots of D-KEFS Total Scores by<br>Visit and Treatment | | |
| Figure 14.2.2.2 | Per<br>Protocol | Boxplots of D-KEFS Total Scores by<br>Visit and Treatment | | |
| Figure 14.2.3.1 | Evaluable | Boxplots of MDS-UPDRS Parts 1-3<br>Scores by Visit and Treatment | | |
| Figure 14.2.3.2 | Per<br>Protocol | Boxplots of MDS-UPDRS Parts 1-3<br>Scores by Visit and Treatment | | |
| Figure 14.2.3.3 | Evaluable | Boxplots of MDS-UPDRS Part 1 Scores<br>by Visit and Treatment | | |
| Figure 14.2.3.4 | Per<br>Protocol | Boxplots of MDS-UPDRS Part 1 Scores<br>by Visit and Treatment | | |
| Figure 14.2.3.5 | Evaluable | Boxplots of MDS-UPDRS Part 2 Scores<br>by Visit and Treatment | | |
| Figure 14.2.3.6 | Per<br>Protocol | Boxplots of MDS-UPDRS Part 2 Scores<br>by Visit and Treatment | | |
| Figure 14.2.3.7 | Evaluable | Boxplots of MDS-UPDRS Part 3 Scores<br>by Visit and Treatment | | |
| Figure 14.2.3.8 | Per<br>Protocol | Boxplots of MDS-UPDRS Part 3 Scores<br>by Visit and Treatment | | |
| Figure 14.3.1.1 | Safety | Hematology Data by Parameter, Visit, and Treatment | | |
| Figure 14.3.1.2 | Safety | Serum Chemistry Laboratory Data by<br>Parameter, Visit, and Treatment | | |
| Figure 14.3.1.3 | Safety | Quantitative Urinalysis Laboratory Data<br>by Parameter, Visit, and Treatment | | |
| Figure 14.3.2.1 | Safety | Hematology: Mean (SD) by Parameter,<br>Visit, and Treatment | | |
| Figure 14.3.2.2 | Safety | Serum Chemistry: Mean (SD) by<br>Parameter, Visit, and Treatment | | |
| Figure 14.3.2.3 | Safety | Quantitative Urinalysis: Mean (SD) by<br>Parameter, Visit, and Treatment | | |

| Number | Population | Title | Safety IA | Efficacy<br>IA |
|---|---|---|---|---|
| Figure 14.3.3.1 | Safety | Vital Signs Data by Parameter, Visit, and Treatment | | |
| Figure 14.3.3.2 | Safety | Vital Signs: Mean (SD) by Parameter,<br>Visit, and Treatment | | |





# 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all TLFs in support of this study. Note that programming notes may be added if appropriate after each TLF shell.





### Page xx of xx Version <Study Population and if applicable subgroup Description> <Title of Table Listing or Figure> Body of Table, Listing or Figure <Table, Listing, Figure> xx.x.x Footnote 1 <if applicable> Recommendation is to keep footnotes to a minimum CONFIDENTIAL Footnote n+1 <ppppgm path and name>, <date> <Note: If directly Applicable> Footnote 2 < if applicable> Footnote n <if applicable> Protocol: ALK6021-201 Alkahest, Inc.





Planned Table Shells

14.2.





Summary of Subject Disposition ITT Set Table 14.1.1

| | Placebo | GREB021 | Owerall |
|---|---|---|---|
| Status | (N=XX) | (XX=N) | (XX=N) |
| Randomized | × | × | × |
| Completed Dosing Period 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Dosing Period 2 | XX (XX.X%) | XX (XX.X%) | (%X'XX) XX |
| Completed Study | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| Did not complete the study per protocol due to COVID-19 | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| Prematurely Discontinued from Study Reason for Discontinuation: | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| Adverse Event | (%X XX) XX | (%X XX) XX | (%X XX) XX |
| Death | XX (XX.X%) | (%XXX)XX | (%X XX) XX |
| Lost to Follow-up | XX (XX:X%) | (%X XX) XX | (%X XX) XX |
| Physician Decision | XX (XX.X%) | (%XXXX) XX | (%XXX)XX |
| Pregnancy | XX (XX.X%) | XX (XX.X%) | XX (XXXXX) |
| Protocol Deviation | XX (XX.X%) | XX (XX.X%) | (%X'XX) XX |
| Study Terminated by Sponsor | XX (XX.X%) | XX (XX.X%) | (%XXXX) XX |
| Withdrawal by Legally Authorized Representative | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| Withdrawal by Subject | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Worsening Condition | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | (%X.X%) XX |
| Completed Study Visit: | | | |
| Visit 1 | XX (XX.X%) | XX (XX.X%) | (%XXXX) XX |
| Visit 2 | XX (XX.X%) | (%XXXX)XX | (%X:XX) XX |
| Visit 3 | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Visit 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 5 | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| Visit 6 | XX (XX.X%) | XX (XX X%) | (%X'XX) XX |

Abbreviation: COVID-19 = novel coronavirus disease 2019; CRF = case report form;

Note: Percentages are based on the number of subjects randomized. A subject is considered to not have completed the study per protocol due to COVID-19 if they had any missing visits that affected treatment administration or collection of end of study efficacy assessments due to COVID-19. If a subject did not complete the study per protocol due to COVID-19, this category supersedes their study status on the study completion CRF.

[1] The ITT Set consists of all randomized subjects.
[2] The Safety Set consists of all subjects who received at least one dose of the study agent.
[3] The Evaluable Set consists of subjects who receive at least 5 of the 10 planned doses and complete through Visit 8.
[4] The Evaluable Set consists of subjects who receive at least 5 of the 10 planned doses, who complete Visit 18 and Visit 19 in window, and who have no protocol deviations that could affect the assessment of efficacy.
[5] The Complete Set is a subset of the PP Set comprised of subjects who did not have any changes to any of the following concomitant medications preferred terms reported at any time deviations that could affect the assessment (Neupro Patch)), Duopa Pump, Pimavanserin Tartate (Nuplazid), Quetiapine Furnarate (Seroquel), Sinemet [(Carbidopa, Levodopa]), Carbidopa, Rytary), Pregabalin (Lyrica), Amantadine, Antipsychotics (e.g. Pimavanserin Tartate (Nuplazid), Clozapine, Quetiapine Furnarate (Seroquel), or benzodiazepines (e.g. Approached per protocol beforeprior to first dose and either changed dose or stopped on study andas well as those that began on study.

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,

Source: Listing 16.2.1

Table 14.1.1 (cont.) Summary of Subject Disposition

| | Placebo | GRF6021 | Overall |
|---|---|---|---|
| Status | (XX=N) | (XX=N) | (XX=N) |
| Completed Study Visit: | | | |
| Visit 7 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 8 | (%X:X%) | XX (XX.X%) | (%X:XX) |
| Visit 9 | XX (XX,X%) | (%X:XX) XX | (%X:XX) XX |
| Visit 10 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 11 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 12 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 13 | (%X:X%) | XX (XX.X%) | XX (XX:X%) |
| Visit 14 | XX (XXXX%) | (%X'XX) XX | (%X:XX) |
| Visit 15 | XX (XX.X%) | XX (XX.X%) | (%X'XX) XX |
| Visit 16 | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| Visit 17 | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Visit 18 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Analysis Sets: | | | |
| [TT Set [1] | (%X:X%) | XX (XX.X%) | XX (XX:X%) |
| Safety Set [2] | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Evaluable Set [3] | (%X:X%) | XX (XX.X%) | (%X:XX) XX |
| Per Protocol Set [4]<br>Complete Set [5] | (%X:X%) | XX (XX.X%) | (%X:XX) XX |

Abbreviation: COVID-19 = novel coronavirus disease 2019.

Note: Percentages are based on the number of subjects randomized. A subject is considered to not have completed the study per protocol due to COVID-19 if they had any missing visits that affected treatment administration or collection of end of study efficacy assessments due to COVID-19.

[1] The ITT Set consists of all randomized subjects.
[2] The Safety Set consists of all subjects who received at least one dose of the study agent.
[3] The Evaluable Set consists of subjects who receive at least 5 of the 10 planned doses and complete through Visit 8.
[4] The Per Protocol Set is a subset of the Evaluable Set comprised of subjects who receive all 10 planned doses, who complete Visit 18 and Visit 19 in window, and who have no protocol deviations that could affect the assessment of efficacy.

[5] The Complete Set is a subset of the PP Set comprised of subjects who did not have any changes to any of the following concomitant medications preferred terms reported at any time on study: Dopaminergic agents (e.g. Rotigotine [Neupro Patch], Duopa Pump, Sinemet [Carbidopa, Levodopa], Carbidopa, Rytary), Pregabalin (Lyrica), Amantadine, Antipsychotics (e.g. Pimavanserin Tartate [Nuplazid], Clozapine, Quetiapine Fumarate [Seroquet]), or benzodiazepines (e.g. Alprazolam). This includes those that were stable per protocol prior to first dose and either changed dose or stopped on study as well as those that began on study. Source: Listing 16.2.1



Table 14,1,2 Demographics and Baseline Characteristics ITT Set

| Vanable | Placebo | GRF6021 | Overall |
|------------------------------|------------|------------|-------------|
| Statistic or Category | (XX=X) | (N=XX) | (N=XX) |
| Age (years) | | | |
| | × | × | ×× |
| Mean (SD) | XXX (XXX) | XXX XXX | XXXX XXX |
| Median | XXX | ××× | XXX |
| Min, Max | XX XX | XX XX | XX XX |
| P value [1] | | XXXXX | to the |
| Sex | | | |
| Male | XX (XX.X%) | (%X XX) XX | (%X XX) XX |
| Female | (%X XX) XX | (%X XX) XX | (%X XX) XX |
| P value [2] | | XXXXX | (ormal) var |
| Child-Bearing Potential? [3] | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX XXX XX |
| No | XX (XX X%) | XX (XX.X%) | XX (XX.X%) |
| Ethnicity | | | |
| Hispanic or Latino | (%X'XX) XX | (%X XX) XX | 1%X XX/ XX |
| Not Hispanic or Latino | XX (XX:X%) | XX (XX.X%) | XX XXX XX |
| P value [2] | | XXXXX | |

Abbreviations: ApoE = polopoprotein E; CRF = case report form; PD = Parkinson's Disease.

Note: Percentages are n/Number of subjects in the ITT Set\*100. Subjects are summarized by randomized treatment. Disease duration = [Enrollment date – PD onset date (as recorded on the Medical History CRF) + 1] / 365.

[1] P value from Wilcoxon rank-sum test.
[2] P value from Chi-square test.
[3] Only captured for female subjects; percentages are based on the number of female subjects in the ITT Set.
[4] Obtained from Visit 3 blood draw.
Source: Listing 16.2.4.1



Table 14.1.2 (cont.) Demographics and Baseline Characteristics ITT Set

| | (X=X) | (N=XX) | (N=XX) |
|---|---|---|---|
| Race | | | |
| White | (%X:XX) | XX (XX.X%) | XX (XX.X%) |
| Black or African-American | (%X:XX) | XX (XX.X%) | XX (XX.X%) |
| Asian | (%X:XX) | XX (XX.X%) | (%X:XX) XX |
| American Indian or Alaska Native | (%X:X%) | XX (XX,X%) | (%X:XX) XX |
| Native Hawaiian or Other Pacific Islander | XX (XX.X%) | XX (XX.X%) | (%X XX) XX |
| More than One Race<br>P value [2] | (%X XX) XX | XX (XX X%)<br>X XXXX | (%XXX)XX |
| Height (cm) | ***** | 100 | |
| | X | X | × |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Min, Max.<br>P value [1] | XX, XX | XX, XX<br>X, XXXX | XX, XX |
| weight (kg) | | | |
| | X | X | × |
| Mean (SD) | XXX (XXX) | XXX (XXX) | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Min, Max | XX, XX | XX, XX | XX.XX |
| P value [1] | | X.XXXX | |
| Body Mass Index (kg/m²) | | | |
| | × | X | × |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XXX | XXX | xxx |
| Min, Max | XX, XX | XX, XX | XX, XX |
| P value [1] | | XXXXX | |

Abbreviations: ApoE = polopoprotein E; CRF = case report form; PD = Parkinson's Disease.

Note: Percentages are n/Number of subjects in the ITT Set\*100. Subjects are summarized by randomized treatment. Disease duration = [Enrollment date - PD onset date (as recorded on the Medical History CRF) + 1] / 365.

<sup>[1]</sup> P value from Wilcoxon rank-sum test.
[2] P value from Chi-square test.
[3] Only captured for female subjects; percentages are based on the number of female subjects in the ITT Set.
[4] Obtained from Visit 3 blood draw.
Source: Listing 16.2.4.1

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



Table 14.1,2 (cont.)
Demographics and Baseline Characteristics ITT Set

| Variable<br>Statistic of Catagoria | Placebo | GRF6021 | Overall |
|------------------------------------|------------|------------|------------|
| Statistic of Category | (XX=X) | (N=XX) | (N=XX) |
| Disease Duration (years) | | | |
| U | × | × | × |
| Mean (SD) | XXX (XXX) | XXX XXX | XXX (XXX) |
| Median | XXX | XXX | XXX |
| Min, Max | XX. XX | XX XX | XX XX |
| P value [1] | | XXXXX | |
| ApoE Genotype [4] | | | |
| 2/2 | XX (XX:X%) | XX (XX.X%) | (%XXXX) XX |
| 2/3 | XX (XX.X%) | XX (XX.X%) | XX XXX XX |
| 3/3 | XX (XX.X%) | (%X:XX) XX | (%X XX) XX |
| 4/3 | XX (XX.X%) | XX (XX.X%) | (%XXXX) XX |
| 4/4 | XX (XX.X%) | XX (XX.X%) | (%X'XX) XX |
| 2/4 | XX (XX.X%) | XX (XX,X%) | (%XXX)XX |
| P value [2] | | XXXXX | |

Abbreviations: ApoE = polopoprotein E; CRF = case report form; PD = Parkinson's Disease.

Note: Percentages are n/Number of subjects in the ITT Set\*100. Subjects are summarized by randomized treatment. Disease duration = [Enrollment date – PD onset date (as recorded on the Medical History CRF) + 11 / 365.

[1] P value from Wilcoxon rank-sum test.

[2] P value from Chi-square test.

[3] Only captured for female subjects; percentages are based on the number of female subjects in the ITT Set.

[4] Obtained from Visit 3 blood draw.

Programming Note: If cell counts are <5, use Fisher's Exact Test and update footnote accordingly.

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



Summary of Medical History by SOC, PT, and Treatment.
Safety Set

| System Organ Class<br>Preferred Term | Placebo<br>(N=XX) | GRF6021<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Subjects with at least 1 Recorded Medical History | (%X'XX) XX | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | (%X'XX) XX | XX (XX:X%) | XX (XX.X%) |
| Preferred Term 3 | (%X'XX) XX | XX (XX.X%) | (%XXXX) |
| System Organ Class 2 | (%X'XX) XX | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: PT = Preferred Term; SOC = System Organ Class.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. Medical histories were coded using MedDRA version 21.0. Subjects were counted once for each system organ class (SOC) and once for each preferred term (PT). Medical history terms are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT.

SOURCE: Listing 16.2.4.2.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell.

Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan, Sponsor Alkahest, Inc.



Table 14.1.3.2 Summary of Parkinson's Disease Medical History by SOC, PT, LLT and Treatment Safety Set

| System Organ Class Preferred Term Lower Level Term | Placebo<br>(N=XX) | GRF6021<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 Recorded Medical History | XX (XX.X%) | (%X.X%) | XX (XX X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX X%) | XX (XX.X%) | XX (XX:X%) |
| Lower Level Term 1 | XX (XX.X%) | (%X'XX) XX | (%X XX) XX |
| Lower Level Term 2 | XX (XX.X%) | (XX.XX) XX | (%X XX) XX |
| System Organ Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| Lower Level Term 1 | | XX (XX.X%) | XX (XX X%) |
| Lower Level Term 2 | XX (XX X%) | XX (XX:X%) | XX (XX.X%) |

Abbreviations: LLT = Lower Level Term; PT = Preferred Term: SOC = System Organ Class.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. Medical histories were coded using MedDRA version 21.0.

This table contains histories of Parkinson's Disease-Mild Cognitive Impairment and Parkinson's Disease-Dementia which includes the following LLTs: Parkinson's Disease, cognitive disorder, cognitive impairment, and dementia. Subjects were counted once for each system organ class (SOC), once for each preferred term (PT) and once for each Lower Level Term (LLT). Medical history terms are displayed by descending frequency of SOC, then PT within SOC, then LLT within PT, and then alphabetically by LLT. SOURCE: Listing 16.2.4.2.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell.

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



Table 14.1.4
Summary of Prior Medications by ATC Class Level 4, PT, and Treatment
Safety Set

| ATC Class Level 4 Preferred Term (ATC Class Level 5) | Placebo<br>(N=XX) | GRF6021<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Subjects with at least 1 Prior Medication | XX (XX.X%) | (%X.XX) XX | XX (XX.X%) |
| Subjects with at least 1 Prior Medication for Cognition Subjects with at least 1 Prior Medication for Cognition | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | XX (XX.X%) | (%XXXX) XX | XX (XX.X%) |
| Preferred Term 1 | XX (XX:X%) | XX (XX.X%) | XX (XX X%) |
| Preferred Term 2 | (%X:XX) XX | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX,X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | (%X'XX) |

Medications that started before first dose will be considered prior medications whether or not they were stopped before dose. Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by PT within ATC, and then alphabetically. Subjects were counted only once for each ATC and PT. Medications for PD are identified from the indication field on the CRF as well as those in ATC Classes N04, N04A, and N04B. Medications for cognition are identified by ATC Class N06D and N06DX. SOURCE: Listing 16.2.8.6 Abbreviations: ATC = Anatomical Therapeutic Chemical; PD = Parkinson's Disease; PT = Preferred Term.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. Medications were coded using WHODrug version March 2018.

Programming note: ATC & PT text should be in proper case in table, as shown in the shell. Ensure correct WHODrug version is printed in footnote.



Table 14.1.5 Summary of Exposure by Treatment Safety Set

| Dosing Period: Overall | | | |
|---|---|---|---|
| Variable / Statistic | Placebo<br>(N=XX) | GRF6021<br>(N=XX) | Overall (N=XX) |
| Evaluable Subjects [1] | (%X`XX) XX | XX (XX.X%) | XX (XX.X%) |
| Total Number of Exposure Days | | | |
| u u | × | ×× | XX |
| Mean (SD) | XXX (XXXXX) | XX XX XXX | (XX XX) X XX |
| Median | XXX | XXX | ××× |
| Min, Max | XX,XX | xx, xx | XX, XX |
| Actual Volume Administered | | | |
| Ü | XX | X | XX |
| Mean (SD) | (XX XXX XXX | (XX XX) X XX | XX XX/ XXX |
| Median | XXX | XXX | ××× |
| Min, Max | XX'XX | XX.XX | ×××× |

Continue for Dosing Period 1 and Dosing Period 2

Note Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. [1] The duration of therapy for a subject to be considered evaluable is 5 exposure days. SOURCE: Listing 16.2.5



Table 14.2.1.1 Summary of Change from Baseline in MoCA Scores by Treatment Evaluable Set

| Parameter, lotal score | | | | | | |
|---|---|---|---|---|---|---|
| Study Visit | | Placebo<br>(N=XX) | | | GRF6021<br>(N=XX) | |
| Statistic | Observed | CFB | %CFB | Observed | CFB | %CFB |
| Baseline [1] | | | | *** | | |
| | × | | | XX | | |
| Mean (SD) | XX.X (XX.XX) | | | (XX XX) | | |
| Median | ××× | | | XXX | | |
| Min, Max | XX.XX | | | XX.XX | | |
| Veek 4 (Visit 9) | | | | | | Ž. |
| | × | × | × | × | × | × |
| Mean (SD) | XXX (XXXX) | XX.X (XX.XX) | XX.X (XX.XX) | XXX (XXXXX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XXX | XXX | XXX | XXX | XXX | XXX |
| Min, Max | XX, XX | xx,xx | XX, XX | ×××× | XX, XX | XX, XX |
| P value [2] | | | | | X.XXXX | |
| Week 16 (Visit 17) | | | | | | |
| | ×× | × | × | × | × | × |
| Mean (SD) | XX.X (XX.XX) | (XX.XX) X.XX | XX.X (XX.XX) | XX.X (XX.XX) | (XX XX) XXX | (XX.XX) X.XX |
| Median | XXX | XXX | XXX | XXX | XXX | XXX |
| Min, Max<br>Divable (2) | XX,XX | XX. XX | XX, XX | XX, XX | XX XX | XX.XX |
| י אמומה [ד] | | | Repeat for all parameters. | | | |

Abbreviations: CFB = change from baseline; MoCA = Montreal Cognitive Assessment.

Note: Higher scores indicate better cognitive function; the total possible score is 30 and a score of 26 or more is considered normal. A positive value of change means an improvement, and a negative value of change means deterioration. Subjects are summarized by randomized treatment.

[1] The baseline value is the MoCA Score from Visit 1 (Screening).
[2] P-value for testing mean change from baseline to subsequent visit is 0 is calculated using a paired I-test. SOURCE: Listing 16.2.6.1

Programming note: Check normality per Section 8.2 of the SAP. If the data are non-normal, use the Wilcoxon signed-rank test and update the footnote accordingly. Parameters will be: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, orientation.



Table 14.2.1.2
Mean Change from Baseline in MoCA Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA Evaluable Set

| Study Visit<br>Stalistic [1] | Placebo<br>(N=XX) | GRF6021<br>(N=XX) |
|---|---|---|
| Week 4 (Visit 9) | | |
| | X | × |
| LS Mean Change from Baseline (SE) | XXX (XXX) | XXX (XXX) |
| (95% Ct for LS Mean Change from Baseline) P value for LS Mean Change from Baseline) [2] | (XXX,XXX) | (XXX, XXX) |
| LS Mean Difference from Placebo (SE) (95% CI for Difference from Placebo) | | (XXX) XXX |
| P value for Difference from Placebo [3] | | XXXXX<br>XXXXX |
| Week 16 (Visit 17) | | |
| | XX | × |
| LS Mean Change from Baseline (SE) | XX.X (X.XX) | XX.X (X.XX) |
| (35% CLTor LS Mean Change from Baseline) P value for LS Mean Change from Baseline) [2] | (XXX, XXX) | (XXX, XXX) |
| LS Mean Difference from Placebo (SE) | | CAA AV A AA |
| (95% CI for Difference from Placebo) | | (XXX, XXX) |
| P value for Difference from Placebo [3] | | XXXXX |

Abbreviations: ANCOVA = analysis of covariance; ApoE = apolopoprotein E; CI = confidence interval; LS = least squares; MoCA = Montreal Cognitive Assessment; SE = standard

Note: Higher scores indicate better cognitive function; the total possible score is 30 and a score of 26 or more is considered normal. A positive value of change means an improvement, and a negative value of change means deterioration. Subjects are summarized by randomized treatment.

[1] Estimates for LS means (change from baseline and difference from placebo [ie, change from baseline for Placebo]) and accompanying 95% Cls and P values are from an ANCOVA model with treatment, visit, and treatment-by-visit interaction as the main effects, and baseline MoCA total score, age,

and ApoE genotype as covariates.
[2] P value for testing mean change from baseline is 0.
[3] P value for testing difference (GRF6021 minus Placebo) in mean change from baseline from is 0. SOURCE: Listing 16.2.6.1

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,

Table 14.2.1.3
Summary of Change from Baseline in MoCA Total Score by Treatment.
Per Protocol Set

### (Same Shell as Table 14.2.1.1)

Table 14.2.14

Mean Change from Baseline in MoCA Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA Per Protocol Set

### (Same Shell as Table 14.2.1.2)

Table 14.2.1.5
Summary of Change from Baseline in MoCA Total Score by Treatment
Complete Set

### (Same Shell as Table 14.2.1.1)

Table 14.2.1.6
Mean Change from Baseline in MoCA Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA Complete Set

## (Same Shell as Table 14,2.1.2)



Summary of Change from Baseline in D-KEFS Scores by Treatment Table 14.2.2.1 Evaluable Set

Programming Note: Parameters will be Total Score, Letter Fluency, Category Fluency, and Category Switching. Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 16), and Week 20 (Visit 18). Add D-KEFs to abbreviations. Update footnote to read [1] The baseline value is the D-KEFS Score from Visit 2 or before." SOURCE: Same Shell as Table 14.2.1.1 Listing 16.2.6.2.

Mean Change from Baseline in D-KEFs Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Table 14.2.2.2 Evaluable Set

Programming Note: Add D-KEFs to abbreviations. SOURCE: Listing 16.2.6.2. Same Shell as Table 14.2.1.2

Table 14.2.2.3

Summary of Change from Baseline in D-KEFs Scores by Treatment

Per Protocol Set

Same Shell as Table 14.2.1.1

Programming Note: Parameters will be Total Score, Letter Fluency, Category Fluency, and Category Switching. Visits will be Baseline (Visit 2), Week 1 (Visit 16), and Week 20 (Visit 18), Add D-KEFs to abbreviations. Update footnote to read [1] The baseline value is the D-KEFS Score from Visit 2 or before." SOURCE: Listing 16.2.6.2. Update footnote to reflect Per Protocol Set. Mean Change from Baseline in D-KEFs Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Table 14.2.2.4

Programming Note: Add D-KEFs to abbreviations. SOURCE: Listing 16.2.6.2. Update footnote to reflect Per Protocol Set. Same Shell as Table 14.2.1.2

Per Protocol Set

Statistical Analysis Plan. Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Summary of Change from Baseline in D-KEFs Scores by Treatment

Complete Set

Programming Note: Parameters will be Total Score, Letter Fluency, Category Fluency, and Category Switching: Visits will be Baseline (Visit 2), Week 1 (Visit 3), Week 8 (Visit 10), Week 10 (Visit 18), Add D-KEFs to abbreviations. Update footnote to read 111 The baseline value is the D-KEFS Score from Visit 2 or before." SOURCE: Listing 16.2.6.2. Update footnote to reflect Complete Set. Same Shell as Table 14.2.1.1

Table 14.2.2.6
Mean Change from Baseline in D-KEFs Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Complete Set

Programming Note: Add D-KEFs to abbreviations, SOURCE: Listing 16.2.6.2. Update footnote to reflect Complete Set. Same Shell as Table 14.2.1.2



Table 14.2.3.1
Summary of Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Scores by Treatment
Evaluable Set

### Same Shell as Table 14.2.1.1

Programming Note: Parameters will be Total Score, Part 1 Score, Part 2 Score and Part 3 Score. Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 17), Week 20 (Vsit 18), and Week 24 (Visit 19), Add MDS-UPDRS to abbreviations. Update footnote to read [1] The baseline value is the MDS-UPDRS Score from Visit 2 or before." SOURCE: Listing 16.2.6.3.

Table 14.2.3.2
Mean Change from Baseline in MDS-UPDRS Parts 1-3 Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Evaluable Set

Same Shell as Table 14,2,1,2,

Programming Note: Add MDS-UPDRS to abbreviations. Age and baseline score will be the only covariates used in the model, update footnote accordingly. SOURCE: Listing 16.2.6.3.

Table 14.2.3.3
Summary of Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Scores by Treatment
Per Protocol Set

Same Shell as Table 14.2.1.1

Programming Note: Parameters will be Total Score, Part 1 Score, Part 2 Score and Part 3 Score. Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 18), Week 8 (Visit 18), Add MDS-UPDRS to abbreviations. Update footnote to read [11] The baseline value is the MDS-UPDRS Score from Visit 2 or before," SOURCE: Listing 16.2.6.3. Update footnote to reflect Per Protocol Set.

Table 14.2.3.4
Mean Change from Baseline in MDS-UPDRS Parts 1-3 Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA

Per Protocol Set Same Shell as Table 14,2,1,2

Programming Note: Add MDS-UPDRS to abbreviations. Age and baseline score will be the only covariates used in the model, update footnote accordingly. SOURCE: Listing 16.2.6.3. Update footnote to reflect Per Protocol Set.

Protocol Number ALK 6021-201 Statistical Analysis Plan, PCN Number ALKA7951 Sponsor Alkahest, Inc.

Summary of Change from Baseline in MDS-UPDRS Parts 1, 2, and 3 and Parts 1-3 Total Scores by Treatment Complete Set Table 14.2.3.5

Programming Note: Parameters will be Total Score, Part 1 Score, Part 2 Score and Part 3 Score. Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 17), Week 20 (Vsit 18), and Week 24 (Visit 19). Add MDS-UPDRS to abbreviations. Update footnote to read [11] The baseline value is the MDS-UPDRS Score from Visit 2 or before." SOURCE: Listing 16.2.6.3. Update footnote to reflect Complete Set. Same Shell as Table 14.2.1.1

Mean Change from Baseline in MDS-UPDRS Parts 1-3 Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Table 14.2.3.6 Complete Set

Programming Note: Add MDS-UPDRS to abbreviations. Age and baseline score will be the only covariates used in the model, update footnote accordingly, SOURCE: Listing 16.2.6.3. Update footnote to reflect Complete Set. Same Shell as Table 14.2.1.2


Table 14.2.4.1 Summary of SE-ADL by Study Visit and Treatment. Evaluable Set

| Baseline [1] 100% = Completely independent, ability to do chores essentially normal. 100% = Completely independent, ability to do chores essentially normal. 100% = Completely independent, above stakes twice as long. 100% = Completely independent. Spend a large part of day with chores. 100% = Not completely independent. Spend a large part of day with chores. 100% = Not completely independent. Spend a large part of day with chores. 100% = Not dependent. Can assist with all chores but few alone. 100% = A busine dependent. Help with half of chores. 100% = Nothing alone. Severe invalid. 100% = Totally dependent, helpless. Complete invalid. 100% = Totally dependent, ability to do chores essentially normal. 100% = Nothing alone. Severe might alex wice as long. 100% = Nothing alone. Severe might alex wice as long. 100% = Nothing alone. Severe might alex with a long. 100% = Completely independent, ability to do chores essentially sowly. 100% = Nothing alone. Severe might alex with a long. 100% = Nothing alone. Severe might alex with a long. 100% = Nothing alone. Severe might alex with a long. 100% = Nothing alone. Severe might alex with a long. 100% = Nothing alone. Severe might alex with all chores. 100% = Nothing alone. Severe might alex with all chores. 100% = Nothing alone. Severe might alex with all chores. 100% = Nothing alone. Severe might alex with all chores. 100% = Nothing alone. Severe method. 100% = Nothing alone. Severe met | Study Visit<br>Statistic | | Placebo<br>(N=XX) | GRF6021<br>(N=XX) |
|---|---|---|---|---|
| ely independent, ability to do chores essentially normal. ely independent, chores might take twice as long. ely independent in most chores, akes twice as long. ely independent in most chores, akes twice as long. pletely independent. Spend a large part of day with chores, pendency. Can do most chores, but exceedingly slowly. pendency. Can do most chores, but few alone. pendent. Help with half of chores. endent. Can assists with all chores but few alone. pendent. Help with half of chores. ependent, Helpless. Complete invalid. pendent, helpless. Complete invalid. gly independent, ability to do chores essentially normal. ely independent, chores might take twice as long. ely independent. Spend a large part of day with chores. pendency. Can do most chores, takes twice as long. pendency. Can do most chores, but exceedingly slowly. pendency. Can do most chores. alone or begins alone. Much help needed. alone. Severe invalid. pendent. Help with half of chores but few alone. ores alone or begins alone. Much help needed. pendent, helpless. Complete invalid. | Baseline [1] | | | |
| inplately independent, chrores might take twice as long. Implately independent, chrores might take twice as long. Inplately independent in most chores, takes twice as long. Completely independent. Spend a large part of day with chores. In a dependent. Help with half of chores. In a dependent, can assist with all chores but few alone. In a dependent, can assist with all chores but few alone. In a dependent, can assist with all chores but few alone. In a dependent, a defider. In a dependent, a defider. In a dependent, a defider. In a dependent, chores might take twice as long. In a dependent, chores might take twice as long. In a dependent, chores might take twice as long. In a dependent, chores might take twice as long. In a dependent. Spend a large part of day with chores. In a dependent. Can assist with all chores but few alone. In a dependent. Can assist with all chores but few alone. In dependent. A ledge with help needed. In a dependent, help with help needed. In a dependent, help with help needed. In a dependent, help less. Complete invalid. In a dependent, helpless. Complete invalid. In a dependent, helpless. Complete invalid. | 100% = Completely independent, ability to do chores esser | tially normal, | XX (XX.X%) | XX (XX,X%) |
| left in the pendent in most chores, takes twee as long. pletely independent. Spend a large part of day with chores, spendency. Can do most chores, but exceedingly slowly. pendent. Can assist with half of chores but few alone. pendent. Can assist with all chores but few alone. pendent. Can assist with all chores but few alone. pendent, helpess, Complete invalid. alone. Severe invalid. pendent, helpess, Complete invalid. a functions. Bedridden. by independent, ability to do chores essentially normal. by independent, chores might take twice as long. all independent. Spend a large part of day with chores. between most chores, but exceedingly slowly. bendent. Can do most chores, but exceedingly slowly. bendent. Can assist with all chores but few alone. ores alone or begins alone. Much help needed. alone. Severe invalid. alone. Severe invalid. but the pless. Complete Invalid. alone invalid. | 90% = Completely independent, chores might take twice a | lang. | XX (XX.X%) | XX (XX X%) |
| pletely independent. Spend a large part of day with chores, spendency. Can do most chores, but exceedingly slowly. Pendency. Can do most chores, but exceedingly slowly. Pendent. Help with half of chores. Bendent. All a sasist with all chores but few alone. Ores alone or begins alone. Much help needed. Bendent. Repliess. Complete invalid. Bendency. Camplete invalid. Punctions. Bedridden. I unctions. Bedridden. | 80% = Completely independent in most chores, takes twice | as long. | XX (XX:X%) | XX (XX.X%) |
| pendency. Can do most chores, but exceedingly slowly. pendent. Help with half of chores. pendent. Can assist with all chores but few alone. pendent. Can assist with all chores. alone. Severe invalid. pendent, helpless. Complete invalid. pendent, helpless. Complete invalid. punctions. Bedridden. pendent, chores, takes twice as long. pethy independent, in most chores, takes twice as long. pethy independent. Spend a large part of day with chores. pendency. Can do most chores, but exceedingly slowly. pendent. Help with half of chores. pendent. Can assist with all chores but few alone. ores alone or begins alone. Much help needed. alone. Severe invalid. pendent, helpless. Complete Invalid. | /0% = Not completely independent. Spend a large part of | ay with chores. | XX (XX:X%) | XX XXX XX |
| pendent. Help with half of chores. endent. Can assist with all chores but few alone. endent. Can assist with all chores but few alone. alone. Severe invalid. ependent, helpless. Complete invalid. a functions. Bedridden. functions. Bedridden. et with a bility to do chores essentially normal. et with independent, chores might take twice as long. et with independent in most chores, takes twice as long. et with independent. Spend a large part of day with chores. pendency. Can do most chores, but exceedingly slowly. endent. Can assist with all chores but few alone. endent. Can assist with all chores but few alone. endent. Can assist with half of chores. alone. Severe invalid. ependent, helpless. Complete invalid. functions. Bedridden. | 60% = Some dependency. Can do most chores, but excee | ingly slowly. | XX (XX.X%) | XX XXX XX |
| endent. Can assist with all chores but few alone. ores alone or begins alone. Much help needed. alone. Severe invalid. spendent, helpless. Complete invalid. stunctions. Bedridden. stunctions. Bedridden. stunctions and state the state of the state | 50% = More dependent. Help with half of chores. | | XX (XXXX%) | XX (XX.X%) |
| ores alone or begins alone. Much help needed. alone. Severe invalid. spendent, helpless. Complete invalid. stunctions. Bedridden. stunctions. Bedridden. stunctions ability to do chores essentially normal. stunctions ability to do chores essentially normal. stunctions ability to do chores essentially normal. stunctions ability to do chores as long. stunctions ability to do chores as long. spendent, can do most chores, but exceedingly slowly. sendent. Can do most chores. sendent. Can assist with all chores but few alone. ores alone or begins alone. Much help needed. solones Severe invalid. stunctions. Bedridden. | 40% = Very dependent. Can assist with all chores but few | lone. | XX (XX:X%) | XX XXXXX |
| alone. Severe invalid. ependent, helpless. Complete invalid. ependent, helpless. Complete invalid. functions. Bedridden. ethy independent, ability to do chores essentially normal. ethy independent, chores might take twice as long. ely independent in most chores, takes twice as long. ely independent in most chores, but exceedingly slowly. pendent. Can do most chores, but exceedingly slowly. pendent. Help with half of chores but few alone. endent. Can assist with all chores but few alone. alone or begins alone. Much help needed. alone. Severe invalid. ependent, helpless. Complete Invalid. | | ed. | (%X:XX) XX | XX XXXXX |
| ependent, helpless. Complete invalid. I functions. Bedridden. I functions. Bedridden. I the pendent, ability to do chores essentially normal. I the pendent, chores might take twice as long. I the pendent in most chores, takes twice as long. I the pendent in most chores, but exceedingly slowy. I the point half of chores. I the point half of chores. I the point half of chores but few alone. I the point half of chores but few alone. I severe invalid. I the pedent invalid. I the pedent invalid. | 20% = Nothing alone. Severe invalid. | | XX (XX.X%) | XX XXX XX |
| tely independent, ability to do chores essentially normal. lety independent, chores might take twice as long. ely independent, chores, takes twice as long. ely independent in most chores, takes twice as long. pletely independent. Spend a large part of day with chores. pendency. Can do most chores, but exceedingly slowly. pendency. Can do most chores. pendency. Lely with half of chores. pendent. Help with half of chores but few alone. pendent. Can assist with all chores but few alone. slone or begins alone. Much help needed. slone. Severe invalid. providence. Severe invalid. | 10% = Totally dependent, helpless. Complete invalid. | | XX (XX:X%) | (%XXX)XX |
| tely independent, ability to do chores essentially normal. ely independent, chores might take twice as long. ely independent in most chores, takes twice as long. pletely independent. Spend a large part of day with chores. spendency. Can do most chores, but exceedingly slowly. pendency. Can assist with half of chores but few alone. endent. Can assist with all chores but few alone. severe invalid. stones. Severe invalid. stunctions. Bedridden. | 0% = Vegetative functions. Bedridden, | | XX (XX:X%) | XX (XX X%) |
| tely independent, ability to do chores essentially normal. ely independent, chores might take twice as long. ely independent in most chores, takes twice as long. ely independent in most chores, takes twice as long. pletely independent. Spend a large part of day with chores. pendency. Can do most chores, but exceedingly slowly. pendent. Help with half of chores endent. Can assist with all chores but few alone. gress alone or begins alone. Much help needed. slone. Severe invalid. pendent, helpless. Complete invalid. | P value [2] | | | XXXXX |
| ompletely independent, ability to do chores essentially normal. Independent, chores might take twice as long. Independent in most chores, takes twice as long. Completely independent in most chores, takes twice as long. Completely independent. Spend a large part of day with chores. The dependency. Can do most chores, but exceedingly slowly. The dependent. Help with half of chores but few alone. The dependent is an assist with all chores but few alone. The dependent is a single with help needed. The dependent is a single with help needed. Thing alone. Severe invalid. The dependent, helpless. Complete invalid. | Veek 8 (Visit 10) | | | |
| mpletely independent, chores might take twice as long. mpletely independent in most chores, takes twice as long. completely independent. Spend a large part of day with chores. ne dependency. Can do most chores, but exceedingly slowly. re dependent. Help with half of chores but few alone. we dependent. Act an assist with all chores but few alone. we chores alone or begins alone. Much help needed. hing alone. Severe invalid. ally dependent, helpless. Complete invalid. | 100% = Completely independent, ability to do chores esser | tially normal. | XX (XX:X%) | (%X'XX) XX |
| npletely independent in most chores, takes twice as long. completely independent. Spend a large part of day with chores. ne dependency. Can do most chores, but exceedingly slowly. re dependent. Help with half of chores. w chores alone or begins alone. Much help needed. hing alone. Severe invalid. ally dependent, helpless. Complete invalid. | 90% = Completely independent, chores might take twice as | long. | XX (XX.X%) | XX (XX.X%) |
| completely independent. Spend a large part of day with chores, ne dependency. Can do most chores, but exceedingly slowly. e dependency. Can do most chores. e dependent. Help with half of chores but few alone. A dependent. Can assist with all chores but few alone. Who chores alone or begins alone. Much help needed. white alone. Severe invalid. ally dependent, helpless. Complete invalid. | 80% = Completely independent in most chores, takes twice | as long. | XX (XX.X%) | XX (XX:X%) |
| ne dependency. Can do most chores, but exceedingly slowly. e dependent. Help with half of chores. y dependent. Can assist with all chores but few alone. y dependent or begins alone. Much help needed. hing alone. Severe invalid, ally dependent, helpless. Complete invalid. | /0% = Not completely independent. Spend a large part of or | ay with chores. | XX (XX.X%) | XX (XX.X%) |
| re dependent. Help with half of chores. y dependent. Can assist with all chores but few alone. y dependent. Can assist with all chores but few alone. wy chores alone or begins alone. Much help needed. ling alone. Severe invalid, ally dependent, helpless. Complete invalid. | 60% = Some dependency. Can do most chores, but excee | ingly slowly. | XX (XX.X%) | XX (XX.X%) |
| y dependent. Can assist with all chores but few alone. sw chores alone or begins alone. Much help needed. hing alone. Severe invalid, alone or begins alone or begins alone alone. Severe invalid, ally dependent, helpless. Complete invalid. | 50% = More dependent. Help with half of chores. | | XX (XX.X%) | XX (XX.X%) |
| sw chores alone or begins alone. Much help needed. hing alone. Severe invalid, ally dependent, helpless. Complete invalid. stative functions. Bedridden. | 40% = Very dependent. Can assist with all chores but few | one. | XX (XX:X%) | XX (XX.X%) |
| hing alone. Severe invalid, ally dependent, helpless. Complete invalid. stative functions. Bedridden. | | ed. | XX (XX X%) | XX (XX XX) |
| ally dependent, helpless. Complete invalid. | 20% = Nothing alone. Severe invalid, | | XX (XX.X%) | (%XXXX)XX |
| stative functions. Bedridden, | 10% = Totally dependent, helpless. Complete invalid. | | XX (XX.X%) | XX (XX.X%) |
| I vaine [7] | 0% = Vegetative functions. Bedridden. | | XX (XX:X%) | (%X'XX) XX |
| | r value [4] | | | XXXXX |

Continue for Week 24 (Visit 19).

Abbreviations: CMH = Cochran-Mantel-Haenszel; SE-ADL = Schwab and England Activities of Daily Living Scale.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized treatment.

[1] The baseline value is the SE-ADL Score from Visit 2.

[2] P value from CMH test.

SOURCE: Listing 16.2.6.4

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,

Table 14.2.4.2 Summary of SE-ADL by Study Visit and Treatment Per Protocol Set

(Same Shell as Table 14.2.4.1)

Programming Note: Update footnote to reflect Per Protocol Set.

Table 14.2.4.3 Summary of SE-ADL by Study Visit and Treatment Complete Set

(Same Shell as Table 14.2.4.1)

Programming Note: Update footnote to reflect Complete Set.

Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan, Sponsor Alkahest, Inc.



Table 14.2.5.1

Summary of Change from Baseline in CISI-PD Scores by Treatment

Evaluable Set

Programming Note: Parameters will be Total Score, Motor Signs, Disability, Motor Complications, and Cognitive Status. Visits will be Baseline (Visit 2), Week 8 (Visit 10), and Week 24 (Visit 19). Add CISI-PD to abbreviations. Update footnote to read [1] The baseline value is the CISI-PD Score from Visit 2 or before." SOURCE: Listing 16.2.6.5. (Same Shell as Table 14.2.1.1)

Mean Change from Baseline in CISI-PD Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Table 14.2.5.2 Evaluable Set

Programming Note: Add CISI-PD to abbreviations, SOURCE: Listing 16.2.6.5. (Same Shell as Table 14.2.1.2)

Table 14.2.5.3 Summary of Change from Baseline in CISI-PD Scores by Treatment Per Protocol Set

Programming Note: Parameters will be Total Score, Motor Signs, Disability, Motor Complications, and Cognitive Status. Visits will be Baseline (Visit 2), Week 8 (Visit 10), and Week 24 (Visit 19). Add CISI-PD to abbreviations. Add CISI-PD to abbreviations. Update footnote to read [1] The baseline value is the CISI-PD Score from Visit 2 or before." SOURCE: Listing 16,2.6.5. Update footnote to reflect Per Protocol Set. (Same Shell as Table 14.2.1.1)

Mean Change from Baseline in CISI-PD Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Per Protocol Set Table 14.2.5.4

Programming Note: Add CISI-PD to abbreviations. SOURCE: Listing 16,2,6.5. Update footnote to reflect Per Protocol Sel. Same Shell as Table 14.2.1.2

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Table 14.2.5.5 Summary of Change from Baseline in CISI-PD Scores by Treatment Complete Set

(Same Shell as Table 14.2.1.1)

Programming Note: Parameters will be Total Score, Motor Signs, Disability, Motor Complications, and Cognitive Status. Visits will be Baseline (Visit 2), Week 8 (Visit 10), and Week 24 (Visit 19). Add CISI-PD to abbreviations. Add CISI-PD to abbreviations. Update footnote to read "[1] The baseline value is the CISI-PD Score from Visit 2 or before." SOURCE: Listing 16.2.6.6. Update footnote to reflect Complete Set.

Table 14.2.5.6
Mean Change from Baseline in CISI-PD Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Complete Set

Same Shell as Table 14.2.1.2 Programming Note: Add CISI-PD to abbreviations. SOURCE: Listing 16.2.6.5. Update footnote to reflect Complete Set.



Summary of Change from Baseline in PDQ-39 Scores by Treatment Evaluable Set Table 14.2.6.1

Note: PDQ-39 is scored on a scale of 0-100 with lower scores indicating better health and high scores indicating more severe symptoms. [1] The baseline value is the PDQ-39 Score Programming Note: Parameters will be Total Score, Mobility, Activities of Daily Living, Emotional Well-Being, Stigma, Social Support, Cognitions, Communication, and Bodily Discomfort. Visits will be Baseline (Visit 2), Week 4 (Visit 9), Week 8 (Visit 10), Week 20 (Visit 18), and Week 24 (Visit 19), Add PDQ-39 to abbreviations. Update footnote to read (Same Shell as Table 14.2.1.1) from Visit 2 or before." SOURCE: Listing 16.2.6.6.

Mean Change from Baseline in PDQ-39 Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Table 14.2.6.2 Evaluable Set

Programming Note: Add PDQ-39 to abbreviations, SOURCE: Listing 16.2.6.6. (Same Shell as Table 14.2.1.2)

Summary of Change from Baseline in PDQ-39 Scores by Treatment Per Protocol Set Table 14.2.6.3

"Note: PDQ-39 is scored on a scale of 0-100 with lower scores indicating better health and high scores indicating more severe symptoms. [1] The baseline value is the PDQ-39 Score from Visit 2 or before." SOURCE: Listing 16.2.6.6. Update footnote to reflect Per Protocol Set. Programming Note: : Parameters will be Total Score, Mobility, Activities of Daily Living, Emotional Well-Being, Stigma, Social Support, Cognitions, Communication, and Bodily Discomfort. Visits will be Baseline (Visit 2), Week 4 (Visit 9), Week 8 (Visit 10), Week 20 (Visit 18), and Week 24 (Visit 19). Add PDQ-39 to abbreviations. Update footnote to read (Same Shell as Table 14.2.1.1)

Mean Change from Baseline in PDQ-39 Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Per Protocol Set Table 14.2.6.4

Programming Note: Add PDQ-39 to abbreviations. SOURCE: Listing 16.2.6.6. Update footnote to reflect Per Protocol Set. (Same Shell as Table 14,2,1,2)

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Table 14.2.6.5
Summary of Change from Baseline in PDQ-39 Scores by Treatment
Complete Set

complete set

Programming Note: : Parameters will be Total Score, Mobility, Activities of Daily Living, Emotional Well-Being, Stigma, Social Support, Cognitions, Communication, and Bodily Discomfort. Visits will be Baseline (Visit 2), Week 4 (Visit 10), Week 20 (Visit 16), and Week 24 (Visit 19). Add PDQ-39 to abbreviations. Update footnote to read "Note: PDQ-39 is scored on a scale of 0-100 with lower scores indicating better health and high scores indicating more severe symptoms. [1] The baseline value is the PDQ-39 Score from Visit 2 or before." SOURCE: Listing 16.2.6.6. Update footnote to reflect Complete Set. (Same Shell as Table 14.2.1.1)

Table 14.2.6.6
Mean Change from Baseline in PDQ-39 Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Complete Set

(Same Shell as Table 14,2.1.2)
Programming Note: Add PDQ-39 to abbreviations.SOURCE: Listing 16.2.6.6. Update footnote to reflect Complete Set.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



| Study Visit<br>Category | Placebo (N=XX) | GRF6021 |
|-------------------------|------------------|-------------|
| Paralline (4) | | (ox-si) |
| Daseline [1] | | |
| S to tellession | XX (XX.X%) | (%X:X%) |
| D-10 Mild depression | XX (XX.X%) | XX (XX:X%) |
| 11 + Severe depression | (%X.X%) | XX (XX X%) |
| Week 8 (Visit 10) | | |
| 0-4 No depression | (%XXXX)XX | (%X XX) XX |
| 5-10 Mild depression | XX XXX XX | (%X XX) XX |
| 11 + Severe depression | XX (XX.X%) | XX (XX.X%) |
| Week 20 (Visit 18) | | |
| 0-4 No depression | (%X XX) XX | 176X XX/ XX |
| 5-10 Mild depression | (%X XX) XX | (%X XX) XX |
| 11 + Severe depression | (marine Armonia) | forward to |

Abbreviation: GDS-15 = Geriatric Depression Scale-15.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized treatment.

[1] The baseline value is the SDS-15 assessment from Visit 2 or before.

SOURCE: Listing 16.2.6.7

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Table 14.2.7.2

Summary of Change from Baseline in GDS-15 Total Score by Treatment

Evaluable Set

Evaluable set

"Note: Each item is recorded as yes or no which is assigned a numeric value of 1 or 0, respectively. The final score is the tally of the number of depressive answers with the following scores indicating depression: [1] The baseline value is the PDQ-39 Score from Visit 2 Programming Note: Parameter will be Total Score Visits will be Baseline (Visit 2), Week 8 (Visit 10), and Week 20 (Visit 18). Add GDS-15 to abbreviations. Update footnote to read (Same Shell as Table 14.2.1.1) or before. "SOURCE: Listing 16.2.6.7.

Table 14.2.7.3

Mean Change from Baseline in GDS-15 Total Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Evaluable Set

(Same Shell as Table 14.2.1.2)

Programming Note: Add GDS-15 to abbreviations. SOURCE: Listing 16.2.6.7.

Table 14.2.7.4

Summary of GDS-15 Categories by Study Visit and Treatment
Per Protocol Set
Same Shell as Table 14.2.7.1

Programming Note: Add GDS-15 to abbreviations. Update footnote to reflect Per Protocol Set. SOURCE: Listing 16.2.6.7.

Table 14.2.7.5
Summary of Change from Baseline in GDS-15 Total Score by Treatment
Per Protocol Set

Same Shell as Table 14,2,1,1

Programming Note: Parameter will be Total Score Visits will be Baseline (Visit 2), Week 8 (Visit 10), and Week 20 (Visit 18). Add GDS-15 to abbreviations. Update footnote to read "Note: Each item is recorded as yes or no which is assigned a numeric value of 1 or 0, respectively. The final score is the tally of the number of depression answers with the following scores indicating depression: 0-4 No depression, 5-10 Suggestive of a mild depression 11 + Suggestive of severe depression. [1] The baseline value is the PDQ-39 Score from Visit 2 or before." SOURCE: Listing 16.2.6.7. Update tootnote to reflect Per Protocol Set.



Mean Change from Baseline in GDS-15 Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Per Protocol Set Table 14.2.7.6

(Same Shell as Table 14.2.1.2)
Programming Note: Add GDS-15 to abbreviations. SOURCE: Listing 16.2.6.7.

Summary of GDS-15 Categories by Study Visit and Treatment Complete Set Table 14.2.7.7

Same Shell as Table 14,2.7.1

Programming Note: Add GDS-15 to abbreviations. Update footnote to reflect Per Protocol Set. SOURCE: Listing 16.2.6.7.

Table 14.2.7.8
Summary of Change from Baseline in GDS-15 Total Score by Treatment Complete Set

Programming Note: Parameter will be Total Score Visits will be Baseline (Visit 2), Week 8 (Visit 10), and Week 20 (Visit 18). Add GDS-15 to abbreviations. Update footnote to read "Note: Each item is recorded as yes or no which is assigned a numeric value of 1 or 0, respectively. The final score is the fally of the number of depression sationed an unmeric value of 1 or 0, respectively. The final score is the raily of the number of depression, 5-10 Suggestive of a mild depression 11 + Suggestive of severe depression. [1] The baseline value is the PDQ-39 Score from Visit 2 or before." SOURCE: Listing 16.2.6.7. Update footnote to reflect Per Protocol Set. Same Shell as Table 14.2.1.1

Mean Change from Baseline in GDS-15 Total Score by Study Visit and Treatment Tabulation of Fitted Summary Statistics from ANCOVA Complete Set Table 14.2.7.9

Programming Note: Add GDS-15 to abbreviations, SOURCE: Listing 16.2.6.7. (Same Shell as Table 14.2.1.2)

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Table 14.2.8.1 Summary of Change from Baseline in dCDT Score by Treatment Evaluable Set

the second second second second

(Same Shell as Table 14.2.1.1)

Programming Note: Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 16), and Week 20 (Visit 18). Add dCDT to abbreviations. Update footnote to read "[1] The baseline value is the dCDT Score from Visit 2 or before." SOURCE: Listing 16.2.6.8.

Table 14.2.8.2
Mean Change from Baseline in dCDT Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Evaluable Set

(Same Shell as Table 14.2.1.2)
Programming Note: Add dCDT to abbreviations. SOURCE: Listing 16.2.6.8.

Table 14.2.8.3

Summary of Change from Baseline in dCDT Score by Treatment

Per Protocol Set

(Same Shell as Table 14.2.1.1)
Programming Note: Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 16), and Week 20 (Visit 18). Add dCDT to abbreviations. Update footnote to read "[1] The baseline value is the dCDT Score from Visit 2 or before." SOURCE: Listing 16.2.6.8.

Table 14.2.8.4
Mean Change from Baseline in dCDT Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Per Protocol Set

(Same Shell as Table 14.2.1.2)

Programming Note: Paramter will be dCDT total score. Add dCDT to abbreviations. SOURCE: Listing 16.2.6.8.



Table 14.2.8.5 Summary of Change from Baseline in dCDT Score by Treatment Complete Set

(Same Shell as Table 14.2.1.1)
Programming Note: Visits will be Baseline (Visit 2), Week 1 (Visit 8), Week 8 (Visit 10), Week 13 (Visit 16), and Week 20 (Visit 18). Add dCDT to abbreviations. Update footnote to read "[1] The baseline value is the dCDT Score from Visit 2 or before." SOURCE: Listing 16.2.6.8.

Table 14.2.8.6
Mean Change from Baseline in dCDT Score by Study Visit and Treatment
Tabulation of Fitted Summary Statistics from ANCOVA
Complete Set

(Same Shell as Table 14.2.1.2)
Programming Note: Paramter will be dCDT total score. Add dCDT to abbreviations. SOURCE: Listing 16.2.6.8.





| Study Visit | Placebo | GRF6021 |
|------------------------|------------|------------|
| Statistic | (N=XX) | (N=XX) |
| Baseline [1] | | |
| Within normal limits | XX (XX.X%) | (%X:XX) |
| Indeterminate | (%X'XX) | (%X XX) XX |
| Outside normal limits | (%X:XX) XX | XX (XX.X%) |
| Unanalyzable | (%X.X%) | XX (XX.X%) |
| Week 1 (Visit 8) | | |
| Within normal limits | (%X'XX) XX | XX (XX.X%) |
| Indeterminate | XX (XX:X%) | XX (XX.X%) |
| Outside normal limits. | XX (XX.X%) | XX (XX X%) |
| Unanalyzable | (XX.X%) | XX (XX.X%) |
| Week 8 (Visit 10) | | |
| Within normal limits | (%X:XX) XX | XX (XX.X%) |
| Indeterminate | XX (XX.X%) | XX (XX.X%) |
| Outside normal limits | XX (XX.X%) | XX (XX.X%) |
| Unanalyzable | XX (XX.X%) | XX (XX.X%) |

### Continue for other visits.

Abbreviation: dCDT = Digital clock drawing test.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized treatment.

[1] The baseline value is the dCDT Score from Visit 2 or before.

SOURCE: Listing 16.2.6.8



Table 14.2.8.8
dCDT Classification by Study Visit and Treatment
Per Protocol Set

(Same shell as Table 14.2.8.7)
Programming Note: Update footnote to reflect Per Protocol Set

Table 14.2.8.9
dCDT Classification by Study Visit and Treatment Treatment
Complete Set

(Same shell as Table 14.2.8.7)
Programming Note: Update footnote to reflect Complete Set





| Calegory | (XX=N) | (N=XX) |
|---------------------------------|-------------|------------|
| Presence of MRI Abnormalities | | |
| | XX (XX.X%) | XX (XX X%) |
| | XX (XX.X%) | XX (XX.X%) |
| Nonevaluable | XX (XX:X%) | XX (XX.X%) |
| Abnormalities Present | | |
| Cerebral edema | XX (XX.X%) | XX (XX.X%) |
| Abnormality Primary Location | | |
| Right frontal | (%X:XX) | (%X XX) XX |
| Right temporal, non hippocampal | XX (XX.X%) | (%X:XX) XX |
| Right parietal | XX (XX.X%) | (%X:XX) |
| Right occipital | (%XXX) | (%X:XX) XX |
| Abnormality Status | | |
| Present | (%X XX) XX | (%X:XX) XX |
| Presence is questionable | (%X XX) XX | %X XXX XX |
| Abnormality Sequence | | |
| 3014 | XX (XX.X%) | (%X:XX) XX |
| FLAIR | XX (XX.X%) | XX (XX.X%) |
| 72* | XX (XX.X%) | XX (XX.X%) |
| 72 | XX (XX:X%) | XX (XX.X%) |
| | XX (XX:X%) | (%X:X%) |
| Other | XX (XX:X%) | (%X XX) XX |
| Microhemorrhage | (%X'XX) | (%X:XX) XX |
| Abnormality Primary Location | | |
| Right frontal | XX (XX.X%) | (%X:XX) XX |
| Abnormality Status | | |
| Present | XX (XX.X%) | XX (XX:X%) |
| Presence is questionable | XX (XX.X%) | XX XXX XX |
| Abnormality Sequence | | |
| 3071 | XX (XX X%) | (%X'XX) XX |
| | 100 000 000 | 200 |

Abbreviations: MRI = magnetic resonance imaging; PD = Parkinson's Disease.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized treatment..

SOURCE: Listing 16.2.6.10

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



## Table 14.2.9.1 (cont.) Screening MRI Results by Study Visit and Treatment Evaluable Set

| VISIC Screening | | | |
|---|---|---|---|
| Test<br>Category | Placebo<br>(N=XX) | GRF6021<br>(N=XX) | |
| | | | ľ |
| White matter disease present | | | |
| No lesions (including symmetrical, well-defined caps or bands) | XX (XX.X%) | XX (XX.X%) | |
| Focal lesions | XX (XX.X%) | XX (XX.X%) | |
| Beginning confluence of lesions | XX (XX.X%) | (%XXXX)XX | |
| Diffuse involvement of entire region, with or without involvement of U-fibers | XX (XX.X%) | (%XXXX)XX | |
| Non Evaluable | XX (XX.X%) | XX (XX.X%) | |
| Potential alternative diagnosis to PD | | | |
| Yes | XX (XX.X%) | (%XXXX)XX | |
| No | XX (XX,X%) | (%X XX) XX | |
| Nonevaluable | XX (XX.X%) | XX (XX.X%) | |

Abbreviations: MRI = magnetic resonance imaging; PD = Parkinson's Disease.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized treatment. SOURCE: Listing 16.2.6.10 Programming Note: Continue for Visit 16 for subjects who consented to additional MRI. Only categories with at least 1 subject should be presented for the following tests: Abnormalities Present, Abnormality Primary Location, and Abnormality Sequence.

Subarachnoid haemomhage; Intraventricular haemomhage; Stroke involving a major vascular territory; Lacunar infarct (10-15 mm); Cortical infarct: Other infarct: Cerebral confusion; Encephaloras ≥ 1 cm in diameter; Meningioma > 1 cm in diameter; Arachnoid cyst ≥ 1 cm in diameter; Other space occupying lesion or Brain tumor; Other. Potential abnormalities are: Cerebral edema, Microhemormage, Microhemormage (>1cm); Superficial siderosis; Subdural hemormage/hematoma; Epidural haemormage;

Potential Abnormality primary locations are: Right frontal; Right temporal, non hippocampal; Right occipital; Right occipital; Right chippocampus; Right cerebellum; Mid-brain; Medulla; Left temporal, non hippocampal; Left parietal; Left occipital; Left chippocampus; Left cerebellum; Hydrocephalus; Pons; Deep grey matter structures; Ventricular system; All brain; Other.

Potential abnormality sequences are: DT1; FLAIR; T2\*, T2; DWI; Other

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Table 14.2.9.2
Screening Safety MRI Results by Study Visit and Treatment
Per Protocol Set

(Same shell as Table 14.2.9.1)

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



Volumetric MRI Results by Study Visit and Treatment Evaluable Set Table 14.2.9.3

Test: Volume (mm3), Visit: Screening

| 7 | | |
|--------------------|---------------|--------------|
| Location | | |
| Laterality | Placebo | GRF6021 |
| Statistic | (N=XX) | (X=XX) |
| Whole Brain | | |
| Bilateral | | |
| u u | × | XX |
| Mean (SD) | (XXXX (XXXXX) | (XX XX) X XX |
| Median | XXX | XXX |
| Min, Max | XX, XX | XX, XX |
| Lateral Ventricles | | |
| Bilateral | | |
| | × | XX |
| Mean (SD) | (XX XX) XXX | (XX XX) X XX |
| Median | XXX | XXX |
| Min, Max | XX, XX | XX, XX |
| Intracranial | | |
| Bilateral | | |
| • | × | XX |
| Mean (SD) | (XX XX) X XX | XX XX/ X XX |
| Median | XXX | XXX |
| Min, Max | XX, XX | XX,XX |
| Cortical | | |
| Left | | |
| T. | × | ×× |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XXX | XXX |
| Min, Max | XX, XX | XX, XX |
| Right | | |
| u u | XX | × |

Abbreviations: MRI = magnetic resonance imaging.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized treatment.

SOURCE: Listing 16.2.6.11

Thickness (mm) and Cerebral Cortex Thickness Average Change (mm). Locations will be Cortical (left, right, bilateral), Mayo (bilateral), Prefrontal Lobe (left, right, bilateral), Superior Temporal Lobe (left, right, bilateral), Interior Parietal Lobe (left, right, bilateral), Interior Parietal Lobe (left, right, bilateral), Interior Parietal Lobe (left, right, bilateral), Precuneus (left, right, bilateral), Isthmuscingulate (left, right, bilateral), Entorhinal Cortex (left, right, bilateral), Repeat table for Test: Atrophy (mm³). Locations Programming note: For Visit: Screening, Additional locations for Test: Volume (mm³) will be Hippocampus (left, right, bilateral). Repeat table for Test: Cerebral Cortex Average

will be the same as Test: Volume with the exception of Intracranial.
Repeat table for Visit: Week 13 (Visit 16).

AD-ST-33.05 Effective date, 22-Jan-2018

Version 4.0 | Date 17-Aug-2020 | AD-PR-109.01 Effective date: 26-Jun-2017

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



| Loiseac | | |
|-----------------------------------------|--------------|----------------|
| TOO | edesce D | GBER031 |
| Laterality | (N=XX) | (XX=N) |
| Claimic | | |
| Frontal Lobe | | |
| Left | X | × |
| | (A) A) A A) | 100 V V V V |
| Mean (SD) | (VV'VV) | (۷۷.۷۷) |
| Median | XX.X | XXX |
| Min, Max | XX XX | XX.XX |
| Right | | 3 |
| | × | × |
| Mean (SD) | XX,X (XX,XX) | (XX XX) XXX |
| Median | XXX | XXX |
| Min, Max | XX, XX | XX, XX |
| Bilateral | | |
| | × | × |
| Mean (SD) | XXXX (XXXXX) | (XXXX (XXXXX) |
| Median | XXX | XXX |
| Min, Max | XX, XX | XX, XX |
| Cingulate Cortex | | |
| Left | 2 | 3 |
| u u | X | X |
| Mean (SD) | XX.X (XX.XX) | (XX XX (XX XX) |
| Median | XXX | XXX |
| Min. Max | ××× | XX XX |

Abbreviations; ASL = arterial-spin labeling; MRI = magnetic resonance imaging.

Note: Percentages are n/Number of subjects in the Evaluable Set\*100. Subjects are summarized by randomized freatment. Cerebral blood flow measurements are presented in mL/100g/min. SOURCE: Listing 16.2.6.12 Programming note: For Visit: Screening, Additional locations will be Frontal lobe, Cingulate cortex, Parietal lobe, Temporal lobe, Occipital lobe, Striatum, Cerebellum, Thalamus, Pallidum, Substantia nigra, Hippocampus. Left, Right, and Bilateral sides will be present for all.
Repeat table for Visit: Week 13 (Visit 16).





| | Placebo | GRF6021 | Overall |
|---|---|---|---|
| Category | (N=XX)<br>(%) u | (N=XX)<br>n (%) | (N=XX) |
| Subjects with at least 1 TEAE | THE STATE AND | | |
| 11 (Percentage, %)<br>95% CI for percentage<br>Difference in percentage<br>95% CI for difference in percentage<br>P Value [1] | XX. (XX. X%)<br>XX. X%, XX. X% | XX (XX.X%) XX.X%, XX.X% XX.X% XX.X% XX.X% XXXXX | XX.X%, XX.X%) |
| Subjects with an SAE n (Percentage, %) 95% CI for percentage Difference in percentage 95% CI for difference in percentage | XX (XX.X%)<br>XX (XX.X%)<br>XX.X%, XX.X% | XX (XX.X%)<br>XX (XX.X%)<br>XX.X%, XX.X%<br>XX.X%, XX.X%<br>XX.X%, XX.X%<br>XX.XXX | XX (XX.X%)<br>XX (XX.X%)<br>XX.XX, XX.X% |

Abbreviations: AESI = adverse event of special interest; CI = confidence interval; CRF = case report form; TEAE = treatment emergent adverse event; SAE = serious adverse

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received,

AEs were coded using MedDRA version 21.0. A TEAE is any AE that occurs after the time of treatment with the study agent. This will include any AE with onset prior to time of treatment with study agent and increased severity after the treatment administration. AESts are TEAEs that are of special interest as defined by the protocol and are only recorded if the PI considers them as Adverse Events.

[1] P value from Chi-square test.
[2] Related TEAEs are those marked as Possibly Related or Definitely Related on the CRF. SOURCE: Listing 16.2.7.1

Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan, Sponsor Alkahest, Inc.



| Category | Placebo<br>(N=XX)<br>n (%) | GRF6021<br>(N=XX)<br>π (%) | Overall<br>(N=XX)<br>n (%) |
|---|---|---|---|
| Maximum Severity of TEAE Mild Moderate Severe | XX (XX.X%) XX (XX.X%) XX | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X.XX) XX (%X.X%) XX (%X.XX) XX |
| Subjects with a Related TEAE [2] | XX (XX.X%) | (%X:XX) XX | (%X XX) XX |
| Subjects with a TEAE Leading to Discontinuation of Study Drug (CRF) Subjects with a TEAE Leading to Discontinuation of Study Drug (Derived) | (%X XX) XX | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Subjects with an AE leading to Death | XX (XX.X%) | XX (XX.X%) | (%X'XX) XX |
| Subjects with an AESI | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AESI = adverse event of special interest; CI = confidence interval; CRF = case report form; TEAE = treatment emergent adverse event; SAE = serious adverse

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received.

treatment with study agent and increased severity after the treatment administration. AESIs are TEAEs that are of special interest as defined by the protocol and are only recorded if the PI considers them as Adverse Event, and the AE occurred between the start of AEs were coded using MedDRA version 21.0. A TEAE is any AE that occurs after the time of treatment with the study agent. This will include any AE with onset prior to time of the first infusion in Period 1 through the final infusion in Period 2, the derived action taken was set to 'study drug withdrawn' regardless of what was indicated on the CRF since treatment is administered during two distinct periods and not on a continuous basis.

[1] P value from Chi-square test.
[2] Related TEAEs are those marked as Possibly Related or Definitely Related on the CRF. SOURCE: Listing 16.2.7.1

Programming note: If Fisher's exact test is used, update footnote [1] accordingly.



Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment Table 14.3.1.2 Safety Set

| System Organ Class | Placebo | GRF6021 | Overall |
|-------------------------------|------------|------------|------------|
| Preferred Term | (XX=N) | (N=XX) | (N=XX) |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| System Organ Class 1 | XX (XX.X%) | (%X'XX) XX | XX (XX X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX:X%) | (%X XX) XX |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | (%X XX) XX |
| Preferred Term 3 | (XX.XX) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX XXX XX |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | (%XXXXXXX |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | (%XXXX) |
| Preferred Term 3 | XX (XX:X%) | XX (XX.X%) | XX (XXXX) |

Abbreviations: PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received.

AEs were coded using MedDRA version 21.0. A TEAE is any AE that occurs after the time of treatment with the study agent. This will include any AE with onset prior to time of treatment with study agent and increased severity after the treatment administration. Subjects are counted once for each SOC and once for each PT. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.7.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote.



Table 14.3.1.3 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Treatment Safety Set

| System Organ Class | Placebo | GRF6021 | Over |
|---|---|---|---|
| Preferred Term<br>Maximum Severity | (N=XX)<br>(%) u | (N=XX)<br>n (%) | (%) u |
| Subjects with at least 1 TEAE | (%X'XX) | (%X.XX) XX | XX (XX.X%) |
| Any Event (Total)<br>Mild | (%X'XX) XX | XX (XX.X%) | XX (XX.X) |
| Moderate | XX (XX.X%) | XX (XX.X%) | (%XXX)XX |
| Severe | (%X'XX) XX | (%X:XX) XX | 6XXXX) |
| System Organ Class 1<br>Any Event (Total) | | | |
| Mild | (%XXX) XX | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | (%X.XX) | XX XXX XX |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | | | |
| PJIW | XX (XX:X%) | (%X:XX) XX | XX (XX.X%) |

Note: Percentages are in/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. AEs were coded using MedDRA version 21.0. A TEAE is any AE that occurs after the time of treatment with the study agent. This will include any AE with onset prior to time of treatment with study agent and increased severity after the treatment administration. Subjects are counted once for each SOC and once for each PT. The severity shown is the greatest severity reported for a particular subject (Severe > Moderate > Mild). AEs with a missing severity were counted as Severe. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.7.1 Abbreviations: PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event.

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote.





Table 14.3.1.4 Incidence of Treatment Emergent Adverse Events by Relationship, SOC, PT, and Treatment Safety Set

| System Organ Class | Placebo | GRF6021 | Overall |
|---|---|---|---|
| Preferred Term<br>Maximum Severity | (N=XX)<br>n (%) | (N=XX)<br>n (%) | (N=XX)<br>n (%) |
| Subjects with at least 1 TEAE | XX (XX.X%) | (%X XX) XX | (%X'XX) XX |
| Any Event (Total)<br>Related<br>Not Related | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (%XXX)<br>XX (XXXX) |
| System Organ Class 1<br>Any Event (Total)<br>Related<br>Not Related | (%X.XX)<br>XX (XX.X%) | (%XXX) XX<br>(%XXX) XX | (%XXX) XX |
| Preferred Term 1<br>Related<br>Not Related | XX (XX.X%)<br>XX (XX.X%) | (%XXX) XX<br>XX (XX.X%) | (%X.XX) XX |

AE that occurs after the time of treatment with the study agent. This will include any AE with onset prior to time of treatment with study agent and increased severity after the treatment administration. Subjects are counted once for each SOC and once for each PT. Subjects are classified according to the closest relationship if the subject reported one or more events. Related TEAEs are those marked as Possibly Related or Definitely Related on the CRF. AEs with a missing relationship will be considered related for this summary. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. AEs were coded using MedDRA version 21.0 A TEAE is any Abbreviations: CRF = case report form; PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event. SOURCE: Listing 16.2.7.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



Table 14.3.2.1 Incidence of Adverse Events Leading to Withdrawal by SOC, PT, and Treatment Safety Set

Same shell as Table 14.3.1.2

Programming note: AEs leading to withdrawal will be based on derived action taken in this table. The following should be added to Note: If the reason for discontinuation entered on the study completion CRF was "Adverse Event" and the AE occurred between the start of the first infusion in Period 1 through the final infusion in Period 2, the derived action taken was set to 'study drug withdrawn' regardless of what was indicated on the CRF since treatment is administered during two distinct periods and not on a continuous basis.

Table 14.3.2.2 Incidence of Serious Adverse Events by SOC, PT, and Treatment. Safety Set.

Same shell as Table 14.3.1.2

Programming note: Add SAE to abbreviations.

Table 14.3.2.3 Incidence of Adverse Events of Special Interest by SOC, PT, and Treatment Safety Set

Same shell as Table 14.3,1.2

Programming note: Add AESI to abbreviations.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



Table 14.3.2.4 Incidence of Adverse Events with Terms Associated with Blood Pressure Changes by Infusion Period, SOC, PT, and Treatment Safety Set

| System Organ Class<br>Preferred Term | (X)<br>(X)<br>(%) | (%) u | (N=XX) |
|---|---|---|---|
| Any Occurrence. System Organ Class 1 Preferred Term 1 (Blood Pressure Decreased) Preferred Term 2 (Blood Pressure Increased) | (%X.XX) XX | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| System Organ Class 2<br>Preferred Term 1 (Blood Pressure Decreased)<br>Preferred Term 2 (Blood Pressure Increased) | XX (XX.X%)<br>XX (XX.X%) | (%XXX) XX<br>(%XXX) XX | XX (XX.X%) XX (%X.X%) |
| Starting During Infusion Period 1 System Organ Class 1 Preferred Term 1 (Blood Pressure Decreased) Preferred Term 2 (Blood Pressure Increased) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (%XXX) XX |
| System Organ Class 2<br>Preferred Term 1 (Blood Pressure Decreased)<br>Preferred Term 2 (Blood Pressure Increased) | (%X.XX) XX (%X.XX) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%) XX |
| Starting After Infusion Period 1 System Organ Class 1 Preferred Term 1 (Blood Pressure Decreased) Preferred Term 2 (Blood Pressure Increased) | XX (XX.X%)<br>XX (XX.X%) | (%XXXX)<br>XX (XXXXX) | (%XXXX)XX |

Abbreviations: CRF = case report form; PT = preferred term; SOC = system organ class; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. AEs were coded using MedDRA version 21.0 A TEAE is any AE that occurs after the time of treatment with the study agent. This will include any AE with onset prior to time of freatment with study agent and increased severity after the treatment administration. Subjects are counted once for each SOC and once for each PT. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.7.1

Programming Note: Continue for "Starting During Infusion Period 2" and "Starting After Infusion Period 2."



Table 14.3.3.1
Listing of Adverse Events Leading to Study Drug Discontinuation
All Subjects

| Subject<br>ID | Subject Treatment<br>ID [1] | TEAE/<br>Intercurrent | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date (Study<br>Day) Start Time /<br>End Date (Study<br>Day) End Time | Severity/<br>Relationship | Outcome/<br>Study Drug Action<br>Taken (CRF)/<br>Other Action Taken | Derived<br>Action<br>Taken | Serious?/<br>Criteria Met | AESI?<br>[2] |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX XXXXXX XXXXX | XXXX | DOXXXXXXXXXXXXXX | DDMMMYYYY (XX)<br>HH:MM/ | AXXXXXXXXX | XXXXXXXXXXXXX | XXXXX | /XX | XXX |
| | | | ACCOCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCC | DDMMMYYYY<br>(XX) HH:MM | XXXXXXXX | XXXXXXXXXXXXXXXX | XXXXX | XXXXXXXXXX | |
| | | | XXXXXXXXXXX | | | xxxxxxxxxxxx | XXXXX | | |
| | xxxx xxxxx | XXXX | XXXXXXXXXX | DDMMMYYYY (XX) | XXXXXXXXXXX | XXXXXXXXXXXX | XXXXX | × | XX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ongoing | XXXXXXXX | | | | |
| | XXXXXX | XXXXXXXXX | XXXXXXXXX | DDMMMYYYY (XX) | XXXXXXXX | XXXXXXXXXXXXX | XXXXX | × | XXX |
| | | | XXXXXXXXXXXX | DDMMMYYYY(XX)<br>HH:MM | XXXXXXX | | | | |
| | | | XXXXXXXXXXXXXXXXXX | | | | | | |

Abbreviation: TEAE = treatment emergent adverse event.

between the start of the first infusion in Period 1 through the final infusion in Period 2, the derived action taken will be set to 'study drug withdrawn' regardless of what was indicated Note: Study day is calculated relative to the date of first dose. AEs were coded using MedDRA version 21.0. A TEAE is any AE that occurs after the time of treatment with the study reported after consent has been signed and prior to initial dosing. If the reason for discontinuation entered on the study completion CRF was "Adverse Event" and the AE occurred agent. This will include any AE with onset prior to time of treatment with study agent and increased severity after the treatment administration. An intercurrent AE is an AE that is on the CRF since treatment is administered during two distinct periods and not on a continuous basis.

[1] Treatment is based on treatment received.
[2] AESIs are TEAEs that are of special interest as defined by the protocol and are only recorded if the PI considers them as Adverse Events.

"Other" with the text. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported."

SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in foolnote. AESI will be Yes or No Programming note: "Other Action Taken" will be either None, Medication Required, Relevant Procedure, or Other, if specify text is needed, concatenate "Relevant Procedure," or

Table 14,3,3,2 Listing of Serious Adverse Events Safety Set

(Same shell as Table 14,3,3,1)

Table 14.3.3.3 Listing of Deaths Safety Set

(Same shell as Table 14.3.3.1)

Table 14.3.3.4 Listing of Adverse Events of Special Interest Safety Set

(Same shell as Table 14.3.3.1)

Programming note: Include column which contains Higher Level Term, Higher Level Group Term, and Lower Level Term next to the SOC/PT/Verbatim Term column.

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



## Parameter: XXXXXXXXX

| Study Visit | SPIA<br>(=N) | (XX) | 25 | (N=XX) | 5 🖔 | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | Observed | CFB | Observed | CFB |
| Baseline [1] | ** | 3 | ** | ** | * | * |
| Mean (SD) | XXXX XXXX | XX.X (XX.XX) | XXX XXXXX | XX.X (XX.XX) | XXXX XXXXX | XXXX XXX |
| Median | XXX | XXX | XX.X | XX | XXX | XXX |
| Min, Max | XX, XX | XX XX | XX, XX | XX, XX | XX, XX | XX'XX |
| Week 1 (Visit 6) | 3 | | 3 | | | |
| | × | × | × | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XXXX (XXXXX) | XX.X (XX.XX) | (XXXX) XXX | XX.X (XX.XX) |
| Median | XXX | XXX | ××× | XXX | XXX | XXX |
| Min Max | XX XX | XX. XX | XX XX | XX XX | XX XX | XX. XX |

Continue for other parameters and visits. Sort alphabetically by parameter.

Abbreviation: CFB = change from baseline.

Note: Subjects are summarized by treatment received.

[1] The baseline value for each variable is the value recorded prior to the first dose. SOURCE: Listing 16.2.8.1.1

Programming Note: Comprehensive labs will be performed at screening/Visit 1, Visit 6, Visit 8, Visit 14, Visit 16, Visit 17, and upon exit/Visit 19.



Table 14.3.5.1.2
Shift from Baseline in Hematology Laboratory Results by Study Visit and Treatment.
Safety Set

Parameter: XXXXXXX

| | | Baseline [ | le [1] | |
|---|---|---|---|---|
| | | Placebo (N=XX | N=XX) | |
| Study Visit<br>Category | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) |
| Week 1 (Visit 6) | | | | |
| Low | (%X'XX) XX | (%X:XX) XX | (%X XX) XX | V70A AAU AA |
| Normal | XX (XX.X%) | (%XXXX)XX | (%X XX) XX | (8/ YXX) XX |
| High | (%X'XX) | (%X XX) XX | (%X XX) XX | (8/2:22) |
| Missing | XX (XX.X%) | (%XXX)XX | XX (XX,X%) | XX (XX.X%) |
| Week 1 (Visit 8) | | | | |
| Low | (%X'XX) XX | (%XXX)XX | (%X XX) XX | 1764 444 44 |
| Normal | XX (XX.X%) | XX (XX.X%) | (%X XX) XX | (%X XX) XX |
| High | XX (XX.X%) | XX (XX.X%) | (%X XX) XX | (SIX XX XX |
| Missing | XX (XX.X%) | XX (XXXX)) | (%X:XX) XX | XX (XX.X%) |

Continue for other parameters and treatment groups (GRF6021 and overall). Sort alphabetically by parameter.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. [1] The baseline value for each variable is the value recorded prior to the first dose.

SOURCE: Listing 16.2.8.1.1

Programming Note: Comprehensive labs will be performed at screening/Visit 1, Visit 6, Visit 9, Visit 14, Visit 16, Visit 17, and upon exit/Visit 19. If table width allows, all three treatment groups (Placebo, GRF6021, Overall) may be displayed in one table with the four shift categories (low, normal, high, missing) underneath (i.e. 12 columns) rather than repeating the table for each treatment group (4 columns).

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Table 14.3.5.2.1
Summary of Serum Chemistry Laboratory Results by Study Visit and Treatment Safety Set

(Same shell as Table 14.3,5,1,1; SOURCE: Listing 16.2,8,1,2)

Table 14.3.5.2.2
Shift from Baseline in Serum Chemistry Laboratory Results by Study Visit and Treatment Safety Set

(Same shell as Table 14.3.5.1.2; SOURCE: Listing 16.2.8.1.2)

Table 14.3.5.3.1 Summary of Quantitative Urinalysis Laboratory Results by Study Visit and Treatment Safety Set

(Same shell as Table 14.3.5.1.1; SOURCE: Listing 16.2.8.1.3)

Table 14.3.5.3.2
Shift from Baseline in Quantitative Urinalysis Laboratory Results by Study Visit and Treatment
Safety Set

(Same shell as Table 14.3.5.1.2; SOURCE: Listing 16.2.8.1.3)





Table 14.3.5.3.3

Summary of Qualitative Urinalysis Laboratory Results by Study Visit and Treatment Safety Set

| Į |
|-------------|
| 5 |
| ξ |
| ξ |
| ? |
| e<br>e<br>e |
| a |
| 7 |

| tion No. | Placebo | GRF6021 | Overall |
|------------------|------------|------------|------------|
| Catanon | (VY-N) | (YY=N) | (N=XX) |
| Calcyony | (%) II | n (%) | (%) تا |
| Baseline [1] | | | |
| Category 1 | (%XXX) XX | XX (XX.X%) | (%XXXXXXX |
| Category 2 | (%XXX) | XX (XX.X%) | XX XXX XX |
| Category 3 | XX (XX.X%) | (%X.XX) XX | XX (XX.X%) |
| Week 1 (Visit 6) | | | |
| Category 1 | (%XXXX) | XX (XX.X%) | (%X XX) XX |
| Category 2 | XX (XX.X%) | XX (XX.X%) | (%XXXX) |
| Category 3 | XX (XX.X%) | XX (XX.X%) | (%X'XX) |

Continue for other parameters. Sort alphabetically by parameter.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. [1] The baseline value for each variable is the value recorded prior to the first dose. SOURCE: Listing 16.2.8.1.3

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Table 14.3.5.4.1 Summary of Coagulation Laboratory Results by Study Visit and Treatment Safety Set

(Same shell as Table 14.3.5.1.1; SOURCE: Listing 16.2.8.1.5)

Table 14.3.5.4.2
Shift from Baseline in Coagulation Laboratory Results by Study Visit and Treatment
Safety Set

(Same shell as Table 14.3.5.1.2; SOURCE: Listing 16.2.8.1.5)



Table 14.3.6.1.1 Summary of Vital Signs by Study Visit and Treatment Safety Set (Same shell as Table 14.3.5.1.1; visits include Visit 1- Visit 19; parameters Include Temperature (C), Respiration Rate (breaths per min), Sitting Systolic Blood Pressure (mmHg), Heart Rate (bpm), Sitting Diastolic Blood Pressure (mmHg), Standing Diastolic Blood Pressure (mmHg), and Supine Diastolic Blood Pressure (mmHg), Weight (kg); SOURCE: Listing 16.2.8.2.)

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



Table 14.3.6.1.2 Summary of Blood Pressures of Special Interest by Study Visit and Treatment Safety Set

| Study Visit Category Baseline [1] SBP > 180mmHg SBP < 90 mmHg SBP < 90 mmHg | Placebo | PODLOGO | - |
|---|---|---|---|
| Study Visit Category Saseline [1] SBP > 180mmHg SBP < 90 mmHg SBP < 90 mmHg | 10.00 | GREDUZI | Overall |
| Calegory Saseline [1] SBP > 180mmHg SBP < 200 mmHg SBP < 90 mmHg | (N=XX) | (XX=N) | (N=XX) |
| Saseline [1] SBP > 180mmHg SBP > 200 mmHg SBP < 90 mmHg | n (%) | u (%) | u (%) |
| SBP > 180mmHg SBP > 200 mmHg SBP < 90 mmHg | The state of the s | | |
| SBP > 200 mmHg SBP < 90 mmHg | XX (XX.X%) | XX (XX.X%) | (%X'XX) XX |
| SBP < 90 mmHg | XX (XX.X%) | XX (XX.X%) | (%XXX) |
| MOIST THE CHICK OF THE PERSON AS A PERSON | XX (XX X%) | XX (XX.X%) | XX (XX XX) |
| Veek (Visit 3) 15 Mily DURING INTUSION | | | |
| SBP > 180mmHg | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SBP > 200 mmHg | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SBP < 90 mmHg | XX (XX.X%) | XX (XX.X%) | (%X XX) XX |
| CFB≥30% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 1 (Visit 3) 30 MIN DURING INFUSION | | | |
| SBP > 180mmHg | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SBP > 200 mmHg | (%X:XX) XX | XX (XX.X%) | (%X:XX) |
| SBP < 90 mmHg | XX (XX.X%) | XX (XX.X%) | (%XXX) XX |
| CFB≥30% | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX |

# Continue for other parameters. Sort alphabetically by parameter.

Abbreviations: CFB = change from baseline; DBP = diastolic blood pressure; SBP = systolic blood pressure.

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. Blood pressures of special interest are as follows: seated systolic blood pressure > 180 mmHg, seated systolic blood pressure > 200 mmHg, seated systolic blood pressure > 120 mmHg, seated diastolic blood pressure > 120 mmHg, seated diastolic blood pressure < 50 mmHg, or a change of ≥ 30% from baseline in seated systolic and/or seated diastolic blood pressure.

[1] The baseline value for each variable is the value recorded prior to the first dose.

SOURCE: Listing 16.2.8.1.3

Programming Note: Parameters Include: Sitting Systolic Blood Pressure (mmHg) and Sitting Diastolic Blood Pressure, the categories with be: DBP < 50, DBP > 110, DBP > 120, and at post baseline visits, CFB ≥ 30%

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



Table 14.3.6.2.1
Summary of 12-Lead Electrocardiogram by Study Visit and Treatment
Safety Set

(Same shell as Table 14.3.5.1.1; visits include Visit 1, Visit 11, and Visit 15; parameters include HR, QT, QTcF; SOURCE: Listing 16.2.8.3)

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Table 14.3.6.2.2
Summary of 12-Lead Electrocardiogram Interpretation by Study Visit and Treatment
Safety Set

| Study Visit<br>Category | // γ/2000 (N=XX)<br>π (%) | СКР6021<br>(N=XX)<br>п (%) | (N=XX) |
|---|---|---|---|
| Baseline [1] Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X.XX) XX<br>(%X.XX) XX<br>(%X.XX) XX |
| Week 1 (VIsit 7) Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | (%XXX)XX<br>(%XXX)XX<br>(%XXX) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X.XX) XX (%X.X%) XX (%X.X%) XX |
| Week 13 (Visit 11)<br>Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | (%X`XX) XX<br>(%X`XX) XX<br>(%X`XX) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X'XX) XX<br>(%X'XX) XX |
| Week 13 (Visit 15)<br>Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X,XX)<br>XX (XX,X%)<br>XX (XX,X%) | (%XXX) XX<br>(%XXX) XX<br>(%XXX) XX |

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received, [1] The baseline value for each variable is the value recorded prior to the first dose SOURCE: Listing 16.2.8.3


Table 14.3.6.3 Summary of Sheehan-Suicidality Tracking Scale (S-STS) by Study Visit and Treatment Safety Set

| Study Visit | Plac<br>(N=) | Placebo<br>(N=XX) | 88<br>8 | GRF6021<br>(N=XX) | WO N | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | Observed | CFB | Observed | CFB |
| Visit 1 | | | | | | |
| | × | X | X | × | ×× | XX |
| Mean (SD) | XXXX (XXXXX) | XX.X (XX.XX) | XXXX XXXX | XX XXX XXX | XX XXX XXX | XX XXX XXX |
| Median | XXX | XXX | XXX | ××× | XXX | XXX |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX,XX |
| Week 1 (Visit 3) | | | | | | |
| n | × | × | X | × | × | XX |
| Mean (SD) | XX.X (XX.XX) | XXXX (XXXXX) | XXXXXXXX | XX XX XXX | XX XXX XXX | XX XX XXX |
| Median | XX.X | XXX | XXX | XXX | ××× | XXX |
| Min, Max | XX.XX | XX, XX | XX, XX | XX, XX | XX,XX | XX, XX |
| Week 1 (Visit 7) | | | | | | |
| | × | × | × | ×× | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | (XX.XX) XXX | XXXXXXXX | (XX XX) X XX | XX XXX XXX |
| Median | XXX | XXX | XXX | XXX | ××× | XXX |
| Min, Max | XX,XX | XX.XX | XX.XX | XXXX | ×××× | XX XX |

Abbreviation: CFB = change from baseline. Note: Subjects are summarized by treatment received. SOURCE: Listing 16.2.8.5

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Table 14.3.6.4
Summary of Concomitant Medications by ATC Class Level 4, PT, and Treatment Safety Set

| ATC Class Level 4<br>Preferred Term (ATC Class Level 5) | Placebo<br>(N=XX)<br>n (%) | GRF6021<br>(N=XX)<br>n (%) | Overall (N=XX) n (%) |
|---|---|---|---|
| Subjects with at least 1 Concomitant Medication | (%X.XX) XX | XX (XX.X%) | (%X:XX) XX |
| ATC Class 1 | (%X'XX)XX | XX (XX.X%) | XX (XX,X%) |
| Preferred Term 1 | (%XXXXXXX | XX (XX:X%) | (%XXX) |
| Preferred Term 2 | (%XXX)XX | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | (%X XX) XX | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | XX (XX.X%) | (%XXX)XX | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety Set\*100. Subjects are summarized by treatment received. Medications were coded using WHODrug version March 2018. Concomitant medications are all medications that were continuing or starting after first dose of study drug. A medication with a missing start date and a stop date that is either missing or on or after the treatment start date will be considered as concomitant. Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by PT within ATC, and then alphabetically. Subjects were counted only once for each ATC and PT. Abbreviations: ATC = Anatomical Therapeutic Chemical; PT = Preferred Term. SOURCE: Listing 16.2.8.6

Programming note: ATC & PT text should be in proper case in table, as shown in the shell. Ensure correct WHODrug version is printed in footnote.



## 4.3. Planned Listing Shells

Listing 16.2.1 Subject Disposition All Subjects

| Subject<br>ID | Treatment [1] | Subject Status | Date of Completion/Discontinuation (Study Day) | Reason for<br>Discontinuation | Date of Last Dose of Study Was the Blind Broken Drug (Study Day) for This Subject? | Was the Blind Broken<br>for This Subject? |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXXXX | Completed | DDMMMYYYY (XX) | | DDMMMYYYY (XX) | |
| XXXXXX | XXXXXX | Early<br>Terminated | DDMMMYYYY (XX) | | DDMMMYYYY (XX) | |
| XXXXXX | XXXXXX | Did not<br>complete per<br>protocol Due<br>to COVID-19 | DDMMMYYYY (XX) | | DDMMMYYYY (XX) | |
| XXXXXX | XXXXXXX | XXXXXX | DDMMMYYYY (X) | XXXXXXX: XXXXXX | DDMMMYYYY (X) | XXX |
| XXXXXX | XXXXXX | XXXXXX | DDMMMYYYY (XX) | XXXXXXXXXXXXXXX DDMMMYYYY (XX) | DDMMMYYYY (XX) | XXX; XXXXXX; |

Abbreviation: COVID-19 = novel coronavirus disease 2019; CRF = case report form; NA = not applicable.

Note: Study day is calculated relative to the date of first dose. A subject is considered to not have completed the study per protocol due to COVID-19 if they had any missing visits that affected treatment administration or collection of end of study efficacy assessments due to COVID-19. If a subject did not complete the study per protocol due to COVID-19, this category supersedes their study status on the study completion CRF. [1] Treatment is based on treatment received. Programming Note: If reason for early termination is Other, concatenate the specify text as follows: "Other, XXXXXXXXX". If reason for early termination is lost to follow-up, concatenate with date of last contact and comments as follows: "Lost to follow-up, date of last contact: DDMMMYYYY; XXXXX". If reason for early termination is death, concatenate with date the blind was broken and with cause of death and date of death as follows: "Lost to follow-up; XXXXX; date of death: DDMMMYYYY". If blind was broken, concatenate with date the blind was broken and reason for breaking the blind as follows: "Yes; DDMMMYYY; XXXXX"

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,

Listing 16.2.2.1 Inclusion and Exclusion Criteria Not Met All Subjects

| Subject ID | Treatment [1] | Date of Informed Consent<br>(Study Day) | nt Visit | Visit Date<br>(Study Day) | All Inclusion<br>Criteria Met?<br>[2] | Any Exclusion<br>Criteria Met?<br>[3] |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | DDMMMYYYY<br>(-X) | Screening | DDMMNYYYY (-X) | | |
| | | DDMMMYYYYY (-X) | Baseline | | No: 02 | Ŷ. |
| XXXXXX | XXXXXX | DDMMMYYYYY (-X) | Screening | DDMMNYYYY (-X) | No: 02 | N<br>N |
| | | DDMMMYYYY<br>(-X) | Baseline | | Yes | Yes: 03 |
| XXXXXX | XXXXXX | DDMMMYYYY<br>(-X) | Screening | DDMMMYYYY (-X) | Yes | ON. |
| | | DDMMMYYYY<br>(-X) | Baseline | | Yes | ON. |

Note: Study day is calculated relative to the date of first dose. [1] Treatment is based on treatment received. IE Description:

Inclusion Criteria:

02 = Diagnosis of clinically established or clinically probable PD according to MDS-PD criteria with at least 1 year of PD symptoms. Exclusion Criteria:

03 = Prior hypersensitivity reaction to any human blood product or any IV infusion; any clinically significant known drug allergy.

Programming note: If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown in the example. If no criteria are present for a column, remove the [2] and/or [3] from the column header.



Listing 16.2.2.2
Protocol Deviations
All Subjects

| Subject ID | Treatment [1] | Event Type | Violation | Description | Excluded from Per Protocol Set? |
|---|---|---|---|---|---|
| XXXXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MAJOR | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ×× |
| XXXXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MINOR | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ×× |
| XXXXXX | XXXXXXXXXX | XXXXXXXXXXXX | MAJOR | XXXXXXXXXXXXXXXXXXXXX | XXX |

[1] Treatment is based on treatment received.

Programming note: The structure of this listing may change depending on the information in the protocol deviations file.

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 Statistical Analysis Plan, PCN Number ALKA7951 Listing 16.2.3 Analysis Sets All Subjects

| Reason(s) for Exclusion | Per Protocol; Had a major protocol deviation | | Evaluable; Did not receive at least 4 of the 10 planned doses |
|---|---|---|---|
| Per Protocol<br>[5] | No | Yes | ON. |
| Evaluable<br>[4] | Yes | Yes | No |
| Safety<br>[3] | Yes | Yes | No. |
| [2] | Yes | Yes | No |
| Treatment [1] | XXXXXX | XXXXXXXX | XXXXXX |
| Subject ID | XXXXXXX | XXXXXX | XXXXXXX |

[1] Treatment is based on treatment received.

[2] The ITT Set includes all randomized participants.
[3] The Safety Set includes all subjects who received at least one dose of study product.
[4] The Evaluable Set includes all subjects who receive at least 5 of the 10 planned doses and complete through Visit 8.
[5] The Per Protocol Set is a subset of the Evaluable Set comprised of subjects who receive all 10 planned doses, who complete Visit 18 and Visit 19 in window, and who have no protocol deviations that could affect the assessment of efficacy.
[6] The Complete Set is a subset of the PP Set comprised of subjects who did not have any changes to any of the following concomitant medications preferred terms reported at any time on study. Dopaminergic agents (e.g. Rotigotine [Neupro Patch], Duopa Pump, Sinemet [Carbidopa, Levodopa], Carbidopa, Rytary), Pregabalin (Lyrica), Amandadine, Antipsychotics (e.g. Pimavansenin Tartate [Nuplazid], Clozapine, Quetiapine Furnarate [Seroquel]), or benzodiazepines (e.g. Alprazolam). This includes those that were stable per protocol prior to first dose and either changed dose or stopped on study as well as those that began on study.

Programming note: Concatenate all reasons for exclusion with a semi-colon.





Listing 16.2.4.1
Demographics and Baseline Characteristics
All Subjects

| XXXXXXX XXXXXXX XXXXXXX No DDMMMYYYY XX XXXXXXXX XXXXXXX XXXXXX XXXXXXX XXXX | Subject ID | Subject ID Treatment [1] | Sex | Child-Bearing<br>Potential? | Date of<br>Birth | Age<br>(years) | Ethnicity | Race | Weight (kg) | Height (cm) | ApoE<br>Genotype | Disease<br>Duration<br>(years) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX | XXXXXX | XXXX | | DDMMMYYY | × | XXXXXXX | XXXXXXX | XXX | XXX | XXX | xxx |
| XXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXXXX XXXXXXXXXX XXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX | XXXXXX | XXXXXX | No | DDMMMYYY | × | XXXXXXX | - 33 | XXX | XXX | XXX | XXX |
| XXXXXXX XXXXXX XX XXXXXXX XXX XXXXXXX XXXX | XXXXXX | XXXXXX | XXXXXX | Yes | DDMMMYYY | × | XXXXXXX | XXXXXX | XXX | XXX | XXX | XXX |
| XXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXX | XXXXXX | XXXXXX | XXXX | | DDMMMYYY | × | XXXXXXX | XXXXX | XXX | XXX | XXX | XXX |
| XXXXXX XXXXXX XXXXXX XXXXXX XXXXXXX XXXX | XXXXXX | XXXXXX | XXXXXX | No | DDMMMYYY | × | XXXXXXX | XXXXXX | XXX | XXX | XXX | XXX |
| | XXXXXX | XXXXXX | XXXX | | DDMMMYYY | X | XXXXXXX | XXXXXX | xxx | XXX | XXX | XXX |

Abbreviations: ApoE = Apolipoprotein E; PD = Parkinson's disease.

Note: Height and weight are the values at Screening. Disease duration = [Enrollment date – PD onset date (as recorded on the Medical History CRF) + 1] / 365.25.[1] Treatment is based on treatment received.

Programming Note: If race is other, concatenate "Other:" with specify text. If subject has multiple races, concatenate them.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Listing 16.2.4.2.1 Medical History All Subjects

| + | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day)/ |
|---|---|---|
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| | XXXXXXXXXX<br>XXXXXXXXXXXXXXXXXXXXXXXXXXX | MMMYYYY (X)/<br>Ongoing |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MMMYYYY (X)/<br>Ongoing |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYYY (X) |

Note: Study day is calculated relative to the date of first dose, Medical history was coded using MedDRA version 21.0. Only subjects with medical history recorded are listed. [1] Treatment is based on treatment received.

Programming note: SOC & PT text should be in proper case in table, as shown in the shell.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



| Subject Treatment | Was Family Medical History | Family | Living/Deceased | Age at Time of | Cause of | History of Neurological | Neurological |
|---|---|---|---|---|---|---|---|
| ID [1] | Collected? | Member | | Death | Death | Disease? | Disease(s) |
| xxxxx xxxx | Yes/No | XXXXXXX | XXXXXX | × | XXXXXXX | Yes/No | XXXXXXXX |

[1] Treatment is based on treatment received.

Programming Note: If not collected, concatenate reason. If neugological disease is 'other' concatenate specify field.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



| | | Social | | | Exercise | Exercise/Activity Level | | |
|---|---|---|---|---|---|---|---|---|
| Treatment [1] | Was Social<br>History/Exercise-<br>Activity Level<br>Assessed? | Describe<br>Where You<br>Currently<br>Live | Bike for 10<br>Minutes<br>Consistently? | How Many<br>Days Do You<br>Bike for 10<br>Minutes? | Time spent Walking or Bicycling for Travel on a Typical Day (minutes) | Do Any Sports,<br>Fitness, or<br>Recreational<br>Activitites? | How Many Days Per<br>Week Do You Do<br>Sports, Fitenss, or<br>Recreational<br>Activities? | Time Spent<br>doing<br>Sports,<br>Fitenss, or<br>Recreational<br>Activities on<br>a Typical<br>Day<br>(Minutes |
| XXXXXX | Yes/No | XXXXXXX | Yes/No | X | XXX | Yes/No | × | XXX |

[1] Treatment is based on treatment received.

Programming Note: If not done, concatenate explanation. If neugological disease is 'other' concatenate specify field. If 'Other' concatenate specify field.



Listing 16.2.4.3
Alcohol, Tobacco, and Substance Use All Subjects

| | | Topac | Tobacco Smoking History | fistory | | | Alcohol | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment [1] | Smoking<br>History/# Years<br>Smoked | # per day:<br>Cigarettes/<br>Cigars/<br>Pipes | If Ex-Smoker,<br>Date Stopped<br>(Study Day) | Have you consumed alcohol in the past 6 months? | # drinks containing alcohol do you have on a typical day when you are drinking? | How often do<br>you have 6+<br>drinks on 1<br>occasion? | Did<br>anybody<br>ever tell you<br>when you<br>were<br>younger<br>that you<br>had a<br>problem<br>with | Have you ever had problems related to consuming alcohol? | Subject used illicit substances (including marijuana) in the past? / Describe |
| × | XXXXXXXX | XX XXXXXXXXXX XXXXXX XXXXX XXXXX XXXX XXXX | × ×× | DDMMMYYYYY (X) | ×× | × | XXXXXX | XX | XX | × |
| * | XXXXXXXXX | XXXXXXXXX XXXXXXXXX XXXXXXXX | | DDMMMYYYY<br>(X) | XX | × | XXXXXX | XX | ××× | × |

Note: Study day is calculated relative to the date of first dose. [1] Treatment is based on treatment received.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



Was Assessment Completed?

Treatment [1]

Subject

XXXXXX

| Date/Time of Assessment (Study Day) | Parameter | Result |
|---|---|---|
| DDMMMYYYYY HH:MM (XX) | Abrupt onset of dementia | |
| | | Present/Absent |
| | Stepwise deterioration of dementia | |
| | | <b>Present/Absent</b> |
| | Somatic complaints | |
| | | Present/Absent |
| | Emotional inconfinence | |
| | | Present/Absent |
| | History or presence of hypertension | |
| | | Present/Absent |
| | History of strokes | |
| | | Present/Absent |
| | Focal neurological symptoms | |
| | | Present/Absent |
| | Focal neurological signs (on | Present/Absent |
| | examination) | |
| | Total Soora | XX |

Abbreviation: MHIS = Modified Hachinski Ischaemia Scale.
Note: Study day is calculated relative to the date of first dose. MHIS is collected at Screening Visit 1 only.
[1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason.



Listing 16.2.4.5 Hoehn and Yahr Scale All Subjects

| Subject ID | Treatment [1] | Was Assessment Completed? | Date/Time of Assessment<br>(Study Day) | Hoehn and Yahr Stage |
|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | DDMMMYYYY/ HH:MM (XX) | X: XXXXXX |

Note: Study day is calculated relative to the date of first dose. Hoehn and Yahr is collected at Screening Visit 1 only. [1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concalenate reason. For stage, include the number and text.



Listing 16,2,5 Drug Infusion All Subjects

| Pump Manufacturer and model | XXXXXXX |
|-----------------------------------------|--------------------------|
| Actual Volume<br>Administered<br>(mL) | XX |
| Rate<br>(mL/hour) | × |
| Date/Time of<br>Infusion<br>(Study Day) | DDMMMYYYY/<br>HH:MM (XX) |
| Time Point | Time X |
| Was the Infusion<br>Performed? | XXX |
| Treatment [1] | XXXXXX XXXXXX |
| Subject<br>ID | XXXXXX |

Note: Study day is calculated relative to the date of first dose. [1] Treatment is based on treatment received.



Listing 16.2.6.1 MoCA All Subjects

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

| 11 | Was Assessment Completed? | MoCA Version | Date/Time of Assessment<br>(Study Day) | Parameter | Result |
|---|---|---|---|---|---|
| | XXX | xx | DDMMMYYYY HH:MM (XX) | Visuospatial/Executive | × |
| | | | | Naming | × |
| | | | | Memory | × |
| | | | | Attention | × |
| | | | | Language | × |
| | | | | Abstraction | × |
| | | | | Delayed Recall | × |
| | | | | Orientation | × |
| | | | | Add 1 point if <=12 years of | × |
| | | | | education | |
| | | | | Total Score | × |

Abbreviation: MoCA = Montreal Cognitive Assessment.

Note: Study day is calculated relative to the date of first dose.

MoCA Total score = sum of Individual item scores, with a range from 0 to 30.

[1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason.

Page 123 of 156

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



| | | | | | | Letter | etter Fluency | cy | Cate | Category Fluency | ucy | Category Switching | tching | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ubject | Treatment<br>[1] | Was<br>Assessment<br>Completed? | Date/Time of<br>Assessment<br>(Study Day) | Interval | jų, | Ą | S | Total<br>Correct | Animals | Boys'<br>Names | Total | Fruits/Furniture | Total<br>Correct<br>Score | Total<br>Correct<br>Score |
| XXXXX | XXXXXX | XXX | DDMMMYYYY/ | 1-15 seconds | × | × | × | × | XXX | XXX | × | XXX | × | × |
| | | | THE WINE (AA) | 16-30 seconds | × | × | × | | XX | XXX | | XXX | | |
| | | | | 31-45 seconds | × | × | × | | XXX | XXX | | XXX | | |
| | | | | 46-60 seconds | × | × | X | | XXX | XX | | XXX | | |

Abbreviation: D-KEFS = Delis-Kaplan Executive Function System.

Note: Study day is calculated relative to the date of first dose.

D-KEFS Letter Fluency Total Correct Score = sum of F+A+S correct responses from 1-15, 16-30, 31-46, and 46-60 seconds.

D-KEFS Category Fluency Total Correct Score = sum of Animals and Boys' Names correct responses from 1-15, 16-30, 31-46, and 46-60 seconds.

D-KEFS Category Switching Total Correct Score = sum of Fruits/Furniture correct responses from 1-15, 16-30, 31-46, and 46-60 seconds.

D-KEFS Category Switching Total Correct Score = sum of Fruits/Furniture correct ategory Fluency Total Correct Score.

[1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason. Total scores over the minute will be displayed on the first row only.



Listing 16,2,6,3 MDS-UPDRS All Subjects

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Statistical Analysis Plan,

| 0 | Subject ID Treatment [1] | Was Assessment<br>Completed? | Primary Source<br>of Information | Date/Time of<br>Assessment<br>(Study Day) | Parameter | Result |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXX | × | XXXXXXXX | DDMMMYYYY/ HH:MM (XX) | Cognitive impairment Hallucinations and psychosis Depressed mood Anxious mood Apathy Features of dopamine dysregulation syndrome Sleep problems Daytime sleepiness Pain and other sensations Uninary problems Constipation problems Lightheadedness on standing Fatigue | XXXX = XXXXX = XXXXXX |

Abbreviation: MDS-UPDRS = Movement Disorder Society's Unified Parkinson's Disease Rating Scale. Note: Study day is calculated relative to the date of first dose.

MDS-UPDRS Part 1 score = sum of all Part 1 individual item scores. Part 1 consists of 13 items on a scale of 0 (normal) to 4 (severe), so the Part 1 score ranges from 0 to 52.

MDS-UPDRS Part 2 score = sum of all Part 2 individual item scores. Part 2 consists of 13 items on a scale of 0 (normal) to 4 (severe), so the Part 2 score ranges from 0 to 52.

MDS-UPDRS Part 3 score = sum of all Part 3 individual item scores. Part 3 consists of 22 33 items on a scale of 0 (normal) to-4 (severe), so the Part 3 score ranges from 0 to 132.

MDS-UPDRS Parts 1-3 total score = sum of Part 1, Part 2, and Part 3 scores. If any of the individual part scores are missing, the total score will be set to missing. [1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason. Continue for Parts 2 and 3. Insert a blank row and add a row for Total Score after Part 3.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Listing 16.2.6.4 SE-ADL Scale All Subjects

| Sublant ID | Treatment [4] | Was Assassment Completed? | Date/Time of Assessment | agnetional of layer |
|---|---|---|---|---|
| onnicor In | Heavillein [4] | Was Assessment Completes: | (for form) | |
| XXXXXXX | XXXXXX | XXX | DDMMMYYYY HH:MM (XX) | XXXXXXXXXXX = %XXX |

Abbreviation: SE-ADL = Schwab & England Activities of Daily Living. Note: Study day is calculated relative to the date of first dose. [1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason.



| Subject ID | Treatment [1] | Was Assessment Completed? | Date/Time of Assessment<br>(Study Day) | Asessment | Result |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | DDMMMYYYY/HH:MM (XX) | Motor Signs<br>Disability<br>Motor Commissions | XXXXXXX = X |
| | | | | (dyskinesia and fluctuations) | X = XXXXXXX |
| | | | | Cognitive Status CISI-PD Total Score | XXXXXXXX |

Abbreviation: CISI-PD = Clinical Impression of Severity Index-Parkinson's Disease.

Note: Study day is calculated relative to the date of first dose.

CISI-PD total score = sum of the four individual item scores (motor signs, disability, motor complications, and cognitive status) rated 0 (not at all) to 6 (very severe or disabled), with a range of 0 to 24.

[1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason.

oremier

Protocol Number ALK6021-201 Statistical Analysis Plan, PCN Number ALKA7951 Sponsor Alkahest, Inc.

Listing 16.2.6.6 All Subjects PDQ-39

| Result | XXXX | XXXX | XXX | XXX |
|---|---|---|---|---|
| Question | Had difficulty doing the leisure activities you would like to do? Had difficulty looking after your home, for example, housework, cooking or | yardwork?<br>Had difficulty carrying grocery bags?<br>Had problems walking half a mile? | Mobility subscale score | Total score |
| Domain | Mobility | | | |
| Date/Time of Assessment<br>(Study Day) | DDMMMYYYY/ HH:MM (XX) | | | |
| Was Assessment<br>Completed? | XX | | | |
| Treatment [1] | XXXXXX | | | |
| Subject ID | XXXXXX | | | |

Abbreviation: PDQ-39 = Parkinson's Disease Quality of Life Questionnaire-39.

Note: Study day is calculated relative to the date of first dose

PDQ.39 Mobility subscore = sum of 10 items in the Mobility domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.

PDQ-39 Activities of Daily Living subscore = sum of 6 items in the Activities of Daily Living domain (converted from a range of 0 inever) to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.

PDQ-39 Emotional Well-Being subscore = sum of 6 items in the Emotional Well-Being domain (converted from a range of 0 inever) to 4 [always/cannot do at all] to a range of 0 to

PDQ-39 Stigma subscore = sum of 4 items in the Stigma domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the 100), divided by the maximum possible score on the scale and multiplied by 100.

PDQ-39 Social Support subscore = sum of 3 items in the Social Support domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100. maximum possible score on the scale and multiplied by 100.

PDQ-39 Cognitions subscore = sum of 4 items in the Cognitions domain (converted from a range of 0 ferever) to 4 [always/cannot do at all] to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.

PDQ-39 Bodily Discomfort subscore = sum of 3 items in the Bodily Discomfort domain (converted from a range of 0 [never] to 4 [always/cannot do at all] to a range of 0 to 100), PDQ-39 Communication subscore = sum of 3 items in the Communication domain (converted from a range of 0 (never) to 4 (always/cannot do at all) to a range of 0 to 100), divided by the maximum possible score on the scale and multiplied by 100.

divided by the maximum possible score on the scale and multiplied by 100.

PDQ-39 Total score = mean of all of the PDQ-39 subscores.

Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason. After each question and answer is listed, list the Total score and the scores for the following subscales: Mobility, Activities of Dally Living, Emotional Well-Being, Stigma, Social Support, Cognitions, Communication, Bodily Discomfort.



Listing 16.2.6.7 GDS-15 All Subjects

| ubject ID | Subject ID Treatment [1] | Was Assessment Completed? | Date/Time of Assessment<br>(Study Day) | Question | Result |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | DDMMMYYYY/ HH:MM (XX) | Are you basically satisfied with your life? | × |
| | | | | Have you dropped many of your activities and interests? | × |
| | | | | Do you feel that your life is empty? | × |
| | | | | Do you often get bored? | × |
| | | | | Total Score | × |

Abbreviation: GDS-15 = Geriatric Depression Scale-15.

Note: Study day is calculated relative to the date of first dose.

GDS-15 Total score = sum of the 15 item questionnaire, with a range of 0 to 15. Each question is answered "yes" or "no". Question numbers 1, 5, 7, 11, 13 indicate presence of depression when answered negatively (no). One point is counted for each depressive answer. A score of 0-4 indicates no depression, a score of 5-10 is suggestive of a mild depression, and a score of 11 or more is suggestive of severe depression. [1] Treatment is based on treatment received.

Programming Note: If assessment was not completed, concatenate reason.





| Feature Result | | | | ck | ciency on XX | | omposite Scale XX |
|---|---|---|---|---|---|---|---|
| Cognitive Feature | Stroke Count Conformity on command clock | Total Time on command clock | Ink Length on command clock | Drawing Size on command clock | Drawing Process Efficiency on command clock | Noise on command clock | Drawing Efficiency Composite Scale |
| dCDT | XXXXXX | | | | | | |
| dDCT | XXX | | | | | | |
| Date/Time of Test<br>(Study Day) | DDMMMYYYY/ HH:MM (XX) | | | | | | |
| Handedness of Subject at Test<br>Time | XXXXXX | | | | | | |
| Treatment<br>[1] | XXXXXX | | | | | | |
| Subject<br>ID | XXXXXX | | | | | | |

Abbreviation: dCDT = Digital clock drawing test.

Note: Study day is calculated relative to the date of first dose.

[1] Treatment is based on treatment received.

Programming Note: Continue listing for simple motor, information processing, and spatial reasoning composite scales and cognitive features.



[1] Treatment is based on treatment received.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951



| Comments | XXXX |
|---|---|
| Potential<br>alternative<br>diagnosis to<br>PD? | Yes/<br>No/<br>Non-<br>evaluable/ |
| Is White Matter<br>Disease Present? | No lesions (including symmetrical, well- defined caps or bands)/ Focal lesions/ Beginning confluence of lesions/ Diffuse involvement of entire region, with or without Involvement of U- fibers / |
| Abnormality<br>Status | Present/<br>Presence is<br>questionable |
| Abnomality<br>Primary<br>Location | XXXXXXX |
| Abnormality<br>Slice<br>Number | XX |
| Abnormality<br>Sequence | 3DT1/<br>FLAIR/<br>T2*/<br>T2*/<br>DWI//<br>Other |
| Abnormality | XXXXXX |
| Presence of MRI<br>Abnormalities? | XXXXXX XXXXXX Yes/No/Nonevaluable XXXXXXX |
| Visit | XXXXX |
| Treatment<br>[1] | XXXXXX |
| Subject | XXXXX |

Non evaluable

Abbreviations: MRI = Magnetic Resonance Imaging; PD = Parkinson's Disease. [1] Treatment is based on treatment received.

Programming Note: If abnormality or abnormality primary location is 'Other' concatenate specify field with a semicolon in the cell.





| XXXXXX XXXXXX XXXXXX Volut | Test | n Laterality | Result (unit) |
|---|---|---|---|
| | Volume Whole Brain | ain Bilateral | XXX |
| | Lateral Ven | Lateral Ventricles Bilateral | XXX |
| | Intracrar | ital Bilateral | XX |
| | Cortice | II Left | XXX |
| | Cortice | d Right | XXX |
| | Cortica | ll Bilateral | XXX |
| | 1 | | |

Abbreviations: MRI = Magnetic Resonance Imaging. [1] Treatment is based on treatment received.

Programming Note: Include all location/lateriality/test results for all visits. Sort by visit, test, location.



| XXXXXXX XXXXXX CBF Frontal Lobe Left XX CBF Right XX CBF Right XX CBF Cingulate Cortex Left XX CBF Cingulate Cortex Left XX CBF CBF Right XX CBF Silateral XX | Subject ID | Treatment [1] | Visit | Test | Location | Laterality | Result (unit) |
|---|---|---|---|---|---|---|---|
| CBF Cingulate Cortex Left CBF Right CBF Bilateral | XXXXX | XXXXXX | XXXXX | 28.<br>28.<br>28.<br>28. | Frontal Lobe | Left<br>Right<br>Bilateral | ××× |
| | | | | <u>888</u> | Cingulate Cortex | Left<br>Right<br>Bilateral | XXX |

Abbreviations: ASL = arterial-spin labeling; CBF = cerebral blood flow, MRI = Magnetic Resonance Imaging.
[1] Treatment is based on treatment received.

Programming Note: Include all location/lateriality/test results for all visits. Sort by visit, test, location.

Listing 16.2.7.1 Adverse Events All Subjects

| Derived<br>on Action | ò | X AX XXXXX | | XXXXX | | XXXXXX XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX XXXXXX XX XXXXX XX XXXXX XX XX |
|---|---|---|---|---|---|---|---|---|
| Outcome/<br>Study Drug Action | 1.0 | 8 | | XXXXXXXXXXXXXXX | ^ | | | |
| | Severity/<br>Relationship | ~ | XXXXXXXX | | | × | × | × × |
| Start Date (Study<br>Day) Start Time / | End Date (Study<br>Day) End Time | DDMMMYYYY (XX) | DDMMMYYYY | WW HH-WW | (XX) HH:MM | DDMMMYYYYY (XX) | DDMMMYYYY (XX) HH:MM / Ongoing | DDMMMYYYY (XX) HH:MM / Ongoing DDMMMYYYY (XX) |
| System Organ Class/ | Preferred Tem/<br>Verbatim Term | XXXXXXXXXXXXXXXXX | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | XXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | TEAE/<br>Intercurrent | | | | | XXX | XXX | AXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXX |
| | Treatment<br>[1] | XXXX XXXXXX XXXXX | | | | XXXXX XXXXX | XXXXXX | XXXXX |
| | Subject | XXXXXX | | | | | | |

Abbreviation: CRF = case report form; TEAE = Treatment emergent adverse event.

Note: Study day is calculated relative to the date of first dose. AEs were coded using MedDRA version 21.0. A TEAE is any AE that occurs after the time of treatment with the study between the start of the first infusion in Period 1 through the final infusion in Period 2, the derived action taken will be set to 'study drug withdrawn' regardless of what was indicated reported after consent has been signed and prior to initial dosing. If the reason for discontinuation entered on the study completion CRF was "Adverse Event" and the AE occurred agent. This will include any AE with onset prior to time of treatment with study agent and increased severity after the treatment administration. An intercurrent AE is an AE that is on the CRF since treatment is administered during two distinct periods and not on a continuous basis. Treatment is based on treatment received.

[2] AESIs are TEAEs that are of special interest as defined by the protocol and are only recorded if the PI considers them as Adverse Events.

Programming note: "Other Action Taken" will be either None, Medication Required, Relevant Procedure, or Other, if specify text is needed, concatenate "Relevant Procedure:" or "Other." with the text. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote. AESI will be Yes or No



Listing 16.2.8.1.1 Clinical Laboratory Data: Hematology All Subjects

| Comments/Reason<br>Not Done | | | | | | | | | XX | |
|---|---|---|---|---|---|---|---|---|---|---|
| Com | | | | | | | | | XXXXXX | |
| Accession | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | | XXXXXXX |
| Reference<br>Range Flag | | | | XXX | | | | | | |
| Reference<br>Range [3] | XX-YY | XX-XX | XX - XX | XX-XX | XX-XX | XX-XX | XX-XX | XX-XX | | XX-XX |
| Change from<br>Baseline [2] | | X | × | × | × | × | × | × | | × |
| Standard<br>Results | × | × | × | × | × | × | × | × | QN | × |
| Date of Assessment<br>(Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | | DDMMMYYYY (X) |
| Parameter<br>(unit) | Red Blood<br>Cell Count | | | | | | | | | |
| Treatment<br>[1] | XXXXXXX | | | | | | | | | |
| Subject | XXXXXX | | | | | | | | | |

Abbreviations: A = abnormal; CS = clinically significant, H = high; L = low, ND = not done. Note: Study day is calculated relative to the date of first dose of study drug.

[1] Treatment is based on treatment received.

[2] Baseline is the Screening Visit 1.

[3] Reference range is used to identify potentially clinically significant laboratory values.

Programming note: update abbreviations to reflect actual data, If test was not done, set results to ND; make sure last column is populated accordingly

Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Statistical Analysis Plan,



Listing 16.2,8.1.2 Clinical Laboratory Data: Serum Chemistry All Subjects

(Same shell as Listing 16.2.8.1.1)

Listing 16.2.8.1.3 Clinical Laboratory Data: Urinalysis All Subjects

(Same shell as Listing 16.2.8.1.1; remove "(unit)" from 2"d column header)

ListIng 16.2.8.1.4
Clinical Laboratory Data: Urine Drug Screen and Pregnancy Tests
All Subjects

(Same shell as Listing 16.2.8.1.1; remove "(unit)" from 2nd column header; do not display Reference Range or Accession number columns)

Listing 16.2.8.1.5 Clinical Laboratory Data: Coagulation All Subjects

(Same shell as Listing 16.2.8.1.1)

Listing 16.2.8.1.6 Clinical Laboratory Data: Immunology All Subjects

(Same shell as Listing 16.2,8.1.1)

Listing 16.2.8.1.7 Clinical Laboratory Data: Serology All Subjects

(Same shell as Listing 16.2.8.1.1; remove "(unit)" from 2nd column header)

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951

Listing 16.2.8.2.1 Vital Signs All Subjects

| XXX | | | | |
|---|---|---|---|---|
| XXX | XXX | XXX | ND | XXX |
| XXX | | | | |
| × | × | × | Q | X |
| X | X | X | QN | × |
| XXX | XXX | XXX | QN | XXX |
| DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) |
| XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXXXX | | | | |
| | XXXXXX DDMMMYYYY (X) XX.X XX XX XXX | XXXXXX DDMMMYYYY (X) XX.X XX XX XX XXX XXX XXX XXX XXX XXX | XXXXXXX DDMMMYYYY (X) XX.X XX X | XXXXXXX DDMMMYYYYY (X) XXX XXX |

Subject ID

XXXXXX

Note: Study day is calculated relative to the date of first dose. Abnormal vital signs are as follows: Heart rate > 100 beats per minute, Temperature > 37.5°C or < 36.5°C, Respiration rate > 20 breaths per minute or < 12 breaths per minute.

[1] Treatment is based on treatment received. Abbreviation: ND = not done.

Programming Note: If a measurement is abnormal, place an asterisk (\*) next to the value in the cell.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951 Listing 16.2.8.2.2 Blood Pressure All Subjects

| | | | Date of | Standir<br>Pressure | Standing Blood<br>Pressure (mmHg) | Supine<br>Pressure | Supine Blood<br>Pressure (mmHg) | Sitting Blood<br>Pressure (mmHg) | Sitting Blood essure (mmHg) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment [1] | Study | Assessment<br>(Study Day) | Systolic | Diastolic | Systolic | Diastolic | Systolic | Diastolic | Abnormal? | BPS1? |
| XXXXXX | XXXXXX | XXXXXX | DDMMMYYYY (X) | XXX | × | XXX | × | XXX | × | XXX | XXX |
| | | XXXXXX | DDMMMYYYY (X) | XXX | × | XXX | × | XXX | × | | |
| | | XXXXXX | DDMMMYYYY (X) | XX | × | XX | × | XXX | × | | |
| | | XXXXXX | DDMMMYYYY (X) | QN | Q | Q | Q | N | Q | | |
| | | XXXXXX | DDMMMYYYY (X) | XXX | ×× | XX | × | XXX | × | | |

Note: Study day is calculated reliative to the date of first dose. Abnormal blood pressure vital signs are as follows: seated systolic blood pressure < 90 mmHg or > 110 mmHg, or incidence of offhostalic hypotension (a decrease in systolic blood pressure of > 20 mm Hg and/or a decrease in diastolic blood pressure of > 10 mm Hg between supine and standing). BPSIs are as follows: seated systolic blood pressure > 180 mmHg, seated systolic blood pressure > 100 mmHg, seated systolic blood pressure > 100 mmHg, seated systolic blood pressure > 100 mmHg, seated diastolic blood pressure > 100 mmHg, seated diastolic blood pressure > 110 mmHg, seated diastolic blood pressure > 100 mmHg, seated diastolic blood bressure > 100 mmHg Abbreviation: BPSI = blood pressure of special interest; ND = not done.

Programming Note: If a measurement is abnormal, place an asterisk (\*) next to the value in the cell.



Listing 16.2.8.3 12-Lead Electrocardiogram (ECG) Results All Subjects

| Subject ID | Treatment [1] | Was ECG Performed? | Date/Time of ECG<br>(Study Day) | Overall<br>Interpretation | Heart Rate<br>(bpm) | OT Interval<br>(msec) | QTcF Interval<br>(msec) |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | DDMMMYYYYI HH:MM XXXXXXX | xxxxxxx | XXX | XXX | XXX |
| | | × | DDMMMYYYY HH:MM XXXXXXXXXXX | XXXXXXXXXX | XXX | XXX | XXX |
| | | XXX | DDMMMYYYY/ HH:MM | XXXXXXXXX | XXX | XXX | XXX |
| | | XXX | DDMMMYYYY/ HH:MM | XXXXXX; XXXXX | XXX | XXX | XXX |
| | | XXX | DDMMMYYYY/ HH:MM | XXXXXXXXXX | XX | xxx | XXX |
| | | XX | DDMMMYYYY/ HH:MM | XXXXXXXXX | XXX | XXX | XXX |
| | | XXX | (XX) | | | | |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY/ HH:MM | XXXXXXXXXXXXX | XXX | XXX | XXX |
| | | XXX | DDMMMYYYY HH:MM (XX) | XXXXXXXXXXX | XXXX | XXXX | XXXX |

Abbreviation: ND = not done.

Note: Study day is calculated relative to the date of first dose.

[1] Treatment is based on treatment received.

Programming note: If ECG was not performed, concatenate with reason.

Statistical Analysis Plan, Sponsor Alkahest, Inc. Protocol Number ALK6021-201 PCN Number ALKA7951


premier



| Subject ID | Treatment [1] | Was Echocardiogram<br>Performed? | Date/Time of<br>Echocardiogram<br>(Study Day) | Cardiologist's<br>Interpretation | If Abnormal,<br>Describe |
|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | DDMMMYYYY | XXXXXXX | XXXXXXXXXXX |
| | | × | DDMMMYYYY | XXXXXXXXXX | |
| | | XXX | DDMMMYYYY/ | XXXXXXXXX | XXX |
| | | XXX | DDMMMYYYY | XXXXXXX | XXXXXXXXXX |
| | | XXX | DDMMMYYYY/ | XXXXXXXXXX | XXXXXXXXXX |
| | | XX | DDMMMYYYY/ | XXXXXXXX | |
| | | XXX | ND ON | | |
| XXXXXX | xxxxx | XXX | DDMMMYYYY | XXXXXXXXXXX | |
| | | xxx | DDMMMYYYY/<br>HH:MM (XX) | XXXXXXXXXX | XXXXXXXXX |

Abbreviation: ND = not done.

Note: Study day is calculated relative to the date of first dose.

[1] Treatment is based on treatment received.

Programming note: If Echocardiogram was not performed, concatenate with reason.



Listing 16.2.8.5.1 Physical Examination All Subjects

Subject

XXXXXX ₽

| Treatment<br>[1] | Was<br>Physical<br>Exam<br>performed? | Date/Time<br>Performed<br>(Study Day) | Body System | Result | Reason Not Done | If Abnormal, Describe |
|---|---|---|---|---|---|---|
| XXXXX | × | (X-) | General Appearance Skin Head and Neck Lymph Nodes Thyroid Musculoskeletal Extremeties Cardiovascular Lungs Abdomen Neurological | Normal<br>Abnormal, CS<br>Normal<br>Normal<br>Normal<br>Normal<br>Normal | | XXXXXXXX |

Abbreviations: CS = clinically significant; NCS = not clinically significant. Note: Study day is calculated relative to the date of first dose.

[1] Treatment is based on treatment received.

Programming Note: If Exam was not performed, concatenate reason.

Listing 16.2.8.5.2
Targeted Physical Examination
All Subjects

Same shell as Listing 16.2.8.4.1. Body Systems will be: Heart, Lungs, and Peripheral Edema.



Listing 16,2.8.6 S-STS All Subjects

| Treatment [1] | Was Questionnaire Collected? | Date I me Collected<br>(Study Day) | Total Scale Score |
|---|---|---|---|
| XXXXXX | XXX | DDMMMYYYY HH:MM (XX) | × |

Abbreviation: S-STS = Sheehan Suicidality Tracking Scale. Note: Study day is calculated relative to the date of first dose. [1] Treatment is based on treatment received.

Programming Note: If questionnaire was not collected, concatenate reason.



## Listing 16.2.8.7 Prior and Concomitant Medications All Subjects

| Route/<br>(unit) Frequency | AXXXXXXXX () | VVVVVVV | C | C |
|---|---|---|---|---|
| Dose (unit) | (xxx) xxx | | (xxx) xxx | (xxx) xxx |
| Start Date (Study Day)/<br>End Date (Study Day) | DDMMMYYYY (X)/ | DDMMMYYYY (X) | DDMMMYYYY (X)/<br>Ongoing | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| ATC Class (Level 4)/<br>Preferred Term (ATC Level 5)/<br>Verbatim Term | XXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Indication | XXXXXXXX | | XXXXXXX | XXXXXX |
| Taken Prior<br>to First Dose<br>of Study<br>Drug? | XXX | | × | XX |
| Subject ID Treatment [1] | XXXXXX | | | |
| Subject ID | XXXXXX | | | |

Abbreviation: ATC = anatomic therapeutic chemical; NA = Not applicable.

Note: Study day is calculated relative to the date of first dose. Medications were coded using WHO-DDE version March 2018.

[1] Treatment is based on treatment received.

Programming note: If Dose unit, Route or Frequency is Other, display other specify text only (le, do not display "Other: XXXXXX" but just "XXXXXXX"). Sort by subject, start date, end date, end date, ATC level 4 & PT. ATC & PT text should be in proper case in table, as shown in the shell. If ongoing, put "Ongoing" for end date.


## 14.4. Planned Figure Shells

Figure 14.2.1.1

Boxplots of MoCA Total Scores by Visit and Treatment

Evaluable Set



Programming notes: Each treatment group will be graphed using a different color. Boxplots will be displayed at each visit.

Reference Table: 14.2.1.1

SOURCE: Listing 16.2.6.1



Figure 14.2.1.2

Boxplots of MoCA Total Scores by Visit and Treatment

Per Protocol Set

Same Shell as Figure 14.2.1.1. Reference Table: 14.2.1.3. SOURCE: Listing 16,2.6.1.

Figure 14.2.2.1

Boxplots of D-KEFS Total Scores by Visit and Treatment
Evaluable Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.2.1. SOURCE: Listing 16.2.6.2.

Figure 14.2.2.2 Boxplots of D-KEFS Total Scores by Visit and Treatment Per Protocol Set Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.2.3. SOURCE: Listing 16.2.6.2.

Figure 14.2.3.1

Boxplots of MDS-UPDRS Parts 1-3 Scores by Visit and Treatment
Evaluable Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.3.1. SOURCE: Listing 16.2.6.3.

Figure 14.2.3.2

Boxplots of MDS-UPDRS Parts 1-3 Scores by Visit and Treatment
Per Protocol Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.3.3, SOURCE: Listing 16.2.6.3.



Figure 14.2.3.3

Boxplots of MDS-UPDRS Part 1 Scores by Visit and Treatment

Evaluable Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits, Reference Table: 14.2.3.1, SOURCE: Listing 16.2.6.3.

Figure 14,2,3,4
Boxplots of MDS-UPDRS Part 1 Scores by Visit and Treatment
Per Protocol Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table; 14.2.3.3. SOURCE: Listing 16.2.6.3.

Figure 14.2.3.5

Boxplots of MDS-UPDRS Part 2 Scores by Visit and Treatment
Evaluable Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.3.1. SOURCE: Listing 16.2.6.3.

Figure 14.2.3.6

Boxplots of MDS-UPDRS Part 2 Scores by Visit and Treatment

Per Protocol Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.3.3. SOURCE: Listing 16.2.6.3.

Figure 14.2.3.7

Boxplots of MDS-UPDRS Part 2 Scores by Visit and Treatment

Evaluable Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.3.1. SOURCE: Listing 16.2.6.3.

Figure 14.2.3.8

Boxplots of MDS-UPDRS Part 2 Scores by Visit and Treatment

Per Protocol Set

Same Shell as Figure 14.2.1.1. Update Y-axis to reflect appropriate score and update X-axis for the appropriate visits. Reference Table: 14.2.3.3. SOURCE: Listing 16.2.6.3.



Figure 14.3.1.1

Boxplots of Hematology Data by Parameter, Visit, and Treatment Safety Set

Y-axis: Parameter: XXXXXX (unit) X-axis: Week X (Visit X)

Programming notes: A separate graph will be produced for each parameter. Each treatment group will be graphed using a different color. Boxplots will be displayed at each visit. The appropriate visits will be displayed for each parameter. Reference Table: 14.3.5.1.1 SOURCE: Listing 16.2.8.1.2




premier

Figure 14.3.1.2

Boxplots of Serum Chemistry Laboratory Data by Parameter, Visit, and Treatment
Safety Set

(Same shell as Figure 14.3.1.1; Reference Table: 14.3.5.2.1; SOURCE: Listing 16.2.8.1.2)

Figure 14.3.1.3

Boxplots of Quantitative Urinalysis Laboratory Data by Parameter, Visit, and Treatment
Safety Set

(Same shell as Figure 14.3.1.1; Reference Table: 14.3.5.3.1; SOURCE: Listing 16.2.8.1.3)



Figure 14.3.2.1 Hematology: Mean (SD) by Parameter, Visit, and Treatment Safety Set

Y-axis: Parameter: XXXXXX (unit)

X-axis: Week X (Visit X)

Programming notes: A separate graph will be produced for each parameter. Each treatment group will be graphed using a different color and symbol. Use light blue for placebo and green for GRF6021, as in the boxplots above. Mean and 1 standard deviation will be plotted. The appropriate visits will be displayed for each parameter. Reference Table: 14.3.5.1.1 SOURCE: Listing 16.2.8.1.1



premier

(Same shell as Figure 14.3.2.1; Reference Table: 14.3.5.2.1; SOURCE: Listing 16.2.8.1.2) Figure 14.3.2.2 Serum Chemistry: Mean (SD) by Parameter, Visit, and Treatment Safety Set

Figure 14.3.2.3

Quantitative Urinalysis: Mean (SD) by Parameter, Visit, and Treatment
Safety Set

(Same shell as Figure 14.3.2.1; Reference Table: 14.3.5.3.1; SOURCE: Listing 16.2.8.1.3)

Figure 14.3.3.1
Vital Signs Data by Parameter, Visit, and Treatment
Safety Set

(Same shell as Figure 14.3.1.1; Reference Table: 14.3.6.1; SOURCE: Listing 16.2.8.2.1 and 16.2.8.2.2)

Figure 14.3.3.2

Vital Signs: Mean (SD) by Parameter, Visit, and Treatment.
Safety Set
Same shell as Figure 14.3.2.1; Reference Table: 14.3.6.1; SOURCE: Listing 16.2.8.2.1 and 16.2.8.2.2)



## Appendix 1: Premier Research Library of Abbreviations

| Abbreviation | Definition |
|---|---|
| aCRF | annotated case report form |
| AE | adverse event |
| AESI | adverse events of special interest |
| ANCOVA | analysis of covariance |
| ATC | anatomical therapeutic chemical |
| ВМІ | body mass index |
| CDR-CCB | Continuity and Power of Attention, Working Memory, and Episodic<br>Memory on the Cognitive Drug Research Computerized Cognition<br>Battery |
| CFR | code of federal regulations |
| CĪ | confidence intervals |
| CISI-PD | Clinical Impression of Severity Index-Parkinson's Disease |
| СМН | Cochran-Mantel-Haenszel |
| CRF | case report form |
| CRO | contract research organization |
| cs | clinically significant |
| CSR | clinical study report |
| DB | database |
| DBL | database lock |
| DBP | diastolic blood pressure |
| dCDT | Digital clock drawing test |



| Abbreviation | Definition |
|---|---|
| DEA | drug enforcement administration |
| DIA | drug information association |
| D-KEFS | Delis-Kaplan Executive Function System |
| DOB | date of birth |
| EC | ethics committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| ЕМА | European medicines agency |
| FDA | food and drug administration |
| GCP | good clinical practice |
| GDS-15 | Geriatric Depression Scale-15 |
| HR | heart rate |
| IC or ICF | informed consent or informed consent form |
| ICH | international council for harmonization |
| ID | identification |
| ITT | intent-to-treat |
| IV | intravenous |
| MDS-UPDRS | the Movement Disorder Society's Unified Parkinson's Disease Rating Scale |
| MedDRA | medical dictionary for regulatory activities |
| MoCA | Montreal Cognitive Assessment |



| Abbreviation | Definition |
|--------------|------------------------------------------|
| MRI | Magnetic resonance imaging |
| N | number |
| NA | not applicable |
| NCS | non-clinically significant |
| PD | Parkinson's Disease |
| PD | protocol deviation |
| PDD | Parkinson's Disease with dementia |
| PD-MCI | PD with mild cognitive impairment |
| PE | physical examination |
| PP | per-protocol |
| PT | Preferred term |
| RR | respiratory rate or relative rate |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS® | a software system used for data analysis |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SOC | system organ class |
| S-STS | Sheehan Suicidality Tracking Scale |
| TEAE | treatment-emergent adverse event |
| tf-MRI | task-free functional MRI |



| Abbreviation | Definition |
|--------------|-------------------------------------------|
| UPCR | Urine protein-to-creatinine ratio |
| WHO | world health organization |
| WHO-DD | world health organization drug dictionary |



## Appendix 2: Bracket Statistical Analysis Plan for CDR